# **16.1.9 Documentation of Statistical Methods**

| Document | Date |
|----------------------------------------------------------|-----------------|
| Statistical Analysis Plan, Part A, Version 2.0 | 13 January 2021 |
| Statistical Analysis Plan, Part B, Version 1.0 | 13 January 2021 |
| Tables, Listings and Figures Shells, Part A, Version 2.0 | 13 January 2021 |
| Tables, Listings and Figures Shells, Part B, Version 2.0 | 22 January 2021 |

Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6



**Verona Pharma** PROTOCOL RPL554-MD-201

Statistical Analysis Plan v2.0 - Part A


# STATISTICAL ANALYSIS PLAN - PART A

# RPL554-MD-201

A Phase II, Randomized Study to Assess the Pharmacokinetics, Safety and Pharmacodynamics of Single and Repeat Doses of RPL554 Administered by Pressurised Metered Dose Inhaler in Patients with COPD

**AUTHOR:** NICHOLAS ROUBINIS/JENNIFER ALLSOPP

VERSION NUMBER AND DATE: V2.0, 13JAN2021

 $\label{locument} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ APV Pa$ 

Author: Nicholas Roubinis / Jennifer Allsopp Version Number: 2.0

Version Date: 13JAN2021

Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# STATISTICAL ANALYSIS PLAN - PART A SIGNATURE PAGE

Statistical Analysis Plan V2.0 – Part A (Dated 13JAN2021) for Protocol RPL554-MD-201.

| | Name | Signature | Date |
|-----------|------------------------|--------------------|-----------|
| Author: | Jennifer Allsopp | DocuSigned by: | 1/19/2021 |
| Position: | Senior Biostatistician | Jennifer allsopp — | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan – Part A, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Mark Shaw | DocuSigned by: | 1/19/2021 |
| Position: | Manager, Biostatistics | Mark Shaw<br>E2A9CBA2FB8F4B7 | ' |
| Company: | IQVIA | | |
| Approved By: | Tara Rheault | DocuSigned by: | 1/19/2021 |
| D :: | VD D C D | Tara Aleault | |
| Position: | VP, R&D | C1B201F76799452 | |
| Company: | Verona Pharma | | |
| Approved By: | Thomas Bengtsson | DocuSigned by: | 1/19/2021 |
| | | Thomas Bengtsson | 2, 23, 2322 |
| Position: | Statistical Consultant to V | 9570C0A2A259423 | |
| Company: | StatMind | | |

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 - Part A


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# **MODIFICATION HISTORY**

| Unique | Date of the | | |
|---|---|---|---|
| Identifier for | Document | | Significant Changes from |
| this Version | Version | Author | Previous Authorized Version |
| 1.0 | 28AUG2019 | Nicholas Roubinis/<br>Jennifer Allsopp | Not Applicable – First Version |
| 1.1 | 01APR2020 | Jennifer Allsopp | Update approver from Verona on signature page from Brian Maurer to Nancy Herje. Update protocol version SAP is based on in Section 1. |
| 1.2 | 09DEC2020 | Jennifer Allsopp | Update approver from Verona on signature page from Nancy Herje.to Tara Rheault |
| 2.0 | 13JAN2021 | Jennifer Allsopp | Add Thomas Bengtsson as an approver for Verona. |


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Version 1.0; 17 May 2021

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# TABLE OF CONTENTS

| 1.<br>2. | INTRODUCTION | |
|---|---|---|
| 2.1. | Primary Objective | .8 |
| 2.2. | Secondary Objectives | .8 |
| 3. | STUDY DESIGN | 9 |
| 3.1. | General Description | .9 |
| 3.2. | Schedule of Events | 10 |
| 3.3. | Changes to Analysis from Protocol | 10 |
| 4. | PLANNED ANALYSES | 0 |
| <ul><li>4.</li><li>4.1.</li></ul> | PLANNED ANALYSES | |
| | | 11 |
| 4.1. | Data Monitoring Committee (DMC) | 11 |
| 4.1.<br>4.2. | Data Monitoring Committee (DMC) | l 1<br>l 1 |
| 4.1.<br>4.2.<br>4.3. | Data Monitoring Committee (DMC) | 11 |
| 4.1.<br>4.2.<br>4.3. | Data Monitoring Committee (DMC) | 11 |

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


| 5.5. | Pharmacokinetics [PK] Analysis Set | 13 |
|---|---|---|
| 6. | GENERAL CONSIDERATIONS | 13 |
| 6.1. | Reference Start Date and Study Day | 13 |
| 6.2. | Baseline | 14 |
| 6.3. | Repeat/reschedule, Unscheduled Visits and Early Termination Data | 14 |
| 6.4. | Windowing Conventions | 14 |
| 6.5. | Statistical Tests | 15 |
| 6.6. | Common Calculations | 15 |
| 6.7. | Software Version | 16 |
| 7. | STATISTICAL CONSIDERATIONS | 16 |
| 7.1. | Adjustments for Covariates and Factors to be Included in Analyses | 16 |
| 7.2. | Multicenter Studies | 16 |
| 7.3. | Missing data | 17 |
| 7.4. | Multiple Comparisons/ Multiplicity | 17 |
| 7.5. | Examination of Subgroups | 18 |
| 8. | OUTPUT PRESENTATIONS | 18 |
| 9. | DISPOSITION AND WITHDRAWALS | 18 |
| <b>10.</b> | DEMOGRAPHIC AND OTHER SCREENING CHARACTERISTICS | 19 |


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Reference: CS\_WI\_BS005

Statistical Analysis Plan v2.0 - Part A


| 10.1. Derivations | | 20 |
|---|---|---|
| 11. SURGICAL, MEDICAL AND CHRONIC OF DISEASE/SMOKING HISTORY | | |
| 12. MEDICATIONS | | |
| 13. STUDY MEDICATION EXPOSURE | | |
| 14. STUDY MEDICATION COMPLIANCE | | |
| 15. EFFICACY OUTCOMES | ••••• | 23 |
| 15.1. Primary Efficacy | | |
| 15.1.1. Primary Efficacy Variable(s) & Derivation(s) | | |
| 15.1.3. Primary Analysis of Primary Efficacy Variable(s) | | |
| 13.1.3. Timary final folia of Final grant Entered Communications | | 20 |
| 15.2. Secondary Efficacy | ••••• | 24 |
| 15.2.1. Secondary Efficacy Variables & Derivations | | |
| 15.2.1.1. Change in baseline in average $FEV_1$ of $AUC_{0-4h}$ | (Average FEV <sub>1</sub> over 4 hour | s) after single dose |
| (Secondary variable 1) | Avaraga EEV, avar 12 haurs | 24 |
| (Secondary variable 2) | | |
| 15.2.1.3. Change from baseline in peak FEV <sub>1</sub> (measured) | | |
| variable 3) 25 | | • |
| 15.2.2. Missing Data Methods for Secondary Efficacy Varia | ble(s) | 26 |
| 15.2.3. Analysis of Secondary Efficacy Variables | | 26 |
| 16. SAFETY OUTCOMES | ••••• | 27 |
| 16.1. Adverse Events | | |
| 16.1.1. All TEAEs | | |
| 16.1.1.1. Severity | | |
| 16.1.1.2. Relationship to Study Medication | | |
| 16.1.2. TEAEs Leading to Discontinuation of Study Medica<br>16.1.3. Serious Adverse Events | | |
| 16.1.4. Adverse Events Leading to Death | | |
| Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Veror | na RPL554-MD-201 SAP v2.0 – Pa | art A |

Effective Date: 01Apr2018

Template No.: CS\_TP\_BS016 Revision 5


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


| 16.2. Laboratory Evaluations 16.2.1. Laboratory Reference Ranges and Markedly Abnormal Criteria | |
|---|---|
| 16.3. ECG Evaluations | 30 |
| 16.4. Vital Signs | 31 |
| 16.5. Physical Examination | 32 |
| 16.6. Other Safety Assessments | 33 |
| 17. PHARMACOKINETIC EVALUATIONS | 33 |
| 18. REFERENCES | 34 |
| APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | 35 |
| IQVIA Output Conventions | 35 |
| Table and Listing Output Conventions | 35 |
| Figure Output Conventions | 38 |
| Dates & Times | 38 |
| Spelling Format | 38 |
| Presentation of Treatment Groups | 38 |
| Presentation of Visits | 39 |
| Listings | 39 |
| APPENDIX 2. PARTIAL DATE CONVENTIONS | 40 |
| Algorithm for Treatment Emergence of Adverse Events | 40 |


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


### 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy, safety and pharmacokinetic (PK)/pharmacodynamic (PD) data for Part A of protocol RPL554-MD-201. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed. This statistical analysis plan (SAP) is based on the protocol version 3.0, dated 24DEC2019. The study will consist of two parts (A and B) and Part A will be described in this SAP while a separate SAP for Part B will be created prior to the start of Part B. Only the protocol sections applicable to Part A will be described in this SAP.

### 2. STUDY OBJECTIVES FOR PART A

### 2.1. PRIMARY OBJECTIVE

The primary objective of Part A is to investigate the PK profile of single doses of RPL554, administered by pressurized metered dose inhaler (pMDI), in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

# 2.2. SECONDARY OBJECTIVES

The secondary objectives of this part are as follows:

- To investigate the safety and tolerability of single doses of RPL554 administered by pMDI, including effects on peak pulse and heart rate.
- To investigate the bronchodilator effect of single doses of RPL554 administered by pMDI, in terms of peak
  FEV<sub>1</sub> (forced expiratory volume in one second), average FEV<sub>1</sub> area under the curve (AUC)<sub>0-4h</sub> and average
  FEV<sub>1</sub> AUC<sub>0-12h</sub>.

 $\label{locumentation} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ A$ 


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 3. STUDY DESIGN

### 3.1. GENERAL DESCRIPTION

This is a Phase II, randomized, double-blind, placebo-controlled, two-part study. Part A is a parallel group, single dose assessment of RPL554 administered by pMDI to evaluate the safety and terminal PK profile of a range of doses of RPL554. Five dose levels, 100 µg, 300 µg, 1000 µg, 3000 µg and 6000 µg (single-blind) were selected, covering a 60-fold increase in doses. A total of approximately 36 COPD patients (as defined by the American Thoracic Society [ATS]/European Respiratory Society [ERS] guidelines with symptoms compatible with COPD for at least 1 year prior to Screening) aged 40 to 80 years (inclusive) will be randomized at two study centres in the United Kingdom (UK). At the end of Part A, a data cut-off will be used, selected data unblinded and analyzed prior to commencing Part B. Up to four active doses will be selected for Part B, which will include all Part A patients. Part B is designed as a complete block crossover, repeat dose assessment of RPL554 administered by pMDI to evaluate the steady state efficacy/PD effect of the doses compared to the effect with placebo pMDI. The patients in Part B will undergo up to five treatment periods.

In Part A, patients will be screened for eligibility, including a reversibility test with albuterol between 7 and 14 days before the single dose of study treatment. Eligible patients will then be given a single dose of RPL554 or placebo and assessed for 12 hours. They will then return to the clinic the following day for a 24-hour post-dose assessment of PK and lung function.

In Part B, the patients from Part A will be randomly assigned in crossover fashion to one of 4 treatment sequences (if there are 4 treatment groups in Part B), or 10 treatment sequences (if there are 5 treatment groups in Part B) each consisting of up to five 1-week treatment periods separated by a 7 to 10-day washout. Each treatment period consists of 6 days of twice daily doses of RPL554, and a single morning dose on Day 7. In each treatment period, patients will undergo assessments over 12 hours on Days 1 and 7. Figure 1 below and Figure 1 in the protocol summarize these details.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


Figure 1 Study Flow Chart



Abbreviations: TBD=to be determined; TP=Treatment Period

# 3.2. SCHEDULE OF EVENTS

Schedule of events can be found in Section 6 of the protocol.

# 3.3. CHANGES TO ANALYSIS FROM PROTOCOL

Not applicable.

# 4. PLANNED ANALYSES

There are no data monitoring committee (DMC) or formal interim analyses to be performed for this study. The study will consist of two separate and independent analyses, Part A and Part B. At the end of Part A, a data cut-off will be used, selected data unblinded and analyzed prior to commencing Part B. At the end of Part B, the database will be locked and unblinded, and the full analyses for each part will be performed.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# 4.1. DATA MONITORING COMMITTEE (DMC)

There will be no DMC analyses for this study.

### 4.2. INTERIM ANALYSIS

No formal interim analysis is planned for the study.

### 4.3. PART A ANALYSIS

Selected Part A analysis will be performed by IQVIA Biostatistics following the data cut-off. All Part A analyses identified in this SAP will be performed by IQVIA Biostatistics following the Part B Database Lock on a clean database:

- All outstanding data issues and queries resolved.
- All irresolvable data issues documented in the Data Handling Report (DHR) from Data Management.
- All coding of medications and adverse events (AEs) completed.
- Serious AE (SAE) reconciliation completed.
- All reconciliation of vendor data with electronic case report form (eCRF) data completed successfully.
- Analysis sets authorized.

It should be noted that the main teams performing the Part A analysis will remain blinded at the time of the Part A data cut-off. This is to avoid any potential risk they could trace what study medication a patient might be receiving in Part B (e.g. if they know they experienced certain AEs while on one treatment in Part A and identify this in Part B).

All verbatim text from the eCRF will be presented in outputs "as is" with no "manual hard coding" corrections for such data. Also, PK analysis will be performed by another party (third party vendor).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# 5. ANALYSIS SETS

Agreement and authorization of patients included/excluded from each analysis set will be conducted prior to the unblinding of the study for Part A.

# 5.1. ALL PATIENTS ENROLLED SET [ENR]

The all patients enrolled (ENR) set will contain all patients who provide informed consent for this study.

# 5.2. ALL PATIENTS RANDOMIZED SET [RND]

The all patients randomized (RND) set will contain all patients who provide informed consent and who are randomized to study medication. For analyses and displays based on RND, patients will be classified according to randomized treatment.

# 5.3. SAFETY ANALYSIS SET [SAF]

The safety analysis set (SAF) will contain all patients in the RND set who received the single dose of study medication during Part A. Patients will be classified according to actual treatment received. If there is any doubt whether a patient was treated or not, they will be assumed treated for the purposes of analysis.

# 5.4. FULL ANALYSIS SET [FAS]

The full analysis set (FAS) will contain all patients in the RND set with data collected after intake of study medication to compute the pharmacodynamic parameters ( $FEV_1$  measurements pre-dose and at least one post-baseline). For analyses and displays based on FAS, patients will be classified according to planned treatment.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 5.5. PHARMACOKINETICS [PK] ANALYSIS SET

The PK analysis set will contain all patients in the RND analysis set who have a blood sampling performed after the single dose of RPL554 and PK parameter data. The PK analysis set will be determined by a third-party vendor and the data will be provided to IQVIA.

# 6. GENERAL CONSIDERATIONS

# 6.1. REFERENCE START DATE AND STUDY DAY

Study day will be calculated from the reference start date and will be used to show start/stop day of assessments and events. Reference start date is defined as the day of the single dose of study medication and will appear in every listing where an assessment date or event date appears.

If the date of the event is on or after the reference date, then:

• Study day = (date of event – reference date) + 1.

If the date of the event is prior to the reference date, then:

• Study day = (date of event – reference date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, and study day, and any corresponding durations will be presented based on the imputations specified in <u>Appendix 2</u>; Partial Date Conventions.

 $\label{locumentation} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ A$ 


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# **6.2.** BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to the single dose assessment (including unscheduled assessments). For FEV<sub>1</sub> and forced vital capacity (FVC), baseline is defined as the average of the two pre-dose assessments (at 1-hour [±5 minutes] and immediately [within 5 minutes] pre-dose).

# 6.3. REPEAT/RESCHEDULE, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the nominal visit will be presented. If a visit is repeated/rescheduled due to variability in  $FEV_1$  or other reason, the repeated/rescheduled visit, will be listed and summarized as the valid visit (same visit number assigned). Unscheduled measurements will not be included in by-visit summaries, but will contribute to the endpoint value. For example, if an unscheduled visit occurred at 10 hours post-dose on the day of the single dose, then this value will be considered in the calculation of the average  $FEV_1$  over 12 hours ( $AUC_{0.12h}FEV_1$ ). Any unscheduled or unplanned readings will be presented within the patient listings.

Early termination data will be mapped according to the visit number the termination occurred for by-visit summaries. In Part A early terminations can occur at Screening, Day 1 and Day 2. If termination is between Part A and Part B, data are to be considered in the Part B SAP. Subject will be a completer of Part A.

Listings will include scheduled, unscheduled, repeat/reschedule and early discontinuation data.

# **6.4.** WINDOWING CONVENTIONS

No visit windows will be applied in this study and the scheduled assessments will be reported and analyzed as per eCRF collection.

 $\label{locumentation} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ A$ 


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# **6.5. STATISTICAL TESTS**

The default significant level will be (5%); confidence intervals will be 95% and all tests will be 2-sided, unless otherwise specified in the description of the analyses. All significant p-values (i.e. < 5%) will be flagged by means of a "\*" for ease of review.

For presentation of summary statistics for quantitative and qualitative variables see <u>Appendix 1</u>; Programming conventions for outputs.

### 6.6. COMMON CALCULATIONS

For quantitative measurements, change from baseline will be calculated as:

• Test value at post-dose timepoint – baseline value.

For quantitative measurement values of FEV1 and FEV1 AUCs will be calculated based on:

- The highest FEV<sub>1</sub> reading from each assessment.
- The baseline value (average of the two pre-dose values [at 1-hour {±5 minutes} and immediately {within 5 minutes}} pre-dose) must be within ± 20% of the pre-albuterol value at Screening; otherwise, the patient will be a screen failure.

Peak effect will be calculated as:

• Maximum value in the first 4 hours after dosing.

Average effect will be calculated as:

• FEV<sub>1</sub> AUC divided by the length of the time interval of interest.

Log-transformations will be performed on  $FEV_1$  data:

FEV<sub>1</sub> will be analyzed using multiplicative models, which means that data will be logged prior to analysis. The
results will then be back-transformed to linear scale (treatment differences will thus be ratios of geometric
means).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# **6.7. SOFTWARE VERSION**

All analyses will be conducted using SAS version 9.4.

### 7. STATISTICAL CONSIDERATIONS

# 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The following covariates are used in the analyses. For details of their inclusion in the models, see the specific analysis section.

- Randomized treatment (fixed).
  - o RPL554 100μg
  - o RPL554 300μg
  - o RPL554 1000μg
  - o RPL554 3000μg
  - o RPL554 6000μg
  - o Placebo
- Baseline value of analyzed variable (covariate).

# 7.2. MULTICENTER STUDIES

This study will be conducted at 2 study centers, in the UK.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 7.3. MISSING DATA

Missing safety data will not be imputed, apart from partial date imputations as specified in <u>Appendix 2</u>. Missing efficacy data will be handled as described in <u>Section 15.1.2</u> and <u>Section 15.2.2</u> of this SAP.

# 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

Significance of treatment effect will be tested for the primary and secondary efficacy endpoints in Part A and will be done for each of the doses of RPL554 against placebo, starting with the highest dose ( $6000 \mu g$ ). To this end, the fixed-sequence testing approach (Maurer et al., 1995; Westfall & Krishen, 2001) will be used.

For the endpoints, let i=0,1,2,3,4 and 5 represent increasing dose levels, 0 denoting placebo. Also, let  $\mu_i$ , i=0,1,2,3,4 and 5 denote the mean change from baseline for the endpoint of interest for placebo and each increasing active dose level, respectively. The null hypotheses are defined as:  $H_i$ :  $\mu_j - \mu_0 = 0$  and will be tested against the 2-sided alternative  $K_i$ :  $\mu_j - \mu_0 \neq 0$ , j=1,2,3,4 and 5.

Finally, let  $p_1$ ,  $p_2$ ,  $p_3$ ,  $p_4$ ,  $p_5$  denote the marginal p-values obtained from the statistical tests associated with  $H_1$ ,  $H_2$ ,  $H_3$ ,  $H_4$ ,  $H_5$  (obtained from the model).

The fixed-sequence testing will begin with the null hypothesis corresponding to the highest dose versus placebo. If a statistically significant difference is found at the 2-sided  $\alpha$  level of 5%, the testing will proceed with the next highest dose. Otherwise, testing stops, and the remaining null hypotheses are considered as failed to reject, without testing.

This testing strategy can be written as the following stepwise algorithm:

- $\bullet \quad \text{Step 1: If } p_5 \leq \alpha \text{ reject } H_5 \text{ and go to Step 2. Otherwise, fail to reject } H_5, H_4, H_3, H_2 \text{ and } H_1 \text{ and stop.} \\$
- Step 2: If  $p_4 \le \alpha$  reject  $H_4$  and go to Step 3. Otherwise, fail to reject  $H_4$ ,  $H_3$ ,  $H_2$  and  $H_1$  and stop.
- $\bullet \quad \text{ Step 3: If } p_3 \leq \alpha \text{ reject } H_3 \text{ and go to Step 4. Otherwise, fail to reject } H_3, H_2 \text{ and } H_1 \text{ and stop.}$
- $\bullet \quad \text{Step 4: If } p_2 \leq \alpha \text{ reject } H_2 \text{ and go to Step 5. Otherwise, fail to reject } H_2 \text{ and } H_1 \text{ and stop.}$
- $\bullet \quad \text{ Step 5: If } p_1 \leq \alpha \text{ reject } H_1. \text{ Otherwise, accept } H_1.$

The fixed-sequence procedure controls the family-wise error rate in the strong sense because, for each null

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


hypothesis, the testing is conditional upon rejecting all hypotheses earlier in the sequence (Dmitrienko, et al., 2009).

Each secondary endpoint will be tested independently and nominally following a hierarchical testing of doses like the one used for the primary endpoint.

# 7.5. EXAMINATION OF SUBGROUPS

No subgroup analyses will be performed for this study.

### 8. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics.

# 9. DISPOSITION AND WITHDRAWALS

All patients who provide informed consent will be accounted for in this study.

Patient disposition, withdrawals and reasons for exclusion from each analysis set and protocol deviations, including exception to the inclusion and exclusion criteria will be presented for all patients, including those with screen failures and summarized by treatment group for the RND analysis set. Number of patients treated and discontinued will also be presented. If the patient discontinued/withdraws, he/she will be allocated to the single dose treatment group administered.

All protocol deviations collected in Part A will be divided into critical, major or minor categories and will be assigned to the single dose treatment group. These which will be summarized by treatment and presented in a listing for the RND analysis set. Protocol deviations affect the integrity of the drug activity data and will be obtained by the

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


clinical research associates (CRAs) and documented in the clinical trial management system (CTMS). Each protocol deviation is categorized into one of the following types, based on CTMS:

- 1. Informed Consent Criteria
- 2. Eligibility and Entry Criteria
- 3. Concomitant Medication Criteria
- 4. Laboratory Assessment Criteria
- 5. Study Procedures Criteria
- 6. Serious Adverse Event Criteria
- 7. Randomization Criteria
- 8. Visit Schedule Criteria
- 9. Investigation Product (IP) Compliance
- 10. Efficacy Criteria
- 11. Administrative Criteria
- 12. Source Document Criteria
- 13. Regulatory or Ethics Approvals Criteria
- 14. Other Criteria

Preliminary assignment to each analysis population, therefore whether a patient is included/excluded in each analysis population (excluding the PK analysis population) will be recorded in an EXCEL sheet by the IQVIA Biostatistician, with the reason for exclusion from each population indicated. The EXCEL sheet should then be authorized by means of a customer authorization form (CAF) and prior to the Database Lock of the study.

### 10. DEMOGRAPHIC AND OTHER SCREENING CHARACTERISTICS

Demographic data and other baseline characteristics (including screening disease characteristics) will be presented for all analysis sets (RND, SAF, FAS, PK), by treatment groups, if the analysis sets differ to each other. If these are the same, as is expected for Part A, the presentation will be limited to just the RND analysis set, or to those that are

 $\label{locumentation} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ A$ 


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


different. No statistical testing will be carried out for demographic or other baseline characteristics. The following demographic and other baseline characteristics will be reported for Part A:

- Age (years)
- Sex
- Childbearing potential
- Race
- Ethnicity
- Height (cm)
- Weight (kg)
- BMI (kg/m<sup>2</sup>)
- Pre (prior to dosing at baseline)/post (post dosing at baseline) bronchodilator FEV<sub>1</sub> (both in liters and in percentage of predicted normal)
- Pre/Post-bronchodilator FEV<sub>1</sub>/FVC
- FEV<sub>1</sub> reversibility test (mL and %)
- Reversibility assessment performed with four puffs of Albuterol
- Met requirements of reversibility test

# 10.1. DERIVATIONS

- Age (years) = (Informed consent date date of birth)
- BMI  $(kg/m^2)$  = weight (kg)/ height  $(m)^2$

Demographic and other screening characteristics recorded on the eCRF will be used as is on the eCRF, without any derivations or adjustments.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 11. SURGICAL, MEDICAL AND CHRONIC OBSTRUCTIVE PULMONARY DISEASE/SMOKING HISTORY

Surgical and Medical History information will be presented in table summaries and listings, for the RND analysis set

- · Surgical History will not be coded.
  - Surgical History conditions are defined as those conditions which stop prior to or at Screening.
- Medical History will be coded by MedDRA dictionary using the version specified in the data management plan.
  - Medical History conditions are defined as those conditions which stop prior to or at Screening.
  - Data captured on the Medical History page of the eCRF will be presented by SOC and PT.
- COPD/Smoking History data captured on the COPD and Smoking History page of the eCRF will be presented for the RND analysis set.
  - COPD history (Duration of COPD [calculated relative to date of first diagnosis {Randomization date –
    first COPD diagnosis date}], date of most recent exacerbation, known to have chronic
    bronchitis/emphysema)
  - Smoking history (current or former smoker, number of packs per day, number of years smoking and number of pack-years [calculated as number of packs per day x number of years smoking])

### 12. MEDICATIONS

Medications will be coded using the World Health Organization – Drug Dictionary (WHO-DD) version specified in the data management plan and will be presented in a listing by Anatomical Therapeutic Chemical (ATC) (the 1st level of the ATC code) and PT for the RND analysis set. Certain medications (or a special grouping of medications) will be classified in a list during the study and signed-off prior to lock by a medical advisor. As this list, may change prior to sign-off they will not be defined in this section of the SAP. Potential medications include, but are not limited to, inhaled corticosteroids (ICS), LAMAs (long-acting muscarinic antagonists), LABAs (long-acting beta2-agonists) etc.

 $\label{locumentation} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ A$ 


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


See <u>Appendix 2</u> for handling of partial dates for medications, in the case where it is not possible to define a medication as prior, concomitant, or post treatment, the medication will be classified by the worst case; i.e. concomitant.

- 'Prior' medications are medications which started and stopped in the 3 months prior to the single dose of study
  medication and are recorded at Screening.
- 'Concomitant' medications are medications which:
  - o Had an onset date on or after the single dose of study medication.
  - o AND ended on or after the date of single dose of medication or were ongoing at the end of Part A.
  - o A patient can report more than 1 concomitant medication with the same PT.

Prior and concomitant medications will be presented in a listing only, by treatment group.

Rescue medications will be recorded on the Rescue Medication/Rescue Medication Canister Collection/Rescue Medication Canister Dispensed/Rescue Medication Canister Weight pages of the eCRF. These are short acting bronchodilators and will be sourced by the study center and dispensed at the Screening visit and end of Part A (Day 2). Rescue medication used during study visits will be documented on the eCRF pages. Protocol procedures must continue even if rescue medication has been taken. Salbutamol/albuterol is to be used for primary rescue use.

Rescue medications used during study visits (by recording the time it was dispensed and collected) and the amount taken between Day 1 and Day 2 (by recording the weight of the canisters), will be presented in a listing for the RND analysis set.

When a rescue medication is used less than 8 or 6 hours (for protocol version 1 or 2 respectively) prior to pre-dose spirometry or between the pre-dose and 12-hour post-dose spirometry a sensitivity analysis will be carried out. For the analysis detailed in Section 15.2.1.2 patients who took rescue medication will be removed. This will only be carried out if at least 1 patient has taken rescue medication less than 8 or 6 hours (for protocol version 1 or 2 respectively) prior to pre-dose spirometry or between the pre-dose and 12-hour post-dose spirometry.

 $\label{locumentation} \textbf{Document:} \qquad Z:\ RPL554\ EZAA8488\ Biostatistics\ Documentation\ SAP\ Verona\ RPL554-MD-201\ SAP\ v2.0-Part\ APV Part\ A$ 


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# 13. STUDY MEDICATION EXPOSURE

Date and time of exposure to the single dose of study medication and the date of completion/discontinuation will be presented in a listing for the RND analysis set. Duration of exposure will not be calculated as this is expected to be one day for all patients in Part A. The information to be listed will be taken from the Drug Exposure and Disposition eCRF pages.

# 14. STUDY MEDICATION COMPLIANCE

All administration of study treatment will be done at the clinic under supervision of the study staff; therefore, no formal analysis of compliance will be performed.

### 15. EFFICACY OUTCOMES

### 15.1. PRIMARY EFFICACY

# 15.1.1. PRIMARY EFFICACY VARIABLE(S) & DERIVATION(S)

• Not applicable – The primary endpoint of Part A will be described in <u>Section 17</u>.

# 15.1.2. MISSING DATA METHODS FOR PRIMARY EFFICACY VARIABLE(S)

Not applicable.

### 15.1.3. PRIMARY ANALYSIS OF PRIMARY EFFICACY VARIABLE(S)

Not applicable.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# 15.2. SECONDARY EFFICACY

The secondary efficacy analyses will be performed for the FAS.

### 15.2.1. SECONDARY EFFICACY VARIABLES & DERIVATIONS

# 15.2.1.1. Change in baseline in average FEV<sub>1</sub> of AUC<sub>0-4h</sub> (Average FEV<sub>1</sub> over 4 hours) after single dose (Secondary variable 1)

Average  $FEV_1$  after single dose is defined as the  $AUC_{0-4h}FEV_1$  collected, divided by the length of the time (in hours).  $AUC_{0-4h}FEV_1$  is derived using the following formula:

$$AUC = \frac{1}{2}(t_1 - t_0)(y_1 + y_0) + \frac{1}{2}(t_2 - t_1)(y_2 + y_1) + \dots + \frac{1}{2}(t_i - t_{i-1})(y_i + y_{i+1})$$

where i are the number of intervals,  $t_i$  are the time values or time intervals (in actual hours) between assessments and  $y_i$  the FEV<sub>1</sub> values at  $t_i$ . The AUC result will then be divided by the actual time (the time elapsed since dosing, until the time of assessment) at 4-hour assessment (as this can occur  $\pm$  10 minutes) to obtain the average FEV<sub>1</sub>. If the assessment at 4-hour is missing, the AUC result will be divided by the actual time of the last collected assessment. For analysis purposes, it will be assumed that the pre-dose value (immediately pre-dose) occurred at time 0 when computing PD parameters. If a patient misses hour 2 and 4 then the AUC<sub>0-4</sub> is set to missing.

Descriptive statistics (see Appendix 1 [Programming conventions for outputs]) for  $AUC_{0.4}$  will be presented for all patients assigned to FAS, at each assessment and change from baseline at each assessment as relevant. All summaries will be presented for each treatment group. In addition, a figure (bar graph) representing mean change from baseline FEV<sub>1</sub> to FEV<sub>1</sub>  $AUC_{0.4}$  by treatment will be presented, including the standard error of the mean.

Change from baseline  $FEV_1$  to  $FEV_1$  AUC<sub>0-4</sub> will be derived to test the hypothesis described in <u>Section 15.2.3</u> with baseline defined as the average of the  $FEV_1$  pre-dose assessments (-60 minutes and -5 minutes) collected.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 15.2.1.2. Change in baseline in average FEV<sub>1</sub> AUC<sub>0-12h</sub> (Average FEV<sub>1</sub> over 12 hours) after single dose (Secondary variable 2)

 $AUC_{0.12h}$  FEV<sub>1</sub> after single dose is defined and derived similarly to secondary endpoint above (see Section 15.2.1.1), but over 12-hours post-dose. If the assessment at 12-hours is missing, the AUC result will be divided by the actual time of the last collected assessment. If patient misses hours 11 and 12 then the  $AUC_{0.12h}$  is set to missing.

# 15.2.1.3. Change from baseline in peak FEV<sub>1</sub> (measured in first 4 hours) after single dose (Secondary variable 3)

Peak  $FEV_1$  is measured in the first 4 hours after single dose. It is collected on the Spirometry Study measurements eCRF page.

Three acceptable readings are performed at each of the timepoints in first 4 hours after the single dose (5, 15 and 30 minutes and 1, 1.5, 2 and 4 hours) and the highest of the 3 is used for analysis purposes. Hence peak FEV<sub>1</sub> is derived as the highest of all these readings.

Descriptive statistics (see Appendix 1 [Programming conventions for outputs]) for peak  $FEV_1$  will be presented for all patients assigned to FAS, at each assessment and change from baseline as relevant. All summaries will be presented for each treatment group. In addition, a figure (bar graph) representing mean change from baseline  $FEV_1$  to peak  $FEV_1$  by treatment will be presented, including the standard error of the mean. A figure also displaying the mean change over time on Day 1 will be presented.

Change from baseline  $FEV_1$  to peak  $FEV_1$  (over 4 hours) will be derived to test the hypothesis described in <u>Section 15.2.3</u> with baseline defined as the average of the  $FEV_1$  pre-dose assessments (-60 minutes and -5 minutes) collected.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


### 15.2.2. MISSING DATA METHODS FOR SECONDARY EFFICACY VARIABLE(S)

No imputation will be applied.

#### 15.2.3. ANALYSIS OF SECONDARY EFFICACY VARIABLES

The secondary variables will be analyzed by comparing the RPL554 treatment groups to each other and placebo by rejecting the null hypothesis described below at significance level  $\alpha$ =0.05 level (2-sided):

```
H_0\text{: }\mu_j\!=\mu_0\text{ versus }H_1\text{: }\mu_j\!\neq\mu_0
```

where  $\mu_j$  and  $\mu_0$  are the mean change from Baseline for each parameter (Peak FEV<sub>1</sub>, AUC<sub>0-4h</sub> and AUC<sub>0-12h</sub>) after single dose for each respective dose of RPL554 and placebo.

ANCOVA analyses will be implemented using the SAS® procedure MIXED as follows:

```
PROC MIXED DATA = ...;

CLASS TREATMENT;

MODEL CHG = TREATMENT BASELINE;

LSMEANS TREATMENT / CL DIFF;

RUN;
```

where CHG = difference in log (parameter) – log (baseline parameter) i.e. log (parameter / baseline parameter) TREATMENT = treatment group (Respective dose of RPL554,  $100\mu g$ ,  $300\mu g$ ,  $1000\mu g$ ,  $3000\mu g$  and  $6000\mu g$  and placebo)

BASELINE = log (baseline parameter)

The primary comparison will be the contrast (difference in least squares mean [LSMEAN]) between  $6000\mu g$  RPL554 and placebo. The parameter value and its baseline will be log-transformed prior to analysis using natural logarithm. The difference between the two (log [parameter] – log [baseline parameter] equals log (parameter /

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 - Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


baseline parameter). The covariate, baseline parameter, will also be log transformed. Therefore, the LSMEAN statement between treatments in the above PROC MIXED will provide the log of the contrasts. Prior to presentations, the antilog of these point estimates and associated 95% confidence intervals will be performed, giving ratios of geometric means on the linear scale. The 2-sided p-value for the exponential (exp)least squares mean, exp(LSM), ratio between each of the 2 treatment groups and placebo will be reported.

Summary statistics for each parameter (Peak  $FEV_1$ ,  $AUC_{0-4h}$  and  $AUC_{0-12h}$ ) will be presented for baseline, at point of interest and change from baseline by treatment group on patients with both assessments, on the original scale.

### 16. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the SAF.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified with the relevant section.

# 16.1. ADVERSE EVENTS

Adverse Events (AEs) will be coded by MedDRA dictionary using the version specified in the data management plan.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the single dose of study medication, based on the investigator assessment of severity. TEAEs will be assigned to treatment groups based on actual treatment received.

See <u>Appendix 2</u> for handling of partial dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, the AE will be classified by the worst case; i.e. treatment emergent.


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


An overall summary of number of patients within each of the categories described in the sub-section below, will be provided as specified in the templates.

Listings will include TEAEs and Non-TEAEs.

### **16.1.1. ALL TEAES**

Incidence of TEAEs will be presented by System Organ Class (SOC) and Preferred Term (PT) and broken down further by maximum severity and relationship to study medication.

### 16.1.1.1. Severity

Severity is classed as mild/ moderate/ severe (increasing severity). TEAEs starting after the single dose of study medication with a missing severity will be classified as severe. If a patient reports a TEAE more than once within that SOC/ PT, the AE with the worst-case severity will be used in the corresponding severity summaries.

### 16.1.1.2. Relationship to Study Medication

Relationship, as indicated by the Investigator, is classed as "yes" or "no". A related TEAE is defined as a TEAE with a relationship to study medication as "yes". TEAEs with a missing relationship to study medication will be regarded as relationship = "yes" to study medication. If a patient reports the same AE more than once within that SOC/ PT, the AE with the worst-case relationship to study medication will be used in the corresponding relationship summaries.

### 16.1.2. TEAES LEADING TO DISCONTINUATION OF STUDY

TEAEs leading to discontinuation from the study will be identified by using the question "Did the AE cause the Patient to discontinue from the study?" from the AE page of the eCRF.

For TEAEs leading to discontinuation from the study, summaries of incidence rates (frequencies and percentages)

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 - Part A

Author: Version Number: 2.0


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


by SOC and PT will be prepared.

### 16.1.3. SERIOUS ADVERSE EVENTS

Serious adverse events (SAEs) are those events recorded as "Serious" on the Adverse Events page of the eCRF. A summary of serious TEAEs by SOC and PT will be prepared, similarly to Section 16.1.1 and Section 16.1.2.

### 16.1.4. ADVERSE EVENTS LEADING TO DEATH

TEAEs leading to Death are those events which are recorded as "Death" on the Adverse Events page of the eCRF. A summary of TEAEs leading to death by SOC and PT will be prepared.

# 16.2. LABORATORY EVALUATIONS

Results from the local laboratory will be included in the reporting of this study for hematology, blood chemistry, urinalysis and viral serology. A list of laboratory assessments to be included in the outputs is included in the protocol, Sections 7.4.3.1, 7.4.3.2,7.4.3.3 and 7.1.4 for hematology, blood chemistry, urinalysis and viral serology, respectively. Presentations will use International system (SI) units.

Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of quantification (BLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

The following summaries will be provided for laboratory data:

- Actual results at Screening.
- Incidence of abnormal values at Screening according to normal range criteria
- Listing of all laboratory evaluations and abnormal values at Screening.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


### 16.2.1. LABORATORY REFERENCE RANGES AND MARKEDLY ABNORMAL CRITERIA

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

In addition to the high and low quantitative laboratory assignments (as identified by means of the laboratory reference ranges), markedly abnormal quantitative blood chemistry values per the table below will also be identified by the Investigator.

| | Blood Chemistry –<br>Markedly Abnormal Definition |
|---|---|
| Alanine Aminotransferase (ALT) | > 3 x ULN |
| Alkaline Phosphatase (ALP) | > 3 x ULN |
| Aspartate Aminotransferase (AST) | > 3 x ULN |
| Creatinine | > 221 μmol/L |
| Gamma Glutamyl Transferase (GGT) | > 3 x ULN |
| Bilirubin (TBL) | > 3 x ULN |

ULN: Upper limit of normal. ALT: Alanine aminotransferase. AST: Aspartate aminotransferase.

ALP: Alkaline phosphatase. TBL: Total bilirubin.

# 16.3. ECG EVALUATIONS

Overall results from the local ECG (Electrocardiogram) lab will be included in the reporting of this study. The overall assessment of ECG parameters will be reported for this study:

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


- Normal
- Abnormal not Clinically Significant (ANCS)
- Abnormal Clinically Significant (ACS)
- Incomplete
- Uninterpretable

The following summaries will be provided for quantitative ECG data, for example heart rate:

- Actual assessments at screening, baseline (pre-dose of single dose) and each post-dose timepoint (1, 2, 4 and 8 hours)
- Change from Baseline at each post-dose timepoint assessment
- Shift of overall assessment baseline to post-dose timepoints according to Normal, ANCS and ACS overall
  assessment criteria
- Listing of all ECG evaluations and abnormal values

Peak heart rate after single dose is defined as the maximum value measured in the first 4 hours post-dose. Peak heart rate and change from baseline to peak will be summarized similarly to <u>Section 15.2.1.3</u>, including the figure presentations. In addition, hypothesis testing as per <u>Section 15.2.3</u>, will be repeated for this endpoint.

### 16.4. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Supine Systolic Blood Pressure (mmHg)
- Supine Diastolic Blood Pressure (mmHg)
- Supine Pulse Rate (bpm)

The following summaries will be provided for vital signs data:

• Actual assessments at screening, baseline (pre-dose of single dose) and each post-dose timepoint (1, 2, 4, 8, 12


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


and 24 hours [Day 2])

- Change from Baseline at each post-dose timepoint assessment
- Incidence of markedly abnormal values based on the criteria presented in the table below:

| | Low | High |
|---|---|---|
| Systolic blood pressure (mmHg) | Value ≤ 90 mmHg | Value ≥ 180 mmHg |
| | Decrease from Baseline of ≥ 40 mmHg | Increase from Baseline of ≥ 40 mmHg |
| Diastolic blood pressure (mmHg) | Value ≤ 50 mmHg | Value ≥ 110 mmHg |
| | Decrease from Baseline of ≥ 20 mmHg | Increase from Baseline of ≥ 20 mmHg |
| Pulse rate (bpm) | Value ≤ 50 bpm | Value ≥ 110 bpm |
| | Decrease from Baseline of ≥ 30 bpm | Increase from Baseline of ≥ 30 bpm |

Peak supine pulse rate after single dose is defined as the maximum value measured in the first 4 hours post-dose. Peak pulse rate and change from baseline to peak will be summarized similarly to <u>Section 15.2.1.3</u>, including the figure presentations. In addition, hypothesis testing as per <u>Section 15.2.3</u>, will be repeated for these endpoints.

# 16.5. PHYSICAL EXAMINATION

The following summaries will be provided for the full physical examination data, covering major body systems (nose, throat, skin, thyroid gland, neurological system, respiratory system, cardiovascular system, abdomen [liver and spleen], lymph nodes and extremities):

• Incidence of abnormalities at screening

The following summaries will be provided for a brief physical examination to be also performed, on skin, respiratory system, cardiovascular system, and abdomen (liver and spleen):

• Incidence of abnormalities pre-dose.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 16.6. OTHER SAFETY ASSESSMENTS

Chest X-ray and inhalation training results will be presented in a listing only. In addition, screening serum and urine pregnancy test results, as well as pregnancy report data (current pregnancy, pregnancy history and details of the mother), will be listed for women of childbearing potential at Screening.

#### 17. PHARMACOKINETIC EVALUATIONS

PK concentrations are measured at the time of the single dosing and are collected on the Pharmacokinetic Samples eCRF page. Based on this information the PK parameters are then derived. All PK analysis will be carried out by a third party and will not be detailed in this SAP.

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 - Part A

Author: Nicholas Roubinis / Jennifer Allsopp Version Number: Version Date: 13JAN2021

Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


# 18. REFERENCES

Dobson, A. J. (2002). An introduction to generalized linear models, 2nd ed. Chapman & Hall/CRC.

Dmitrienko, A., Bretz, F., Westfall, P. H., Troendle, J., Wiens, B. L., Tamhane, A. C., & Hsu, J. C. (2009). Multiple testing methodology. Multiple Testing Problems in Pharmaceutical Statistics. Chapman and Hall/CRC Press. New York.

Maurer, W., Hothorn, L. A., & Lehmacher, W. (1995). Multiple Comparisons in Drug Clinical Trials and Preclinical Assays: A-priori ordered Hypotheses. Testing Principles in Clinical and Preclinical Trials (J. Vollmar, editor) STuttgart, Gustav Fisher Verlag, 3-18.

SAS Institute, Inc. (1999). SAS Procedures Guide, version 8. Cary, NC: SAS Institute.


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

# **IQVIA OUTPUT CONVENTIONS**

Outputs will be presented according to the following:

### TABLE AND LISTING OUTPUT CONVENTIONS

### General:

- The first row in the body of the table or listing should be blank
- The left-hand column should start in column 1. No indenting or centering of the output should occur.
- Rounding should be done with the SAS function ROUND.
- Numbers in tables should be rounded, not truncated.
- Alphanumeric output should be left aligned.
- Numbers should be decimal point aligned.
- Whole numbers should be right aligned.
- Text values should be left aligned.
- The first letter of a text entry should be capitalized
- Listings of adverse events, concomitant medications, medical histories etc. should be sorted in chronological order, with earliest adverse event, medication or history coming first.
- The study drug should appear first in tables with treatments as columns
- In general, only present totals (across treatment groups) at baseline/randomization, and do not present them post randomization, unless the customer specifically requests it.
- All listing outputs should be sorted (preferably by Treatment, Site Number and Patient Number).
- Exponentiation will be expressed using a superscript with ODS RTF.
- All variables that are output in the CRF (which have data present) should appear in the listings, along with all derived data appearing in the corresponding tables

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018
DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


• The width of the entire output should match the linesize.

#### Univariate Statistics:

- Statistics should be presented in the same order across tables (i.e., n, Mean, SD, Minimum, Median, Maximum and equivalently, n, GeoMean, CV, Minimum, Median, Maximum)
- Table statistics should line up under the N part of the (N=XXX) in the table header. All decimal points should line up. If the minimum and maximum are output on 1 line as Minimum, Maximum then the comma should line up with the decimal point.
- If the original data has N decimal places, then the summary statistics should have the following decimal places: Minimum and maximum: N

Mean, median and CV%: N + 1

SD: N+2

#### Frequencies and percentages (n and %):

• Percent values should be reported inside parentheses, with 1 space between the count and the left parenthesis of the percentage. Parentheses should be justified to accept a maximum of 100.0 as a value and padded with blank space if the percent is less than 100.0. An example is given below:

77 (100.0%)

50 (64.9%)

0 ( 0.0%)

• Percentages will be reported to 1 decimal place, except percentages <100.0% but >99.9% will be presented as '>99.9%' (e.g., 99.99% is presented as >99.9%); and percentages <0.1% will be presented as <0.1%' (e.g., 0.08% is presented as <0.1%). Rounding will be applied after the <0.1% and >99.9% rule.

e.g. ( <0.1%)

(6.8%)

(>99.9%)

Percentages may be reported to 0 decimal places as appropriate (for example, where the denominator is relatively

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

# Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


#### small).

• Where counts are zero, percentages of 0.0% should appear in the output.

#### Confidence Intervals:

- As a rule, confidence intervals are output to 1 place more than the raw data, and standard deviations and standard errors to 2 places more than the raw data
- Confidence intervals should be justified so that parentheses displayed on consecutive lines of a table "line up".
- Boundary values of confidence intervals should be separated by a comma.
- Boundary values should be padded as necessary to accept negative values and to allow alignment of the decimal place.
- An example is given below:

(-0.12, -0.10)

(9.54, 12.91)

#### P-values:

• P-values should be reported to 4 decimal places, except values <1.000 but >0.9999 will be presented as '>0.9999' (e.g., 0.9999 is presented as >0.9999); and values <0.0001 will be presented as '<0.0001' (e.g., 0.00009 is presented as <0.0001). Rounding will be applied after the <0.0001 and >0.9999 rule

#### Ratios

• Ratios should be reported to 1 more decimal place than the original data.

## Spacing:

• There must be a minimum of 1 blank space between columns (preferably 2)

#### Denominators

• If a different count other than the population count is used for a denominator (within the table) to calculate percentages, there should be a row in the table that identifies that number "n".


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018

# Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 453F084F-F7EA-4BA3-B81B-02A299D593C6




Statistical Analysis Plan v2.0 - Part A


• Alternatively, a footnote should be included in each table with percentages to indicate the denominator for percentages.

### Missing values

- A "0" should be used to indicate a zero frequency.
- A blank will be used to indicate missing data in an end-of-text table or patient listing.

## FIGURE OUTPUT CONVENTIONS

- Figures should be provided in RTF files generated by SAS.
- Should contain the title or footer.
- The image should be clear and of high quality when viewed in the Word document, and when printed.
- In general, boxes around the figures should be used.

#### **DATES & TIMES**

Depending on data available, dates and times will take the form DDMMMYYY THH:MM:SS.

## **SPELLING FORMAT**

English US.

## PRESENTATION OF TREATMENT GROUPS

For outputs, treatment groups will be represented as follows and in this order:

| Treatment Group | For Tables, Graphs and Listings |
|----------------------------|---------------------------------|
| RPL554 100 μg double blind | RPL554 100μg |
| RPL554 300 µg double blind | RPL554 300µg |

Document: Z:\ RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v2.0 – Part A


Template No.: CS TP BS016 Revision 5 Reference: CS WI BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


| Treatment Group | For Tables, Graphs and Listings |
|-----------------------------------|---------------------------------|
| RPL554 1000 μg double blind | RPL554 1000μg |
| RPL554 3000 µg double blind | RPL554 3000μg |
| RPL554 6000 µg single blind | RPL554 6000μg |
| Placebo | Placebo |
| Non-randomized (where applicable) | Non-randomized |

## PRESENTATION OF VISITS

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Screening | Scr |
| Day 1 | Day 1 |
| Day 2 | Day 2 |

#### LISTINGS

All listings will be ordered by the following (unless otherwise indicated in the template):

Randomized treatment group (or treatment received if it's a safety output), first by active dose [by ascending dose group] and then placebo.

Center-patient ID,

Date (where applicable),

For listings where non-randomized patients are included, these will appear in a category after the randomized treatment groups labeled 'Non-randomized'.

 $\label{locumentation} \textbf{Document:} \qquad \textbf{Z:} \\ \textbf{RPL554} \\ \textbf{EZAA8488} \\ \textbf{Biostatistics} \\ \textbf{Documentation} \\ \textbf{SAP} \\ \textbf{Verona RPL554-MD-201 SAP v2.0-Part APV v2.0-Part$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


# APPENDIX 2. PARTIAL DATE CONVENTIONS

Imputed dates will NOT be presented in the listings.

## ALGORITHM FOR TREATMENT EMERGENCE OF ADVERSE EVENTS

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| | Partial | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| | Missing | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| Partial, but known | Known | Not TEAE |
| components show that it | | |
| cannot be on or after study | | |
| med start date | | |
| | Partial | Not TEAE |
| | Missing | Not TEAE |
| Partial, could be on or after | Known | If stop date < study med start date, then not TEAE |
| study med start date | | If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month |
| | | if day unknown or 31st December if day and month are |
| | | unknown), then: |
| | | If stop date < study med start date, then not TEAE |


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


| START DATE | STOP DATE | ACTION |
|---|---|---|
| | | If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |
| Missing | Known | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month |
| | | if day unknown or 31st December if day and month are |
| | | unknown), then: |
| | | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |

## ALGORITHM FOR PRIOR / CONCOMITANT MEDICATIONS

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |
| | | If stop date >= study med start date and start date > end of treatment, assign |
| | | as post study |

 $\label{locumentation} \textbf{Document:} \qquad \textbf{Z:} \\ \textbf{RPL554} \\ \textbf{EZAA8488} \\ \textbf{Biostatistics} \\ \textbf{Documentation} \\ \textbf{SAP} \\ \textbf{Verona RPL554-MD-201 SAP v2.0 - Part A representation} \\ \textbf{SAP v2.0 - Part A representation} \\ \textbf{SAP$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


| START DATE | STOP DATE | ACTION |
|---|---|---|
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day |
| | | unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |
| | | If stop date >= study med start date and start date > end of treatment, assign |
| | | as post treatment |
| | Missing | If stop date is missing could never be assumed a prior medication |
| | | If start date <= end of treatment, assign as concomitant |
| | | If start date > end of treatment, assign as post treatment |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month if day |
| | | unknown or 1st January if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |
| | | If stop date >= study med start date and start date > end of treatment, assign |
| | | as post treatment |


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v2.0 - Part A


| START DATE | STOP DATE | ACTION |
|---|---|---|
| | Partial | Impute start date as earliest possible date (i.e. first day of month if day |
| | | unknown or 1st January if day and month are unknown) and impute stop |
| | | date as latest possible date (i.e. last day of month if day unknown or 31st |
| | | December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |
| | | If stop date >= study med start date and start date > end of treatment, assign |
| | | as post treatment |
| | Missing | Impute start date as earliest possible date (i.e. first day of month if day |
| | | unknown or 1st January if day and month are unknown), then: |
| | | If stop date is missing could never be assumed a prior medication |
| | | If start date <= end of treatment, assign as concomitant |
| | | If start date > end of treatment, assign as post treatment |
| Missing | Known | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date, assign as concomitant |
| | | Cannot be assigned as 'post treatment' |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day |
| | | unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date, assign as concomitant |
| | | Cannot be assigned as 'post treatment' |
| | Missing | Assign as concomitant |


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# STATISTICAL ANALYSIS PLAN - PART B

# RPL554-MD-201

A Phase II, Randomized Study to Assess the Pharmacokinetics, Safety and Pharmacodynamics of Single and Repeat Doses of RPL554

Administered by Pressurised Metered Dose Inhaler in Patients with COPD

**AUTHOR:** JENNIFER ALLSOPP

VERSION NUMBER AND DATE: V1.0, 13JAN2021

Document: \(\text{\lector-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201}\)
\(SAP \text{v1.0 - Part B}\)

SAF VI.0 – Falt B

Author: Jennifer Allsopp Version Number: 1.0


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v1.0 - Part B


# STATISTICAL ANALYSIS PLAN – PART B SIGNATURE PAGE

Statistical Analysis Plan V1.0 – Part B (Dated 13JAN2021) for Protocol RPL554-MD-201.

| | Name | Signature | Date |
|---|---|---|---|
| Author: | Jennifer Allsopp | —Docusigned by:<br>Junifer allsopp | 1/19/2021 |
| Position: | Senior Biostatistician | 5E9C02A5CC0A47C | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan – Part B, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Approved By: | Mark Shaw | Docusigned by: Mark Shaw | 1/19/2021 |
| Position: | Associate Director | E2A9CBA2FB8F4B7 | |
| Company: | IQVIA | | |
| Approved By: | Tara Rheault | DocuSigned by: | 1/19/2021 |
| Position: | VP, R&D | C1B201F76799452 | · |
| Company: | Verona Pharma | | |
| Approved By: | Thomas Bengtsson | Docusigned by: Thomas Bengtsson | 1/19/2021 |
| Position: | Statistical Consultant to | 9570C0A2A259423 | |
| Company: | StatMind | | |

 $\begin{tabular}{ll} \begin{tabular}{ll} Document: & \label{tabular} $$ \begin{tabular}{ll} \begin{tabula$ 

Jennifer Allsopp Version Number:


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

# Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# **MODIFICATION HISTORY**

| Unique | Date of the | | |
|---|---|---|---|
| Identifier for | Document | | Significant Changes from |
| this Version | Version | Author | Previous Authorized Version |
| 1.0 | 13JAN2021 | Jennifer Allsopp | Not Applicable – First Version |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v1.0 - Part B


# **TABLE OF CONTENTS**

| 1.<br>2. | INTRODUCTION 9<br>STUDY OBJECTIVES FOR PART B 9 | | |
|---|---|---|---|
| 2.1. | Primary Objective | | 9 |
| 2.2. | Secondary Objectives | | 9 |
| 2.3. | Exploratory Objectives | | 10 |
| 3. | STUDY DESIGN 10 | | |
| 3.1. | General Description | | 10 |
| 3.2. | Schedule of Events | | 11 |
| 3.3. | Changes to Analysis from Protocol | | 11 |
| 4. | PLANNED ANALYSES 11 | | |
| 4.1. | Data Monitoring Committee (DMC) | | 12 |
| 4.2. | Interim Analysis | | 12 |
| 4.3. | Part B Analysis | | 12 |
| 5. | ANALYSIS SETS 13 | | |
| 5.2. | All Patients Randomized Set in Part B [RND] | •••••• | 13 |
| 5.3. | Safety Analysis Set [SAF] | •••••• | 13 |
| 5.4. | Full Analysis Set [FAS] | •••••• | 14 |
| Docum | ment: \\ieedc-vnasc01\\biosdata\\Verona_Pharma\\RPL554\\EZAA8488\\Biostatis SAP v1.0 - Part B | stics\Documentation\SAP\V | erona RPL554-MD-201 |
| Author | Or: Jennifer Allsopp | Version Number: | 1.0 |
| Templa | plate No.: CS_TP_BS016 Revision 5 | Reference: | CS_WI_BS005 |

Effective Date: 01Apr2018




| Stat | stical Analysis Plan V1.0 – Part B | | |
|---|---|---|---|
| | | | - |
| 5.5. | Completers Analysis Set [CAS] | | 14 |
| 5.6. | Pharmacokinetics [PK] Analysis Set | | 14 |
| 6. | GENERAL CONSIDERATIONS 14 | | |
| 6.1. | Reference Start Date and Study Day | | 14 |
| 6.2. | Baseline | ••••• | 15 |
| 6.3. | Repeat/reschedule, Unscheduled Visits and Early Term | ination Data | 15 |
| 6.4. | Windowing Conventions | | 16 |
| 6.5. | Statistical Tests | | 16 |
| 6.6. | Common Calculations | | 16 |
| 6.7. | Software Version | | 17 |
| 7. | STATISTICAL CONSIDERATIONS 18 | | |
| 7.1. | Adjustments for Covariates and Factors to be Included | in Analyses | 18 |
| 7.2. | Multicenter Studies | | 18 |
| 7.3. | Missing data | | 18 |
| 7.4. | Multiple Comparisons/ Multiplicity | | 19 |
| 7.5. | Examination of Subgroups | | 19 |
| 8. | OUTPUT PRESENTATIONS 20 | | |
| 9. | DISPOSITION AND WITHDRAWALS 20 | | |
| 10. | DEMOGRAPHIC AND OTHER SCREENIN | NG CHARACTERIS | TICS 21 |
| 10.1. | Derivations | | 22 |
| Docum | ent: \\ieedc-vnasc01\biosdata\\Verona_Pharma\\RPL554\\EZAA8488\\Bi SAP v1.0 - Part B | ostatistics\Documentation\SAP\V | erona RPL554-MD-201 |
| Author | Jennifer Allsopp | Version Number: | 1.0 |
| | te No.: CS_TP_BS016 Revision 5 | Reference: | CS_WI_BS005 |
| Effectiv | e Date: 01Apr2018 | | |




Statistical Analysis Plan v1.0 - Part B


| 11. SURGICAL, MEDICAL AND CHRONIC OBSTRUCTIVE PULMONARY | |
|---|---|
| DISEASE/SMOKING HISTORY 22 | |
| 12. MEDICATIONS 23 | |
| 13. STUDY MEDICATION EXPOSURE 24 | |
| 14. STUDY MEDICATION COMPLIANCE 25 | |
| 15. EFFICACY OUTCOMES 25 | |
| 15.1. Primary Efficacy | |
| 15.1.1. Primary Efficacy Variable(s) & Derivation(s) | |
| 15.1.2. Missing Data Methods for Primary Efficacy Variable(s) | |
| 15.2. Secondary Efficacy | |
| 15.2.1. Secondary Efficacy Variables & Derivations | 28 |
| 15.2.1.1. Change in baseline in average FEV <sub>1</sub> of AUC <sub>0-4h</sub> (Average FEV <sub>1</sub> over 4 hours), average FEV <sub>1</sub> of AUC <sub>0-12h</sub> (Average FEV <sub>1</sub> over 12 hours) and (morning) trough FEV <sub>1</sub> on Day 7 (Secondary variables 1, 2 and . | 3) |
| 28 | ٠, |
| 15.2.1.2. Change in baseline in peak FEV <sub>1</sub> measured after first dose, average FEV <sub>1</sub> of AUC <sub>0.4h</sub> on Day 1 are | |
| average FEV <sub>1</sub> of AUC <sub>0-12h</sub> FEV <sub>1</sub> on Day 1 (Secondary variables 4, 5 and 6) | |
| 15.2.1.5. Change from baseline in rescue medication use (Secondary variable 9) | 30<br>31 |
| 15.2.3. Analysis of Secondary Efficacy Variables | |
| 15.2.3.1. Analysis of Secondary Variables 1, 2, 3, 4, 5 and 6 | |
| 15.2.3.2. Analysis of Secondary Variable 7 | |
| 15.2.3.3. Analysis of Secondary Variable 8 | |
| 15.2.3.4. Analysis of Secondary Variable 9 | 33 |
| 15.3. Exploratory Efficacy | 33 |
| 15.3.1. Exploratory Efficacy Variables & Derivations | |
| 15.3.1.1. Evaluation of dose response of RPL554 on peak and average FEV1 AUC0-12h after morning dos | |
| on Day 7, and morning trough FEV1 prior to the last dose on Day 7 | 33 |
| 15.3.1.2. Change from baseline in Likert dyspnea scale measured after morning dose on Day 7 | |
| 15.3.2. Missing Data Methods for Exploratory Efficacy Variable(s) | |
| 15.5.5. Milarysis of Exploratory Efficacy Variables | 5-1 |
| 4/ CAPPEN OVERCOMES AA | |
| 16. SAFETY OUTCOMES 34 | |
| 16.1. Adverse Events | 34 |
| | 54 |
| Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B | |
| Template No.: CS_TP_BS016 Revision 5 Reference: CS_WI_BS005 | |
| Effective Date: 01Apr2018 | |
| Copyright © 2009, 2010, 2012, 2016, 2018 IQVIA. All rights reserved. The contents of this document are confidential and propriet to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited. | ary |




Statistical Analysis Plan v1.0 - Part B


| 16.1.1. All TEAEs | 35 |
|---|---|
| 16.1.1.1. Severity | |
| 16.1.1.2. Relationship to Study Medication | |
| 16.1.2. TEAEs Leading to Discontinuation from Study medication | |
| 16.1.3. Serious Adverse Events | |
| 16.1.4. Adverse Events Leading to Death | 30 |
| 16.2. Laboratory Evaluations | |
| 16.2.1. Laboratory Reference Ranges and Markedly Abnormal Criteria | 3′ |
| 16.3. ECG Evaluations | 38 |
| 16.4. Vital Signs | 38 |
| 16.5. Physical Examination | 39 |
| 16.6. Other Safety Assessments | 40 |
| 17. REFERENCES 41 APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS 42 | |
| IQVIA Output Conventions | |
| IQVIA Output Conventions Table and Listing Output Conventions | 42 |
| | 42 |
| Table and Listing Output Conventions | 42 |
| Table and Listing Output Conventions | 42 |
| Table and Listing Output Conventions Figure Output Conventions Dates & Times | |
| Table and Listing Output Conventions Figure Output Conventions Dates & Times Spelling Format | |
| Table and Listing Output Conventions Figure Output Conventions Dates & Times Spelling Format Presentation of Treatment Groups | |
| Table and Listing Output Conventions Figure Output Conventions Dates & Times Spelling Format Presentation of Treatment Groups Presentation of Visits | |

 $SAP\ v1.0-Part\ B$ Author:

Jennifer Allsopp Version Number: 1.0


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

# Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 – Part B


 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy, safety and pharmacokinetic (PK)/pharmacodynamic (PD) data for Part B of protocol RPL554-MD-201. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed. This statistical analysis plan (SAP) is based on the protocol version 3.0, dated 24DEC2019. The study will consist of two parts (A and B) and Part B will be described in this SAP. Only the protocol sections applicable to Part B will be described in this SAP.

### 2. STUDY OBJECTIVES FOR PART B

## 2.1. PRIMARY OBJECTIVE

The primary objective of Part B is to investigate the bronchodilator effect of repeat doses of RPL554 administered by pMDI (pressurized metered dose inhaler), assessed in terms of peak FEV<sub>1</sub> (forced expiratory volume in one second).

## 2.2. SECONDARY OBJECTIVES

The secondary objectives of this part are as follows:

- To investigate the safety and tolerability of repeat doses of RPL554 administered by pMDI.
- To investigate the bronchodilator effect of RPL554 administered by pMDI, in terms of average FEV<sub>1</sub> area under the curve (AUC)<sub>0.4h</sub>, average FEV<sub>1</sub> AUC<sub>0.12h</sub> and trough FEV<sub>1</sub>.
- To determine the onset of action of RPL554 administered by pMDI.
- To evaluate the PK profile of RPL554 administered by pMDI.
- To evaluate the amount of rescue medication use during treatment periods.

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 2.3. EXPLORATORY OBJECTIVES

The exploratory objectives of this part are as follows:

- To assess the dose response of RPL554 on peak and FEV1 AUC<sub>0-12h</sub> after morning dose on Day 7, and morning trough FEV<sub>1</sub> prior to the last dose on Day 7.
- To examine the effect of RPL554 administered by pMDI on a Likert dyspnea scale.

## 3. STUDY DESIGN

# 3.1. GENERAL DESCRIPTION

This is a Phase II, randomized, double-blind, placebo-controlled, two-part study. Part A was a parallel group, single dose assessment of RPL554 administered by pMDI to evaluate the safety and terminal PK profile of a range of doses of RPL554. Five dose levels, 100 µg, 300 µg, 1000 µg, 3000 µg and 6000 µg (single-blind) were selected, covering a 60-fold increase in doses. A total of approximately 36 COPD patients (as defined by the American Thoracic Society [ATS]/European Respiratory Society [ERS] guidelines with symptoms compatible with COPD for at least 1 year prior to Screening) aged 40 to 80 years (inclusive) were randomized at two study centres in the United Kingdom (UK). At the end of Part A, a data cut-off will be used, selected data unblinded and analyzed prior to commencing Part B. Three dose levels, 300 µg, 1000 µg, 3000 µg were selected for Part B, using the same Part A patients. Part B is designed as a complete-block crossover, repeat dose assessment of RPL554 administered by pMDI to evaluate the steady state efficacy/PD effect of the three RPL554 doses compared to the effect with placebo pMDI. The patients in Part B will be expected to complete four treatment periods.

In Part B, the patients from Part A will be randomly assigned in crossover fashion to one of 4 treatment sequences (see <u>Appendix 1</u>; Presentation of Treatment Sequences) each consisting of four 1-week treatment periods separated by a 7 to 10-day washout. Each treatment period consists of 6 days of twice daily doses of RPL554, and a single morning dose on Day 7. In each treatment period, patients will undergo assessments over 12 hours on Days 1 and 7.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 3.2. SCHEDULE OF EVENTS

Schedule of events can be found in Section 6 of the protocol.

## 3.3. CHANGES TO ANALYSIS FROM PROTOCOL

The secondary analysis of change from baseline in rescue medication collected via patient diaries will not be carried out as rescue medication data is only collected during the treatment periods. The rescue medication will be summarized by treatment group for the between visit periods.

An initial formal sample size computation was made for Part B. This was a complete block crossover study. Assuming a residual CV of 6% for peak FEV1, it was estimated that 30 evaluable patients would give an 80% power to detect a pairwise difference in peak FEV1 of 4.6%. Assuming a mean baseline FEV1 of 1.5 L this corresponded to a difference of about 70 mL. To account for withdrawals, 36 patients were to be randomized to Part A. Due to the COVID-19 pandemic, there was a longer than expected period between the completion of Part A and the start of Part B. The long pause made it difficult to re-recruit all patients from Part A and further study conduct with long clinic visits would be more difficult to perform in an ongoing pandemic. It was therefore decided to decrease the patient numbers for Part B to a minimum needed to show efficacy of ensifentrine MDI at doses giving at least 110 mL benefit over placebo on peak FEV1. With 14 fully evaluable patients it was estimated that Part B would have 80% power to fulfill this revised objective.

# 4. PLANNED ANALYSES

There are no data monitoring committee (DMC) or formal interim analyses to be performed for this study. The study will consist of two separate and independent analyses, Part A and Part B. At the end of each part, the database will be locked and unblinded, and the analyses for each part will be performed.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Reference: CS\_WI\_BS005

Template No.: CS\_TP\_BS016 Revision 5 Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 4.1. DATA MONITORING COMMITTEE (DMC)

There will be no DMC analyses for this study.

## 4.2. INTERIM ANALYSIS

No formal interim analysis is planned for the study.

## 4.3. PART B ANALYSIS

All Part B analyses identified in this SAP will be performed by IQVIA Biostatistics following Database Lock on a clean database:

- All outstanding data issues and queries resolved.
- All irresolvable data issues documented in the Data Handling Report (DHR) from Data Management.
- All coding of medications, medical history and adverse events (AEs) completed.
- Serious AE (SAE) reconciliation completed.
- All reconciliation of vendor data with electronic case report form (eCRF) data completed successfully.
- Analysis sets authorized.

It should be noted that the main teams that worked with the Part A analysis remained blinded at the time of the Part A data cut-off, an independent unblinded team performed the Part A unblinded analysis. This was to avoid any potential risk they could trace what study medication a patient might be receiving in Part B (e.g. if they know they experienced certain AEs while on one treatment in Part A and this was identifiable in Part B). Summary data tables for the Part A dose finding analysis were generated. Individual data listings were not provided to the Verona or IQVIA clinical teams to avoid any potential unblinding.

All verbatim text from the eCRF will be presented in outputs "as is" with no "manual hard coding" corrections for such data. Also, PK analysis will be performed by another party (third party vendor), and details of this analysis will not be specified in this SAP.

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 5. ANALYSIS SETS

Agreement and authorization of patients included/excluded from each analysis set will be conducted prior to the unblinding of the study for Part B.

In the case of dosing errors leading to duplication of treatment period or that treatment during period is undetermined, the period data for a patient could be excluded from the analysis. These will be agreed and documented prior to unblinding.

### 5.1. PART A COMPLETERS SET

This set will contain all patients who completed Part A of the study.

# 5.2. ALL PATIENTS RANDOMIZED SET IN PART B [RND]

The all patients randomized (RND) set will contain all patients who completed Part A and who are randomized to study medication in Part B (two randomizations are expected for this study, one for each part). For analyses and displays based on RND, patients will be classified per randomized sequence/treatment.

# 5.3. SAFETY ANALYSIS SET [SAF]

The safety analysis set (SAF) will contain all patients in the RND set who received at least one dose of study medication during Part B. Patients will be classified per actual sequence/treatment received. If there is any doubt whether a patient was treated or not, they will be assumed treated for the purposes of analysis. If a patient is treated based on a non-pre-specified sequence, which is not one of the 4 listed treatment sequence, this will be reported as 'Undefined' for analysis by actual sequence/ treatment per <u>Appendix 1</u>; Presentation of Treatment Sequences. For analysis by treatment group a patient should be counted once for each time a specific treatment was received.

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:




Statistical Analysis Plan v1.0 - Part B


# 5.4. FULL ANALYSIS SET [FAS]

The full analysis set (FAS) will contain all patients in the RND set with sufficient data (pre-dose and at least one post-dose assessment of spirometry) collected after intake of study medication to compute the pharmacodynamic parameters (FEV<sub>1</sub>, FVC measurements) on at least 2 treatment periods in Part B. For analyses and displays based on FAS, patients will be classified per randomized sequence/treatment.

# 5.5. COMPLETERS ANALYSIS SET [CAS]

The completers analysis set (CAS) will contain all patients in the SAF analysis set who complete all treatment periods i.e., a patient who receives a first and last dose intake plus 1 day for all 4 treatment periods per schedule of events (see section 6 of the protocol for schedule details). In the case of dosing errors leading to duplication of treatment period or that treatment during period is undetermined, the patient will be excluded from the completer analysis set. These will be agreed and documented prior to unblinding.

# 5.6. PHARMACOKINETICS [PK] ANALYSIS SET

The PK analysis set will contain all patients in the RND analysis set who have a blood sampling performed after at least one dose of RPL554 in Part B and with data sufficient to calculate PK parameter data. The PK analysis set will be determined by a third-party vendor and the data will be provided to IQVIA.

## 6. GENERAL CONSIDERATIONS

## 6.1. REFERENCE START DATE AND STUDY DAY

Study day will be calculated from the reference start date (treatment period [TP] 1, day 1) and will be used to show start/stop day of assessments and events. Relative day will be calculated from the reference start date (each TP, day 1) and will be used to show start/stop day of assessments and events relative to each treatment period. Reference

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)

Jennifer Allsopp Version Number: 1.


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


start date is defined as the day of the study medication and will appear in every listing where an assessment date or event date appears.

If the date of the event is on or after the reference date, then:

• Study day = (date of event – reference date) + 1.

If the date of the event is prior to the reference date, then:

Study day = (date of event – reference date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, and study day, and any corresponding durations will be presented based on the imputations specified in <a href="Appendix 2">Appendix 2</a>; Partial Date Conventions.

## **6.2.** BASELINE

Baseline definitions are related to the treatment period the patient enters. For majority of endpoints (primary endpoint, relevant secondary/exploratory endpoints and safety endpoints assessed post-dose in the treatment periods), this will be the pre-dose assessment on Day 1 of each treatment period (treatment period 1 to treatment period 4). Baseline for peak FEV<sub>1</sub>, FEV<sub>1</sub> AUC<sub>0-4h</sub>, FEV<sub>1</sub> AUC<sub>0-12h</sub> and morning trough is defined as the average of the FEV<sub>1</sub> pre-dose assessment (-60 minutes and -5 minutes) collected on relevant day of each treatment period. Baseline pre-dose FEV<sub>1</sub>/FVC will be derived from 3 acceptable readings (performed up to 8 times to obtain these), with the highest result from each assessment being used for analysis. For safety assessments with pre-dose assessments, baseline will be defined as the pre-dose assessment for each treatment period.

# 6.3. REPEAT/RESCHEDULE, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the nominal visit will be presented. If a visit is repeated/rescheduled due to variability in FEV<sub>1</sub> or other reason, the repeated/rescheduled visit, will be listed and

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


summarized as the valid visit (same visit number assigned). Unscheduled measurements will not be included in byvisit summaries, but will contribute to the endpoint value. For example, if an unscheduled visit occurred at 10 hours post-dose on Day 1, then this value will be considered in the calculation of the average  $FEV_1$  over 12 hours (AUC<sub>0-12h</sub>  $FEV_1$ ). Any unscheduled or unplanned readings will be presented within the patient listings.

Early termination data will be mapped according to the visit number the termination occurred for by-visit summaries. If termination is between the end of Part A and the beginning of Part B, data are to be considered in the Part B SAP and patient is considered a Part A completer.

Listings will include scheduled, unscheduled, repeat/reschedule and early discontinuation data.

## **6.4.** WINDOWING CONVENTIONS

No visit windows will be applied in this study and the scheduled assessments will be reported and analyzed as per eCRF collection.

## **6.5. STATISTICAL TESTS**

The default significant level will be (5%); confidence intervals will be 95% and all tests will be 2-sided, unless otherwise specified in the description of the analyses. All significant p-values (i.e. < 5%) will be flagged by means of a "\*" for ease of review.

For presentation of summary statistics for quantitative and qualitative variables see <u>Appendix 1</u>; Programming conventions for outputs.

# **6.6. COMMON CALCULATIONS**

Assessments assigned to treatment periods:

Based on the day of assessment relative to the start date of each treatment period as defined by the first

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

# Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


treatment administration for that specific treatment period:

- o Treatment period 1
- o Treatment period 2
- o Treatment period 3
- o Treatment period 4

For quantitative measurements, change from baseline will be calculated as:

• Test value at post-dose timepoint – baseline value.

For quantitative measurement values of FEV1 and FEV1 AUCs will be calculated based on:

- The highest FEV<sub>1</sub> reading from each assessment.
- The baseline value (average of the two pre-dose values [at 1-hour {±5 minutes} and immediately {within 5 minutes}} pre-dose) must be within ± 20% of the pre-albuterol value at Screening; otherwise, the patient will be a screen failure.

Peak effect will be calculated as:

Maximum value in the first 4 hours after dosing.

Average effect will be calculated as:

• FEV<sub>1</sub> AUC divided by the length of the time interval of interest.

Log-transformations will be performed on FEV1 data:

FEV<sub>1</sub> will be analyzed using multiplicative models, which means that data will be logged prior to analysis. The
results will then be back-transformed to linear scale (treatment differences will thus be ratios of geometric
means).

## **6.7. SOFTWARE VERSION**

All analyses will be conducted using SAS version 9.4.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 7. STATISTICAL CONSIDERATIONS

# 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The following covariates are used in the analyses. For details of their inclusion in the models, see the specific analysis section.

- Randomized treatment (fixed).
  - o RPL554 300μg
  - RPL554 1000μg
  - o RPL554 3000μg
  - o Placebo
- Treatment period (fixed).
  - o Treatment period 1
  - o Treatment period 2
  - o Treatment period 3
  - o Treatment period 4
- Baseline value of analyzed variable (covariate).

# 7.2. MULTICENTER STUDIES

This study is being conducted at 2 study centers in the UK.

## 7.3. MISSING DATA

Missing safety data will not be imputed, apart from partial date imputations as specified in <u>Appendix 2</u>. Missing efficacy data will be handled as described in <u>Section 15.1.2</u> and <u>Section 15.2.2</u> of this SAP.

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

Significance of treatment effect will be tested for the primary and secondary efficacy endpoints in Part B and will be done for each of the doses of RPL554 against placebo, starting with the highest dose (3000 µg). To this end, the fixed-sequence testing approach (Maurer et al., 1995; Westfall & Krishen, 2001) will be used.

For the endpoints, let i=0,1,2 and 3 represent increasing dose levels, 0 denoting placebo. Also, let  $\mu_i$ , i=0,1,2 and 3 denote the mean change from baseline for the endpoint of interest for placebo and each increasing active dose level, respectively. The null hypotheses are defined as:  $H_i$ :  $\mu_j - \mu_0 = 0$  and will be tested against the 2-sided alternative  $K_i$ :  $\mu_j - \mu_0 \neq 0$ , j=1,2 and 3.

Finally, let  $p_1$ ,  $p_2$ ,  $p_3$  denote the marginal p-values obtained from the statistical tests associated with  $H_1$ ,  $H_2$ ,  $H_3$  (obtained from the model).

The fixed-sequence testing will begin with the null hypothesis corresponding to the highest dose versus placebo. If a statistically significant difference is found at the 2-sided  $\alpha$  level of 5%, the testing will proceed with the next highest dose. Otherwise, testing stops, and the remaining null hypotheses are considered as failed to reject, without testing.

This testing strategy can be written as the following stepwise algorithm:

- Step 1: If  $p_3 \le \alpha$  reject  $H_3$  and go to Step 2. Otherwise, fail to reject  $H_3$ ,  $H_2$  and  $H_1$  and stop.
- Step 2: If  $p_2 \le \alpha$  reject  $H_2$  and go to Step 3. Otherwise, fail to reject  $H_2$  and  $H_1$  and stop.
- Step 3: If  $p_1 \le \alpha$  reject  $H_1$ . Otherwise, accept  $H_1$ .

The fixed-sequence procedure controls the family-wise error rate in the strong sense because, for each null hypothesis, the testing is conditional upon rejecting all hypotheses earlier in the sequence (Dmitrienko, et al., 2009).

Each secondary endpoint will be tested independently and nominally following a hierarchical testing of doses like the one used for the primary endpoint.

# 7.5. EXAMINATION OF SUBGROUPS

No pre-planned subgroup analyses will be performed for this study.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 - Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 8. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics.

## 9. DISPOSITION AND WITHDRAWALS

All patients who completed Part A of the study will be accounted for in Part B of the study.

Patient disposition, withdrawals and reasons for exclusion from each analysis set will be presented for all patients, summarized by treatment sequence for the patients who completed Part A and were randomized in Part B. Number of patients treated and discontinued in each treatment period will also be presented. If the patient discontinued/withdrew, he/she will be allocated to the last treatment period attended.

All protocol deviations collected in Part B will be divided into critical, major or minor categories and will be assigned to the actual treatment group. The major and critical protocol deviations (PD) will be summarized by treatment and all PDs will be presented in a listing for the RND analysis set. Protocol deviations affect the integrity of the drug activity data and will be obtained by the clinical research associates (CRAs) and documented in the clinical trial management system (CTMS).

Each protocol deviation is categorized into one of the following types, as reported in CTMS:

- 1. Informed Consent Criteria
- 2. Eligibility and Entry Criteria
- 3. Concomitant Medication Criteria
- 4. Laboratory Assessment Criteria
- 5. Study Procedures Criteria
- 6. Serious Adverse Event Criteria
- 7. Randomization Criteria
- 8. Visit Schedule Criteria

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

# Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


- 9. Investigation Product (IP) Compliance
- 10. Efficacy Criteria
- 11. Administrative Criteria
- 12. Source Document Criteria
- 13. Regulatory or Ethics Approvals Criteria
- 14. Other Criteria

Preliminary assignment to each analysis set, therefore whether a patient is included/excluded in each analysis set (excluding the PK analysis set, as this set will be defined later in a separate authorization with input, as required, from the PK scientist) will be recorded in an EXCEL sheet by the IQVIA Biostatistician, with the reason for exclusion from each population indicated. The EXCEL sheet should then be authorized by means of a customer authorization form (CAF) and prior to the Database Lock of the study.

## 10. DEMOGRAPHIC AND OTHER SCREENING CHARACTERISTICS

Demographic data and other screening characteristics (including screening disease characteristics) will be presented for each unique set, as described in Section 5. No statistical testing will be carried out for demographic or other screening characteristics. The following demographic and other screening characteristics will be reported for Part B:

- Age (years)
- Sex
- Childbearing potential
- Race
- Ethnicity
- Height (cm)
- Weight (kg)
- BMI (kg/m<sup>2</sup>)
- Pre (prior to dosing at screening)/post (post dosing at screening) bronchodilator FEV<sub>1</sub> (both in liters and in percentage of predicted normal)
- Post-bronchodilator FEV<sub>1</sub>/FVC

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


- Reversibility test (mL and %)
- · Reversibility assessment performed with four puffs of Albuterol
- Met requirements of reversibility test

## 10.1. DERIVATIONS

Demographic and other screening characteristics recorded on the eCRF will be used as is on the eCRF, without any derivations or adjustments.

# 11. SURGICAL, MEDICAL AND CHRONIC OBSTRUCTIVE PULMONARY DISEASE/SMOKING HISTORY

Surgical and Medical History information will be presented in listings, for the RND analysis set.

- Surgical History will be coded by Medical Dictionary for Regulatory Activities (MedDRA) dictionary using the version specified in the data management plan.
  - o Surgical History conditions are defined as those conditions which stop prior to or at Screening.
  - Data captured on the Surgical Procedure History page of the eCRF will be presented by SOC (System Organ Class) and PT (Preferred Term).
- Medical History will be coded by MedDRA dictionary using the version specified in the data management plan.
  - Medical History conditions are defined as those conditions which stop prior to or at Screening.
  - O Data captured on the Medical History page of the eCRF will be presented by SOC and PT.
- COPD/Smoking History data captured on the COPD and Smoking History page of the eCRF will be presented for each unique set, as described in Section 5.
  - COPD history (Duration of COPD (years) [calculated relative to date of first diagnosis {Randomization date, as recorded in Part A first COPD diagnosis date}/365.25], date of most recent exacerbation, known to have chronic bronchitis/emphysema).
  - Smoking history (current or former smoker, number of packs per day, number of years smoking and number of pack-years [calculated as number of packs per day x number of years smoking])

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 12. MEDICATIONS

Medications will be coded using the World Health Organization – Drug Dictionary (WHO-DD) version specified in the data management plan and will be presented in a listing by Anatomical Therapeutic Chemical (ATC) (the 1st level of the ATC code) and PT for the RND analysis set. Certain medications (or a special grouping of medications) will be classified in a list during the study and signed-off prior to lock by a medical advisor. As this list, may change prior to sign-off they will not be defined in this section of the SAP. Potential medications include, but are not limited to, inhaled corticosteroids (ICS), LAMAs (long-acting muscarinic antagonists), LABAs (long-acting beta2-agonists) etc.

See <u>Appendix 2</u> for handling of partial dates for medications. In the case where it is not possible to define a medication as prior or concomitant, the medication will be classified by the worst case; i.e. concomitant.

- 'Prior' medications are medications which started and stopped in the time between Part A and Part B (prior to the study medication at TP1, Day 1) and have Started prior to start of study medication? = "Yes" on the Concomitant medications eCRF page.
- 'Concomitant' medications are medications which:
  - o Had an onset date on or after the start of study medication for Part B (TP1, Day 1).
  - o AND ended on or after the date of medication or were ongoing at the end of Part B.
  - o A patient can report more than 1 concomitant medication with the same PT.

Prior and concomitant medications will be presented in a listing only, by treatment sequence. For concomitant medications, the treatment period when the medication was taken will also be reported in the listing.

Rescue medications will be recorded on the Rescue Medication/Rescue Medication Inhaler Dispensed/Rescue Medication Inhaler Weight/Rescue Medication Inhaler Collection/Rescue Medication Diary Dispense/Patient Diary for Rescue Medication pages of the eCRF. These are short acting bronchodilators and will be sourced by the study center and dispensed as needed during the Screening, treatment and washout periods. Rescue medication used during the study will be documented on the eCRF pages. Protocol procedures must continue even if rescue medication has been taken. Salbutamol/albuterol is to be used for primary rescue use, but others are also permitted

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Reference: CS\_WI\_BS005

Template No.: CS\_TP\_BS016 Revision 5

Effective Date: 01Apr2018

Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


(e.g. ipratropium). Rescue medications must be withheld for at least 6 hours prior to pre-dose spirometry until completion of the 12-hour post-dose spirometry (per below), and this is to be confirmed in the eCRF at the start of each treatment period. If this withhold is not met, the patient should be rescheduled for a repeat visit within permitted windows.

Rescue medications used during study visits in Part B will be primarily provided by patients on paper diaries, which will be transcribed into the eCRF. In the event of missing or incomplete diaries, rescue medication will be determined analytically (by recording the weight of the canister dispensed at the end of Day 1 and start of Day 7 per period). Rescue medication analysis will be described in Section 15.2.1.5.

When a rescue medication is used less than 6 hours prior to study medication a sensitivity analysis will be carried out for the  $AUC_{0-12h}FEV_1$  analysis detailed in Section 15.2.1.1 and 15.2.1.2 which will remove patients from the treatment periods where rescue medication was taken less than 6 hours prior to study medication or patients who took rescue medication during the 12 hour assessments. This will only be carried out if at least 1 patient has taken rescue medication less than 6-hours prior to study medications.

## 13. STUDY MEDICATION EXPOSURE

Exposure to study medication in days will be presented by treatment for the SAF analysis set. The date of first study medication inhalation, per treatment, will be taken from the Drug Exposure eCRF page for treatment period 1. The date of last study medication inhalation, per treatment sequence, will also be taken from the Drug Exposure eCRF page, based on the last end time of inhalation for the last treatment period of a patient.

Drug accountability i.e. the number of pMDIs used per treatment period, as measured on the Drug Exposure eCRF page will be summed to get the total number of pMDIs used and presented similarly to exposure, by treatment sequence for the SAF analysis set.

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


# 13.1. DERIVATIONS

- Duration of exposure per treatment period (days) in Part B = date of last study medication administration, per treatment – date of first study medication administration, per treatment +1.
- Duration of exposure per treatment sequence (days) in Part B = Duration of exposure for period 1 + Duration of exposure for period 2 + Duration of exposure for period 3 + Duration of exposure for period 4.
- Drug accountability (number of capsules) = Number of pMDIs dispensed number of pMDIs returned by treatment period.

### 14. STUDY MEDICATION COMPLIANCE

In Part B, patients will be dosed at the study center on the morning and evening of Day 1 and on the morning of Day 7. Patients will self-administer study medication for the other dosing times (i.e. on Days 2 through 6). Compliance will be assessed by recording the number of pMDIs dispensed and returned, as per drug accountability described in Section 13.

# 15. EFFICACY OUTCOMES

The primary efficacy analyses will be performed for the FAS. Patients withdrawn after only one treatment period will not be included in the analyses of the primary efficacy variable. If the CAS differs from the FAS, the primary efficacy analysis will also be carried out on the CAS.

#### 15.1. PRIMARY EFFICACY

## 15.1.1. PRIMARY EFFICACY VARIABLE(S) & DERIVATION(S)

The primary efficacy variable is peak  $FEV_1$  (measured in first 4 hours after morning dosing). This will be measured after dosing on Day 7 and is collected on the Spirometry Study measurements eCRF page. The primary efficacy endpoint is change from baseline in peak  $FEV_1$ .

Document: \\ieedc-vnasc01\biosdata\\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\\Verona\_RPL554-MD-201

SAP v1.0 – Part B

Jennifer Allsopp

Version Number:


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:




Statistical Analysis Plan v1.0 - Part B


Three acceptable readings are performed at each of the timepoints in first 4 hours after morning dosing on Day 7 (5, 15 and 30 minutes and 1, 1.5, 2 and 4 hours) and the highest of the 3 is used for analysis purposes. Hence, peak  $FEV_1$  is derived as the highest of all these readings. Patients withdrawn after only one treatment period will not be included in the analysis.

Descriptive statistics (see Appendix 1 [Programming conventions for outputs]) for  $FEV_1$  will be presented for all patients assigned to FAS, at each assessment and change from baseline at each assessment. All summaries will be presented for each treatment group by day and timepoint. In addition, a figure (bar graph) representing mean change from baseline  $FEV_1$  to peak  $FEV_1$  by treatment will be presented, including the standard error of the mean.

Change from baseline  $FEV_1$  to peak  $FEV_1$  (over 4 hours) at Day 7 will be derived to test the hypothesis described in section 15.1.3 with baseline defined as the average of the  $FEV_1$  pre-dose assessment (-60 minutes and -5 minutes) collected on Day 1 of each treatment period. Peak  $FEV_1$  at Day 7 is defined as the maximum post-dose value among the 5, 15, 30 minutes, 1, 1.5, 2 and 4-hour assessments collected at after morning dose on Day 7 of each treatment period.

#### 15.1.2. MISSING DATA METHODS FOR PRIMARY EFFICACY VARIABLE(S)

No imputation will be applied.

#### 15.1.3. PRIMARY ANALYSIS OF PRIMARY EFFICACY VARIABLE(S)

The primary efficacy objective of the study is to show that at least 1 RPL554 treatment group (RPL554 3000 $\mu$ g, RPL554 1000 $\mu$ g, RPL554 300 $\mu$ g) will increase peak FEV<sub>1</sub> (change from Baseline) compared to placebo at Day 7 (measured in first 4 hours after morning dosing) by rejecting the null hypothesis described below at significance level  $\alpha$ =0.05 level (2-sided):

 $H_0$ :  $\mu_j = \mu_0$  versus  $H_1$ :  $\mu_j \neq \mu_0$ 

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


where  $\mu_j$  and  $\mu_0$  are the mean change from Baseline in peak FEV<sub>1</sub> at Day 7 (measured in first 4 hours after morning dosing) for 1 RPL554 treatment group (RPL554 3000 $\mu$ g, RPL554 1000 $\mu$ g, RPL554 3000 $\mu$ g) and placebo respectively.

An ANCOVA will be used to test the hypothesis with change from baseline  $FEV_1$  to peak  $FEV_1$  (measured in first 4 hours after morning dosing) on Day 7 as response variable, and treatment and treatment period as fixed factors, patient as random and baseline  $FEV_1$  as covariates. Analyses will be implemented using the SAS® procedure MIXED as follows:

```
PROC MIXED DATA = ...;

CLASS USUBJID PERIOD TREATMENT;

MODEL CHG = TREATMENT PERIOD BASELINE;

RANDOM USUBJID;

LSMEANS TREATMENT / CL DIFF;

RUN;

where CHG = difference in log (peak FEV<sub>1</sub> - baseline FEV<sub>1</sub>)

TREATMENT = treatment group (RPL554 3000μg, RPL554 1000μg, RPL554 300μg, and placebo)

PERIOD = treatment period (treatment period 1, 2, 3, and 4)

BASELINE = log (baseline FEV<sub>1</sub>)

USUBJID = subject ID
```

The primary comparison will be the contrast (difference in least squares mean [LSMEAN]) between RPL554 3000µg and placebo on Day 7 (in first 4 hours after morning dosing).

Peak  $FEV_1$  and the covariate, baseline  $FEV_1$ , will be log-transformed prior to analysis using natural logarithm. The difference between the two is log (peak  $FEV_1$ ) – log (baseline  $FEV_1$ ). Therefore, the LSMEAN statement between treatments in the above PROC MIXED will provide the log of the contrasts. Prior to presentations, the antilog of these point estimates and associated 95% confidence intervals will be performed, giving ratios of geometric means on the linear scale. The 2-sided p-value for the exponential (exp) least squares mean, exp(LSM), ratio between each of the 2 treatment groups and placebo will be reported.

Summary statistics for FEV<sub>1</sub> will be presented for baseline, peak on Day 7 (in first 4 hours after morning dosing)

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


and change from baseline to peak by treatment group on patients with both assessments, on the original scale. A figure displaying the mean change from baseline FEV<sub>1</sub> over time by treatment and day will also be presented.

## 15.2. SECONDARY EFFICACY

The secondary efficacy analyses will be performed for the FAS. Patients withdrawn after only one treatment period will not be included in the analyses of any of the secondary efficacy variables.

#### 15.2.1. SECONDARY EFFICACY VARIABLES & DERIVATIONS

15.2.1.1. Change in baseline in average FEV<sub>1</sub> of AUC<sub>0-4h</sub> (Average FEV<sub>1</sub> over 4 hours), average FEV<sub>1</sub> of AUC<sub>0-12h</sub> (Average FEV<sub>1</sub> over 12 hours) and (morning) trough FEV<sub>1</sub> on Day 7 (Secondary variables 1, 2 and 3)

Average  $FEV_1$  is defined as the  $AUC_{0-4h}FEV_1$ , divided by the length of the time (in hours).  $AUC_{0-4h}FEV_1$  is derived using the following formula:

$$AUC = \frac{1}{2}(t_1 - t_0)(y_1 + y_0) + \frac{1}{2}(t_2 - t_1)(y_2 + y_1) + \dots + \frac{1}{2}(t_i - t_{i-1})(y_i + y_{i+1})$$

where i are the number of intervals,  $t_i$  are the time values or time intervals (in actual hours) between assessments and  $y_i$  the FEV $_1$  values (highest of the three acceptable readings) at  $t_i$ . The AUC result will then be divided by the actual time (the time elapsed since dosing, until the time of assessment) at 4-hour assessment (as this can occur  $\pm$  10 minutes) to obtain the average FEV $_1$ . If the assessment at 4-hour is missing, the AUC result will be divided by the actual time of the last collected assessment. For analysis purposes, it will be assumed that the pre-dose value (immediately pre-dose) occurred at time 0 when computing PD parameters. If a patient misses hour 2 and 4 then the AUC $_{0.4}$  is set to missing.

Descriptive statistics (see <u>Appendix 1</u> [Programming conventions for outputs]) for AUC<sub>0-4</sub> will be presented for all patients assigned to FAS, at each assessment and change from baseline at each assessment as relevant. All summaries will be presented for each treatment group.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B

Jennifer Allsopp Version Number: 1.0


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


Change from baseline  $FEV_1$  to  $FEV_1$  AUC<sub>0-4</sub> will be derived to test the hypothesis described in <u>Section 15.2.3</u> with baseline defined as the average of the  $FEV_1$  pre-dose assessments (-60 minutes and -5 minutes) collected.

 $AUC_{0-12h}$  FEV<sub>1</sub> is defined and derived similarly to  $AUC_{0-4h}$  above, but over 12-hours post-dose. If patient misses hours 11 and 12 then the  $AUC_{0-12h}$  is set to missing. If the assessment at 12-hours is missing, the AUC result will be divided by the actual time of the last collected assessment.

Morning trough  $FEV_1$  is the average of the  $FEV_1$  pre-dose assessments (-60 minutes and -5 minutes) on Day 7 and the change from baseline will be analyzed similarly to  $AUC_{0.4h}$  and  $AUC_{0.12h}$ .

### 15.2.1.2. Change in baseline in peak FEV<sub>1</sub> measured after first dose, average FEV<sub>1</sub> of AUC<sub>0-4h</sub> on Day 1 and average FEV<sub>1</sub> of AUC<sub>0-12h</sub> FEV<sub>1</sub> on Day 1 (Secondary variables 4, 5 and 6)

Peak  $FEV_1$  measured after first dose is defined as the peak  $FEV_1$  (after 4 hours of dosing) on Day 1. It is defined as the change from baseline to peak  $FEV_1$  and derived similarly to primary analysis (see <u>section 15.1.1</u>), but instead at Day 1.

 $AUC_{0.4h}$  FEV<sub>1</sub> and  $AUC_{0.12h}$  FEV<sub>1</sub> on Day 1 are defined and derived similarly to secondary endpoint above (see section 15.2.1.1), but at Day 1. Parameters will be calculated over 4 and 12 hours, respectively (on Day 1 of each treatment period). If patient misses hours 2 and 4 then the  $AUC_{0.4h}$  is set to missing. Similarly, if patient misses hours 11 and 12 then the  $AUC_{0.12h}$  is set to missing. If the assessment at 12-hours is missing, the AUC result will be divided by the actual time of the last collected assessment.

### 15.2.1.3. Determination of onset of action (>10% increase in FEV<sub>1</sub>, from pre-first dose, censored at 120 minutes) on Day 1 (Secondary variable 7)

Onset of action is defined as a >10% increase in FEV<sub>1</sub> from pre-dose on Day 1 over the next 120 minutes (2 hours) after morning dosing on Day 1 (5, 15 and 30 minutes and 1, 1.5, 2 hours). Time to onset will be derived as the time to onset of action is achieved. For analysis purposes, it will be assumed that the pre-dose value occurred at time 0. Patients not experiencing an onset of action will be censored at 120 minutes (2 hours) or at time of premature

Document: \(\text{\lector-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201}\)
\(SAP \text{v1.0 - Part B}\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


discontinuation (if withdrawn before 120 minutes). If the number of patients censored regarding onset of action is deemed to be too high (number of patients with onset of action censored >50%), the Kaplan-Meier estimates and accompanying figure will not be presented. Patients receiving placebo will not be summarized in either tables or figure.

### 15.2.1.4. RPL554 steady state pharmacokinetics (AUC $_{0-12h}$ , Cmax, time to maximum concentration [tmax]) (Secondary variable 8)

Concentration of RPL554 and computed PK parameters (AUC<sub>0-12h</sub>,  $C_{max}$  [maximum concentration],  $t_{max}$  [time to maximum concentration]) on Day 7 of each treatment period (pre-dose, 30 minutes and 1, 1.5, 2, 4, 8 and 12-hours post dose).

### 15.2.1.5. Rescue medication use during treatment periods (Secondary variable 9)

Use of medication per treatment period is calculated as the mean use daily over the treatment period, (Day 1 to Day 7) calculated only based on the days data was recorded/verified in the patient diary for rescue mediation.

If less than 4 days of data are available for the treatment period, the weekly mean is set to missing, e.g. if data is entered for less than 4 days between Day 1 and Day 7 then no result will be presented for that treatment period.

This will be documented in the "Rescue Medication Diary Dispense" page of the eCRF, as well as in the "Patient Diary for Rescue Medication" entry.

The rescue medication use will be confirmed in the diary using the following rules:

- 1. If patient has put in rescue medication use then analyse as expected.
- 2. If patient has not put in rescue medication use, then to confirm that there was no diary compliance issue, question "Rescue medication taken?" will be answered "No" to make sure it is filled in correctly.
- 3. If patient has not put in rescue medication use and question "Rescue medication taken?" was not filled in correctly then this will be treated as diary compliance issue and therefore this day will not be used as the day recorded for the weekly means calculation.

Rescue medication use, in terms of weight (mcg) of rescue medication during the treatment periods will be collected from the Rescue Medication Inhaler Dispensed, Rescue Medication Inhaler Collected and Rescue Medication

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


Inhaler Weight eCRF pages and will be summarized by treatment group in a listing.

### 15.2.2. MISSING DATA METHODS FOR SECONDARY EFFICACY VARIABLE(S)

No imputation will be applied.

### 15.2.3. ANALYSIS OF SECONDARY EFFICACY VARIABLES

### 15.2.3.1. Analysis of Secondary Variables 1, 2, 3, 4, 5 and 6

The secondary variables listed above will be analyzed by comparing the RPL554 treatment groups to each other and placebo by rejecting the null hypothesis described below at significance level  $\alpha$ =0.05 level (2-sided):

$$H_0\!\colon \mu_j\!=\mu_0 \text{ versus } H_1\!\colon \mu_j\!\neq\mu_0$$

where  $\mu_j$  and  $\mu_0$  are the mean change from Baseline for each parameter for each respective dose of RPL554 and placebo.

ANCOVA analyses will be implemented using the SAS® procedure MIXED as follows:

```
PROC MIXED DATA = ...;

CLASS USUBJID PERIOD TREATMENT;

MODEL CHG = TREATMENT PERIOD BASELINE;

LSMEANS TREATMENT / CL DIFF;

RANDOM USUBJID;

RUN;

where CHG = difference in log (parameter – baseline parameter)

TREATMENT = treatment group (Respective dose of RPL554, 300µg, 1000µg and 3000µg and placebo)

PERIOD = treatment period (treatment period 1, 2, 3, and 4)

BASELINE = log (baseline parameter)

USUBJID = subject ID
```

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


The primary comparison will be the contrast (difference in least squares mean [LSMEAN]) between 3000µg RPL554 and placebo using hierarchical testing. The parameter value and its baseline covariate will be log-transformed prior to analysis using natural logarithm. The difference between the two log (parameter) – log (baseline parameter). Therefore, the LSMEAN statement between treatments in the above PROC MIXED will provide the log of the contrasts. Prior to presentations, the antilog of these point estimates and associated 95% confidence intervals will be performed, giving ratios of geometric means on the linear scale. The 2-sided p-value for the exponential (exp)least squares mean, exp(LSM), ratio between each of the 2 treatment groups and placebo will be reported.

Summary statistics for each parameter will be presented for baseline, at point of interest (if applicable) and change from baseline by treatment group on patients with both assessments, on the original scale.

### 15.2.3.2. Analysis of Secondary Variable 7

Onset of action will be summarized by treatment and a Kaplan-Meier plot illustrating time to onset constructed. The SAS® procedure LIFETEST, will be used as follows to calculate the median, 25<sup>th</sup> and 75<sup>th</sup> percentile:

```
PROC LIFETEST DATA=... OUTSURV =... CONFTYPE = LINEAR METHOD =

KM ALPHA = 0.05 ALPHAQT = 0.05 PLOTS = (SURVIVAL (FAILURE NOCENSOR));

TIME ONSET*STATUS (1);

STRATA TREATMENT;

RUN;

where ONSET = time to onset of action

TREATMENT = treatment group (Respective dose of RPL554, 300μg, 1000μg and 3000μg)

STATUS (1) = indicates an event of onset of action
```

To calculate the mean difference to RPL554  $3000\mu g$ , the SAS procedure LIFETEST will be carried for each treatment comparison pair individually.

If a patient does not have onset of action from pre-dose on Day 1 over the next 120 minutes (2 hours) the data will be censored at 120 minutes or if a patient prematurely discontinued before 120 minutes, the last available

Document: \\ieedc-vnasc01\biosdata\\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


assessment time post-dose (1 indicates censored variables). Median differences to the highest dose (RPL554 3000  $\mu$ g) will be estimated and the p-value based on the PROC LIFETEST above (Wilcoxon signed rank sum test) between each treatment groups and the highest dose will also be presented.

### 15.2.3.3. Analysis of Secondary Variable 8

As described in <u>section 4.3</u>, this SAP will not summarise the analyses related to the PK concentrations and parameters and this will be handled by a third-party vendor.

### 15.2.3.4. Analysis of Secondary Variable 9

Summary statistics will be presented by treatment group. In addition, all rescue medication used during the serial spirometry assessments (Days 1 and 7) will be listed to assess the accuracy of the  $FEV_1$  recordings.

### 15.3. EXPLORATORY EFFICACY

### 15.3.1. EXPLORATORY EFFICACY VARIABLES & DERIVATIONS

### 15.3.1.1. Evaluation of dose response of RPL554 on peak and average FEV1 AUC0-12h after morning dose on Day 7, and morning trough FEV1 prior to the last dose on Day 7

The association of dose response for the primary and secondary endpoints listed in this section title will be performed by pairwise comparisons of RPL554 doses (ie,  $1000\mu g$  vs  $300\mu g$ , and  $3000\mu g$  vs  $1000\mu g$ ) using ANCOVA models in the same ways as the primary endpoint detailed in Section 15.1.3.

### 15.3.1.2. Change from baseline in Likert dyspnea scale measured after morning dose on Day 7

An 11-point Likert scale will be utilized, with patients being asked the following question by a blinded member of staff: "On a scale of zero to ten, please rate your current shortness of breath, with zero indicating no shortness of breath and ten indicating the worst shortness of breath that you can imagine". This scale will be an instantaneous

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


measurement of their dyspnea at that moment, and not reflective. It will be administered on Day 7 pre-dose and 30 minutes, 1, 1.5, 2, 4, 8, 11 and 12 hours post-dose of each treatment period. Baseline will be considered the pre-dose assessment on Day 1 of each treatment period and change from baseline will be assessed at each timepoint on Day 1 and Day 7.

### 15.3.2. MISSING DATA METHODS FOR EXPLORATORY EFFICACY VARIABLE(S)

No imputation will be applied.

### 15.3.3. ANALYSIS OF EXPLORATORY EFFICACY VARIABLES

Dyspnea score and the change in dyspnea score will be summarized at each timepoint of interest on Day 7 (pre-dose and 30 minutes, 1, 1.5, 2, 4, 8, 11 and 12 hours post-dose). Treatment comparisons of change from baseline will be performed using an ANCOVA adjusting for treatment, treatment period and patient, and using pre-dose Day 1 baseline value as a covariate, like the hypothesis described in section 15.1.3. The model will be additive; therefore no log-transformation will be applied.

### **SAFETY OUTCOMES** 16.

All outputs for safety outcomes will be based on the SAF.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified with the relevant section.

### 16.1. ADVERSE EVENTS

Adverse Events (AEs) will be coded by MedDRA dictionary using the version specified in the data management plan.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the

Document:

SAP v1.0 - Part B Jennifer Allsopp


Version Number:

Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


first dose of study medication in Part B, based on the investigator assessment of severity. TEAEs will be assigned to treatment groups based on actual treatment received. TEAEs, like medications, may be assigned to multiple treatment groups due to the cross-over design of the study. This will depend on the occurrence date and duration of each TEAE.

See Appendix 2 for handling of partial dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, the AE will be classified by the worst case; i.e. treatment emergent.

An overall summary of number of patients within each of the categories described in the sub-section below, will be provided as specified in the templates.

Listings will include TEAEs and Non-TEAEs.

### **16.1.1. ALL TEAES**

Incidence of TEAEs will be presented by System Organ Class (SOC) and Preferred Term (PT) and broken down further by maximum severity and relationship to study medication.

### 16.1.1.1. Severity

Severity is classed as mild/ moderate/ severe (increasing severity). TEAEs starting after the first dose of study medication with a missing severity will be classified as severe. If a patient reports a TEAE more than once within that SOC/ PT, the AE with the worst-case severity will be used in the corresponding severity summaries.

### 16.1.1.2. Relationship to Study Medication

Relationship, as indicated by the Investigator, is classed as "yes" or "no". A related TEAE is defined as a TEAE with a relationship to study medication as "yes". TEAEs with a missing relationship to study medication will be regarded as relationship = "yes" to study medication. If a patient reports the same AE more than once within that SOC/ PT, the AE with the worst-case relationship to study medication will be used in the corresponding relationship summaries.

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


### 16.1.2. TEAES LEADING TO DISCONTINUATION FROM STUDY

TEAEs leading to discontinuation from the study will be identified by using the question "Did the AE cause the Patient to discontinue from the study?" from the AE page of the eCRF.

For TEAEs leading to discontinuation from the study, summaries of incidence rates (frequencies and percentages) by SOC and PT will be prepared.

### 16.1.3. SERIOUS ADVERSE EVENTS

Serious adverse events (SAEs) are those events recorded as "Serious" on the Adverse Events page of the eCRF. A summary of serious TEAEs by SOC and PT will be prepared, similarly to <u>Section 16.1.1</u> and <u>Section 16.1.2</u>.

### 16.1.4. ADVERSE EVENTS LEADING TO DEATH

TEAEs leading to Death are those events which are recorded as "Death" on the Adverse Events page of the eCRF. A summary of TEAEs leading to death by SOC and PT will be prepared.

### 16.2. LABORATORY EVALUATIONS

Results from the local laboratory will be included in the reporting of this study for hematology, blood chemistry, and urinalysis. A list of laboratory assessments to be included in the outputs is included in the protocol, Sections 7.4.3.1, 7.4.3.2, and 7.4.3.3 for hematology, blood chemistry, and urinalysis, respectively. Presentations will use International system (SI) units.

Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of quantification (BLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

The following summaries will be provided for laboratory data:

Actual and change from baseline (pre-dose at Day 1 for each treatment period) to each pre-dose time point at
 Day 7 (for quantitative measurements), including overall (where overall is regardless of treatment period, day

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:




Statistical Analysis Plan v1.0 - Part B


and timepoint to assess treatment group, as a whole).

- Shift from baseline based on normal range criteria (for quantitative measurements and categorical measurements)
- Incidence of abnormal values according to normal range criteria (in the case of Biochemistry only).
- Listing of all abnormal values occurring after the first dose of study medication.

### 16.2.1. LABORATORY REFERENCE RANGES AND MARKEDLY ABNORMAL CRITERIA

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

In addition to the high and low quantitative laboratory assignments (as identified by means of the laboratory reference ranges), markedly abnormal quantitative blood chemistry values per the table below will also be identified by the Investigator.

| | Blood Chemistry – |
|----------------------------------|------------------------------|
| | Markedly Abnormal Definition |
| Alanine Aminotransferase (ALT) | > 3 x ULN |
| Alkaline Phosphatase (ALP) | > 3 x ULN |
| Aspartate Aminotransferase (AST) | > 3 x ULN |
| Creatinine | > 221 μmol/L |
| Gamma Glutamyl Transferase (GGT) | > 3 x ULN |
| Bilirubin (TBL) | > 3 x ULN |

ULN: Upper limit of normal.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


### 16.3. ECG EVALUATIONS

Overall results from the local ECG lab will be included in the reporting of this study. The overall assessment of ECG parameters will be reported for this study:

- Normal
- Abnormal not Clinically Significant (ANCS)
- Abnormal Clinically Significant (ACS)
- Incomplete Analysis
- Uninterpretable

The following summaries will be provided for quantitative ECG data, for example heart rate:

- Actual assessments at baseline (pre-dose at Day 1 for each treatment period) and each pre-dose time point at
  Day 7, including overall (where overall is regardless of treatment period, day and timepoint to assess treatment
  group as a whole).
  - Shift of overall assessment baseline to post-dose timepoints per Normal, ANCS and ACS overall
    assessment criteria.
  - Listing of all ECG evaluations and abnormal values occurring after the first dose of study medication.

### 16.4. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Supine Systolic Blood Pressure (mmHg)
- Supine Diastolic Blood Pressure (mmHg)
- Supine Pulse Rate (bpm)

The following summaries will be provided for vital signs data:

 Actual assessments at screening, baseline (pre-dose at each treatment period) and each post-dose time points, including end of study visit and overall (where overall is regardless of treatment period, day and timepoint to

Document: \(\text{\lector-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201}\)
\(SAP \text{v1.0 - Part B}\)

Jennifer Allsopp

Version Number: 1.0

Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:




Statistical Analysis Plan v1.0 - Part B


assess treatment group as a whole).

• Incidence of markedly abnormal values (number and percent) based on the criteria presented in the table below:

| | Low | High |
|---|---|---|
| Systolic blood pressure (mmHg) | Value ≤ 90 mmHg | Value ≥ 180 mmHg |
| | Decrease from Baseline of ≥ 40 mmHg | Increase from Baseline of ≥ 40 mmHg |
| Diastolic blood pressure (mmHg) | Value ≤ 50 mmHg | Value ≥ 110 mmHg |
| | Decrease from Baseline of ≥ 20 mmHg | Increase from Baseline of ≥ 20 mmHg |
| Pulse rate (bpm) | Value ≤ 50 bpm | Value ≥ 110 bpm |
| | Decrease from Baseline of ≥ 30 bpm | Increase from Baseline of ≥ 30 bpm |

Peak supine pulse rate after study medication is defined as the maximum value measured in the first 4 hours post-dose. Peak pulse rate and change from baseline to peak on Day 1 and after morning dosing on Day 7 will be summarized similarly to Section 15.1.3, including the figure presentation described in the same section. Treatment comparisons of change from baseline will be performed using an ANCOVA adjusting for treatment, treatment period and patient, and using pre-dose pulse rate as a covariate, like the hypothesis described in Section 15.1.3. The model will be additive; therefore no log-transformation will be applied.

### 16.5. PHYSICAL EXAMINATION

The following summaries will be provided for the full physical examination data, covering major body systems (nose, throat, skin, thyroid gland, neurological system, respiratory system, cardiovascular system, abdomen [liver and spleen], lymph nodes and extremities):

- Incidence of abnormalities at end of study visit (4-10 days after last treatment period).
- Shifts from baseline at end of study visit.

The following summaries will be provided for a brief physical examination to be also performed, on skin,

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


respiratory system, cardiovascular system, and abdomen (liver and spleen):

- Incidence of abnormalities pre-dose on Day 1 and 7 by treatment period.
- Shifts from baseline by treatment period and timepoint.

### 16.6. OTHER SAFETY ASSESSMENTS

Inhalation training results on Day 1 pre-dose will be presented in a listing only. In addition, urine pregnancy test results will be listed for women of childbearing potential at Day 1 pre-dose and end of study visits.

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


### 17. REFERENCES

Dobson, A. J. (2002). An introduction to generalized linear models, 2nd ed. Chapman & Hall/CRC.

Dmitrienko, A., Bretz, F., Westfall, P. H., Troendle, J., Wiens, B. L., Tamhane, A. C., & Hsu, J. C. (2009). Multiple testing methodology. Multiple Testing Problems in Pharmaceutical Statistics. Chapman and Hall/CRC Press, New York.

Maurer, W., Hothorn, L. A., & Lehmacher, W. (1995). Multiple Comparisons in Drug Clinical Trials and Preclinical Assays: A-priori ordered Hypotheses. Testing Principles in Clinical and Preclinical Trials (J. Vollmar, editor) STuttgart, Gustav Fisher Verlag, 3-18.

SAS Institute, Inc. (1999). SAS Procedures Guide, version 8. Cary, NC: SAS Institute.

Document: \\ieedc-vnasc01\biosdata\\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v1.0 - Part B


### **APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS**

### **IQVIA OUTPUT CONVENTIONS**

Outputs will be presented according to the following:

### TABLE AND LISTING OUTPUT CONVENTIONS

### General:

- The first row in the body of the table or listing should be blank
- The left-hand column should start in column 1. No indenting or centering of the output should occur.
- Rounding should be done with the SAS function ROUND.
- Numbers in tables should be rounded, not truncated.
- Alphanumeric output should be left aligned.
- Numbers should be decimal point aligned.
- Whole numbers should be right aligned.
- Text values should be left aligned.
- The first letter of a text entry should be capitalized
- Listings of adverse events, concomitant medications, medical histories etc. should be sorted in chronological order, with earliest adverse event, medication or history coming first.
- The study drug should appear first in tables with treatments as columns
- In general, only present totals (across treatment groups) at baseline/randomization, and do not present them post randomization, unless the customer specifically requests it.
- All listing outputs should be sorted (preferably by Treatment, Site Number and Patient Number).
- Exponentiation will be expressed using a superscript with ODS RTF.
- All variables that are output in the CRF (which have data present) should appear in the listings, along with all derived data appearing in the corresponding tables
- The width of the entire output should match the line size.

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)

Jennifer Allsopp Version Number: 1


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


### Univariate Statistics:

- Statistics should be presented in the same order across tables (i.e., n, Mean, SD, Minimum, Median, Maximum and equivalently, n, GeoMean, CV, Minimum, Median, Maximum)
- Table statistics should line up under the N part of the (N=XXX) in the table header. All decimal points should line up. If the minimum and maximum are output on 1 line as Minimum, Maximum then the comma should line up with the decimal point.
- If the original data has N decimal places, then the summary statistics should have the following decimal places: Minimum and maximum: N

Mean, median and CV%: N + 1

SD: N+2

Frequencies and percentages (n and %):

• Percent values should be reported inside parentheses, with 1 space between the count and the left parenthesis of the percentage. Parentheses should be justified to accept a maximum of 100.0 as a value and padded with blank space if the percent is less than 100.0. An example is given below:

77 (100.0%)

50 (64.9%)

0 (0.0%)

• Percentages will be reported to 1 decimal place, except percentages <100.0% but >99.9% will be presented as <99.9%' (e.g., 99.99% is presented as >99.9%); and percentages <0.1% will be presented as <0.1%' (e.g., 0.08% is presented as <0.1%). Rounding will be applied after the <0.1% and >99.9% rule.

e.g. ( <0.1%)

(6.8%)

(>99.9%)

Percentages may be reported to 0 decimal places as appropriate (for example, where the denominator is relatively small).

 $\bullet$  Where counts are zero, percentages of 0.0% should appear in the output.

### Confidence Intervals:

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018


DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


- As a rule, confidence intervals are output to 1 place more than the raw data, and standard deviations and standard errors to 2 places more than the raw data
- Confidence intervals should be justified so that parentheses displayed on consecutive lines of a table "line up".
- Boundary values of confidence intervals should be separated by a comma.
- Boundary values should be padded as necessary to accept negative values and to allow alignment of the decimal place.
- An example is given below:

(-0.12, -0.10) (9.54, 12.91)

### P-values:

• P-values should be reported to 4 decimal places, except values <1.0000 but >0.9999 will be presented as '>0.9999' (e.g., 0.9998 is presented as >0.9999); and values <0.0001 will be presented as '<0.0001' (e.g., 0.0000 is presented as <0.0001). Rounding will be applied after the <0.0001 and >0.9999 rule

### Ratios:

• Ratios should be reported to 1 more decimal place than the original data.

### Spacing:

• There must be a minimum of 1 blank space between columns (preferably 2)

### Denominators:

- If a different count other than the population count is used for a denominator (within the table) to calculate percentages, there should be a row in the table that identifies that number "n".
- Alternatively, a footnote should be included in each table with percentages to indicate the denominator for percentages.

### Missing values:

- A "0" should be used to indicate a zero frequency.
- A blank will be used to indicate missing data in an end-of-text table or patient listing.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

DocuSign Envelope ID: 51DC1E96-B8E2-4815-9E6C-9E3AAB2E5FEE




Statistical Analysis Plan v1.0 - Part B


### FIGURE OUTPUT CONVENTIONS

- Figures should be provided in RTF files generated by SAS.
- Should contain the title or footer.
- The image should be clear and of high quality when viewed in the Word document, and when printed.
- In general, boxes around the figures should be used.

### **DATES & TIMES**

Depending on data available, dates and times will take the form DDMMMYYY THH:MM:SS.

### **SPELLING FORMAT**

English US.

### PRESENTATION OF TREATMENT GROUPS

For outputs, treatment groups will be represented as follows and in this order:

| Treatment Group | For Tables, Graphs and Listings |
|-----------------------------------|---------------------------------|
| RPL554 300 μg double blind | RPL554 300μg |
| RPL554 1000 μg double blind | RPL554 1000μg |
| RPL554 3000 μg double blind | RPL554 3000μg |
| Placebo | Placebo |
| Non-randomized (where applicable) | Non-randomized |

### PRESENTATION OF TREATMENT SEQUENCES

For outputs, treatment sequences will be represented as follows and in that order:

| Treatment Group | For Tables, Graphs and Listings |
|---|---|
| RPL554 300 mcg db/RPL554 3000 mcg db/Placebo/RPL554 1000 mcg db | Seq 1 |

Document: \(\text{\lecturedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 SAP v1.0 - Part B\)

Jennifer Allsopp Version Number: 1


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:




Statistical Analysis Plan v1.0 - Part B


| Treatment Group | For Tables, Graphs and Listings |
|---|---|
| RPL554 1000 mcg db/Placebo/RPL554 3000 mcg db/RPL554 300 mcg db | Seq 2 |
| RPL554 3000 mcg db/RPL554 1000 mcg db/RPL554 300 mcg db/Placebo | Seq 3 |
| Placebo/RPL554 300 mcg db/RPL554 1000 mcg db/RPL554 3000 mcg db | Seq 4 |
| Undefined sequence, not mentioned above | Undefined |
| Non-randomized (where applicable) | Non-randomized |

db = double blind

### PRESENTATION OF VISITS

For outputs, visits will be represented as follows and in that order, considering there will be 4 treatment periods (1 to 4):

| Long Name (default) | Short Name |
|----------------------------|------------|
| Screening | Scr |
| Day 1 | Day 1 |
| Day 7 | Day 7 |
| End of Study | EOS |
| Overall (where applicable) | Overall |

### LISTINGS

All listings will be ordered by the following (unless otherwise indicated in the template):

Randomized treatment group (or treatment received if it's a safety output), first by active dose [by ascending dose group] and then placebo.

Center-patient ID,

Date (where applicable),

For listings where non-randomized patients are included, these will appear in a category after the randomized treatment groups labeled 'Non-randomized'.

 $\begin{tabular}{ll} \begin{tabular}{ll} Document: & \label{tabular} $$ \begin{tabular}{ll} \begin{tabula$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Author:




Statistical Analysis Plan v1.0 - Part B


### APPENDIX 2. PARTIAL DATE CONVENTIONS

Imputed dates will NOT be presented in the listings.

### ALGORITHM FOR TREATMENT EMERGENCE OF ADVERSE EVENTS

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known, | If start date < study med start date, then not TEAE |
| | Partial or | If start date >= study med start date, then TEAE |
| | Missing | |
| Partial, but known | Known, | Not TEAE |
| components show that it | Partial or | |
| cannot be on or after study | Missing | |
| med start date | | |
| Partial, could be on or after | Known | If stop date < study med start date, then not TEAE |
| study med start date | | If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month |
| | | if day unknown or 31st December if day and month are |
| | | unknown), then: |
| | | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |
| Missing | Known | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month |
| | | if day unknown or 31st December if day and month are |

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v1.0 - Part B


| START DATE | STOP DATE | ACTION |
|------------|-----------|----------------------------------------------------|
| | | unknown), then: |
| | | If stop date < study med start date, then not TEAE |
| | | If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |

### ALGORITHM FOR PRIOR / CONCOMITANT MEDICATIONS

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |
| | | If stop date >= study med start date and start date > end of treatment, assign |
| | | as post study |
| | Partial | impute stop date as latest possible date (i.e. last day of month if day |
| | | unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | ssign as concomitant |
| | Missing | If stop date is missing could never be assumed a prior medication |
| | | If start date <= end of treatment, assign as concomitant |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month if day |
| | | unknown or 1st January if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona\_RPL554-MD-201

SAP v1.0 – Part B


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018




Statistical Analysis Plan v1.0 - Part B


| CT + DT D + TT | CTOP DATE | L OFFICIAL |
|---|---|---|
| START DATE | STOP DATE | ACTION |
| | Partial | Impute start date as earliest possible date (i.e. first day of month if day |
| | | unknown or 1st January if day and month are unknown) and impute stop |
| | | date as latest possible date (i.e. last day of month if day unknown or 31st |
| | | December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date and start date <= end of treatment, |
| | | assign as concomitant |
| | Missing | Impute start date as earliest possible date (i.e. first day of month if day |
| | | unknown or 1st January if day and month are unknown), then: |
| | | If stop date is missing could never be assumed a prior medication |
| | | If start date <= end of treatment, assign as concomitant |
| Missing | Known | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date, assign as concomitant |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day |
| | | unknown or 31st December if day and month are unknown), then: |
| | | If stop date < study med start date, assign as prior |
| | | If stop date >= study med start date, assign as concomitant |
| | Missing | Assign as concomitant |

 $SAP\ v1.0-Part\ B$ 


Template No.: CS\_TP\_BS016 Revision 5 Reference: CS\_WI\_BS005

Effective Date: 01Apr2018

Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3



# TABLES, LISTINGS AND FIGURES SHELLS - PART A

RPL554-MD-201

Single and Repeat Doses of RPL554 Administered by Pressurised Metered Inhaler in Patients with A Phase II, Randomized Study to Assess the Pharmacokinetics, Safety and Pharmacodynamics of COPD

**AUTHOR:** NICHOLAS ROUBINIS/JENNIFER ALLSOPP

VERSION NUMBER AND DATE: V2.0, 13JAN2021

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

Version: 2.0 Date: 13JAN2021

Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

# TABLES, LISTINGS AND FIGURES SHELLS – PART A SIGNATURE PAGE

Tables, Listings and Figures Shells V2.0 - Part A (Dated 13JAN2021) for Protocol RPL554-MD-201.

| Date | 1/19/2021 | | | |
|---|---|---|---|---|
| Signature | DocuSigned by: | No is is its in Michael | Jama de musepp | |
| Name | Jennifer Allsopp | | Senior Biostatistician | IQVIA |
| | Author: | | Position: | Company: |

Upon review of this document, the undersigned approves this version of the Tables, Listings and Figures Shells – Part A, authorizing that the content is acceptable for the reporting of this study.

| Date | 1/19/2021 | | | | 1/19/2021 | | | | 1/19/2021 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Signature | Docusigned by: | F2A9CBA2FB8F4B7 | | | DocuSigned by: | Town OleanA | C18201276700452 | | DocuSigned by: | T. 4.00 P. 1. Ace. | Lumas Cura sour | 907 000427208420 |
| Name | Mark Shaw | Manager, Biostatistics | IQVIA | | Tara Rheault | | VP, R&D | Verona Pharma | Thomas Bengtsson | | Statistical Consultant to Verona | StatMind |
| | Approved by: | Position: | Company: | Customer Representative | Approved by: | | Position: | Company: | Approved by: | | Position: | Company: |


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

 $Version \ 1.0; \ 17 \ May \ 2021$  Docusign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

# Modification History

| Unique Identifier for<br>this Version | Date of the Document Author | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| 1.0 | 27SEP2019 | Nicholas | Not Applicable – First Draft Version |
| | | Roubinis/ | |
| | | Jennifer | |
| | | Allsopp | |
| 1.1 | 04MAY2020 | Jennifer | 1. Update figure numbering from Figure 14.2.5-14.2.8 to 14.3.1-14.3.4. |
| | | Allsopp | 2. Update listing numbering from Listing 16.2.2.1 to 16.2.3.1. |
| | | | 3. Update lisiting numbering from Listing 16.2.3.1 to 16.2.2.1. |
| | | | 4. Remove DOB from the demographic listing. |
| | | | 5. Update customer representative from Brian Maurer to Nancy Herje. |
| | | | 6. Update footnotes following review of Part A dose finding analysis. |
| | | | 7. Add shell for F14.2.5 - requested as part of the additional dose finding outputs. |
| 1.2 | 09DEC2020 | Jennifer | 1. Update customer representative from Nancy Herje to Tara Rheault. |
| | | Allsopp | 2. Aded footnote to table 14.1.5.1 detailing how patients met protocol requirements of |
| | | | the reversibility test. |
| | | | 3. Update title for tables 14.3.5 and 14.3.9 to clarify that the tables are displaying |
| | | | discontinuation of study rather than study medication. |
| | | | 4. Added column for patients who discontinued between Part A and Part B to listing |
| | | | 16.2.1.1. |
| 2.0 | 13JAN2021 | Jennifer | Add Thomas Bengtsson as an approver for Verona. |
| | | Allsopp | |


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


# Table of Contents

| ables | |
|---|---|
| le 14.1.1 Par | |
| Table 14.1.2 Analysis Sets (All Patients Enrolled in Part A) | |
| Table 14.1.3 Critical/Major/Winor Protocol Deviations (ALL Randomised Analysis Set in Part A) | |
| Table 14.1.4.1 Demographic Characteristics (All Randomized Analysis Set in Part A) | |
| Table 14.1.4.2 Demographic Characteristics (Safety Analysis Set in Part A)14 | |
| Table 14.1.4.3 Demographic Characteristics (Full Analysis Set in Part A) | |
| Table 14.1.4.4 Demographic Characteristics (Pharmacokinetics Analysis Set in Part A) | |
| Table 14.1.5.1 Screening Disease Characteristics (All Randomized Analysis Set in Part A) | |
| Table 14.1.5.2 Screening Disease Characteristics (Safety Analysis Set in Part A) | |
| Table 14.1.5.3 Screening Disease Characteristics (Full Analysis Set in Part A) | |
| Table 14.1.5.4 Screening Disease Characteristics (Pharmacokinetics Analysis Set in Part A) | |
| Table 14.1.6 COPD and Smoking History (All Randomized Analysis Set in Part A) | |
| 14.2 Efficacy | |
| Secondary Efficacy | |
| Table 14.2.1 FEV1 by Treatment and Timepoint Pre- and Post- Single Dose (Full Analysis Set in Part A) | |
| Table 14.2.2 Change from Baseline FEV; to Average FEV; (over 4 hours) After Single Dose (Full Analysis Set in Part A) 25 | |
| Table 14.2.3 Change from Baseline FEV1 to Average FEV1 (over 12 hours) After Single Dose (Full Analysis Set in Part A) | |
| Table 14.2.3a Change from Baseline FEV; to Average FEV; (over 12 hours) After Single Dose - Sensitivity Analysis (Full Analysis Set in Part A) | |
| Table 14.2.4 Change from Baseline FEV; to Peak FEV; (over 4 hours) After Single Dose (Full Analysis Set in Part A) | |
| 14.3 Safety | |
| Adverse Event | |
| Table 14.3.1 Treatment-emergent Adverse Events Summary (Safety Analysis Set in Part A) | |
| Table 14.3.2 Treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part A) 31 | |
| Table 14.3.3 Treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part A) | |
| Table 14.3.4 Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Analysis Set in Part A) 33 | |
| Table 14.3.5 Treatment-emergent Adverse Events Leading to Discontinuation of Study by System Organ Class and Preferred Term (Safety Analysis Set in Part A) | |
| Table 14.3.6 Serious treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part A) . 35 | |
| ocument: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | |
| hypor Michalse Bouhinis/Jamifar 1112000 Date: 12.1120000 | 2.0 |
| | 7 7 0 7 |

CONFIDENTIAL Verona Pharma plc

 $Version~1.0;~17~May~2021\\ DocuSign~Envelope~1D:~5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3$ 

| Version: 2 | nitton. Nicholo Doibisi / Townifor 11 looms |
|---|---|
| | Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A |
| 59 | Figure 14.3.4 Mean Change from Baseline in Pulse Rate over Time by Treatment (Safety Analysis Set in Part A) |
| 65 | Figure 14.3.3 Mean Change from Baseline in Pulse Rate by Treatment (Safety Analysis Set in Part A) |
| | Figure 14.3.2 Mean Change from Baseline in Heart Rate over Time by Treatment (Safety Analysis Set in Part A) |
| | Figure 14.3.1 Mean Change from Baseline in Heart Rate by Treatment (Safety Analysis Set in Part A) |
| 57 | Figure 14.2.5 Change from Pre-dose FEV1 over Time by Treatment by Subject (Full Analysis Set in Part A) |
| 56 | Figure 14.2.4 Mean Change from pre-dose FEV; during spirometry over Time by Treatment (Full Analysis Set in Part A) |
| Part A) 55 | (over 4 hours) to pre-dose $\ensuremath{\text{FEV}}_1$ by Treatment (Full Analysis Set in |
| in Part A) 54 | Figure 14.2.2 Geometric Mean of ratios of Average FEV, (over 12 hours) to pre-dose FEV, by Treatment (Full Analysis Set |
| Part A) . 54 | Figure 14.2.1 Geometric Mean of ratios of Average FEV; (over 4 hours) to pre-dose FEV; by Treatment (Full Analysis Set in |
| 54 | Figures |
| 53 | Table 14.3.26 Physical Examination Data by Timepoint (Safety Analysis Set in Part A) |
| 53 | Physical Examination |
| in Part A) 52 | Table 14.3.25 Change from Baseline Pulse Rate to Peak Pulse Rate (over 4 hours) After Single Dose (Safety Analysis Set |
| 50 | Table 14.3.24 Vital Sign Data - Markedly Abnormal Values (Safety Analysis Set in Part A) |
| 48 | Table 14.3.23 Vital Sign Data - Change from Pre- to Post- dose by Timepoint (Safety Analysis Set in Part A) |
| 48 | Vital Signs |
| n Part A) 47 | Table 14.3.22 Change from Baseline Heart Rate to peak Heart Rate (over 4 hours) After Single Dose (Safety Analysis Set . |
| Part A) 46 | Table 14.3.21 12-Lead Electrocardiogram - Shifts from Pre-Dose Local Lab Assessment by Timepoint (Safety Analysis Set in |
| 44 | Table 14.3.20 12-Lead Electrocardiogram Data by Timepoint (Safety Analysis Set in Part A) |
| 44 | BCG |
| 43 | Table 14.3.19 Hematology Laboratroy Data at Screening - Markedly Abnormal Values (Safety Analysis Set in Part A) |
| 42 | Table 14.3.18 Viral Serology Laboratroy Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A) |
| 42 | Table 14.3.17 Urinalysis Laboratroy Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A) |
| 42 | Table 14.3.16 Biochemistry Laboratroy Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A) |
| 41 | Table 14.3.15 Hematology Laboratroy Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A) |
| 40 | Table 14.3.14 Viral Serology Laboratroy Data at Screening (Safety Analysis Set in Part A) |
| 39 | Table 14.3.13 Urinalysis Laboratroy Data at Screening (Safety Analysis Set in Part A) |
| 388 | Table 14.3.12 Biochemistry Laboratroy Data at Screening (Safety Analysis Set in Part A) |
| 37 | Table 14.3.11 Hematology Laboratroy Data at Screening (Safety Analysis Set in Part A) |
| 37 | Laboratory |
| Analysis Set | Table 14.3.10 Treatment-emergent Adverse Events with Outcome of Death by System Organ Class and Preferred Term (Safety in Part A) |
| Preferred Term | Table 14.3.9 Serious treatment-emergent Adverse Events Leading to Discontinuation of Sutdy by System Organ Class and Pro (Safety Analysis Set in Part A) |
| (Safety Analysis | Table 14.3.8 Serious treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safe' Set in Part A) |
| Term (Safety 35 | Table 14.3.7 Serious treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Analysis Set in Part A) |
| | 1/ 3 7 Morious troutmost Douglasson Dispared Doluthod to Attack Modication Strategic Organ Creates Department |


| Listings |
|---|
| Listing 16.2.1.1 Completed/Discontinued Patients (All Randomized Analysis Set in Part A) |
| Listing 16.2.2.1 Protocol Deviations (All Randomized Analysis Set in Part A) |
| Listing 16.2.3.1 Patients Excluded from Analysis Sets (All Randomized Analysis Set in Part A) |
| Listing 16.2.4.1 Demographic Characteristics (All Randomized Analysis Set in Part A) |
| Listing 16.2.4.2 Screening Disease Characteristics (All Randomized Analysis Set in Part A) 64 |
| Listing 16.2.4.3 COPD and Smoking History (All Randomized Analysis Set in Part A) |
| Listing 16.2.4.4 Medical History (All Randomized Analysis Set in Part A) |
| Listing 16.2.4.5 Surgical Procedure History (All Randomized Analysis Set in Part A) |
| Listing 16.2.4.6 Prior and Concomitant Medications (All Randomized Analysis Set in Part A) |
| Listing 16.2.5.1 Drug Exposure and Accountability (All Randomized Analysis Set in Part A) |
| Listing 16.2.6.1 Spirometry: FEV1 Results (Full Analysis Set in Part A)70 |
| Listing 16.2.6.2 Spirometry: FEV1 Derived Measurements (Full Analysis Set in Part A) |
| Listing 16.2.6.3 Rescue Medications Taken at Site (All Randomized Analysis Set in Part A) |
| Listing 16.2.6.4 Rescue Medication Taken between Visits (All Randomized Analysis Set in Part A) |
| Listing 16.2.7.1 All Adverse Events (Safety Analysis Set in Part A)74 |
| Listing 16.2.7.2 Treatment-emergent Adverse Events Leading to Study Discontinuation (Safety Analysis Set in Part A) 75 |
| Listing 16.2.7.3 Treatment-emergent Adverce Events Leading to Death (Safety Analysis Set in Part A) |
| Listing 16.2.7.4 Serious Treatment-emergent Adverse Events (Safety Analysis Set in Part A)75 |
| Listing 16.2.7.5 Serious Treatment-emergent Adverse Events - Details (Safety Analysis Set in Part A) |
| Listing 16.2.8.1 Hematology (Safety Analysis Set in Part A) 78 |
| Listing 16.2.8.2 Biochemistry (Safety Analysis Set in Part A) 78 |
| Listing 16.2.8.3 Urinalysis (Safety Analysis Set in Part A)79 |
| Listing 16.2.8.4 Viral Serology (Safety Analysis Set in Part A) 79 |
| Listing 16.2.9.1 Electrocardiogram Local Reading Overall Evaluation (Safety Analysis Set in Part A) |
| Listing 16.2.9.2 12-Lead ECG (Safety Analysis Set in Part A) 81 |
| Listing 16.2.9.3 Vital Signs (Safety Analysis Set in Part A) |
| Listing 16.2.9.4 Derived Safety Measurements (Safety Analysis Set in Part A) |
| Listing 16.2.9.5 Brief Physical Examination (Safety Analysis Set in Part A) |
| Listing 16.2.9.6 Full Physical Examination (Safety Analysis Set in Part A) |
| Listing 16.2.9.7 Chest X-ray (All Randomized Analysis Set in Part A) |
| Listing 16.2.9.8 Inhalation Training (All Randomized Analysis Set in Part A) |
| Listing 16.2.9.9 Pregnancy Serum and Urine Test at Screening (All Randomized Analysis Set in Part A) |
| Listing 16.2.9.10 Pregnancy Report at Screening (All Randomized Analysis Set in Part A) |

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


**Tables** 14.1 Demographic Data

Table 14.1.1 Patient Disposition (All Patients Enrolled in Part A)

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.1.1

Part A Page X of Y

Patient Disposition

(All Patients Enrolled in Part A)

| | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | | |
|---|---|---|---|---|---|---|---|
| | 100µg | 300µg | 1000µg | 3000μg | 6000µg | Placebo | Overall |
| Description, n (%) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Number of patients enrolled | | | | | | | XX |
| Screen failures | | | | | | | ×× |
| Number of patients randomized | xx (100.0) | xx (100.0) | )) xx (100.0) | xx (100.0) | xx (100.0) | xx (100.0) | xx (100.0) |
| Number of patients treated | xx (xx.x) | xx (xx.x) | (xxxx) xx ( | xx (xx.x) | (xx.x) xx | xx (xx.x) | xx (xx.x) |
| Number of patients who completed<br>Part A | xx (xx.x) | (x.xx) | (xx.x) | xx (xx.x) | xx (xx.x) | (x.x.x) | xx (xx.x) |
| Number of patients who discontinued | xx (xx.x) | xx (xx.x) | (x.xx) xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of patients who discontinued between Part A and Part B | | | | | | | |
| Primary reason for early study discontinuation | | | | | | | |
| Adverse event | xx (xx.x) | xx (xx.x) | (xx.x) xx ( | xx (xx.x) | (xxx) xx | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | (xx.x) (xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | (xx.x) (xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | (xx.x) xx ( | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol violation | xx (xx.x) | xx (xx.x) | (xx.x) (xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | xx (xx.x) | xx (xx.x) | (xx.x) (xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | xx (xx.x) | (x.xx) | (x.x.x) (xx | xx (xx.x) | (xxxx) xx | xx (xx.x) | xx (xx.x) |
| Withdrawal by patient | xx (xx.x) | xx (xx.x) | (xx.x) (xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | (xx.x) (xx ( | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | cumentation/ | SAP\Verona F | PL554-MD-201 TI | LF Shells v2.0 | - Part A | | |
| Author: Nicholas Roubinis/Jennifer Allsopp | | | | | | | Version: 2.0<br>Date: 13JAN2021 |

CONFIDENTIAL Verona Pharma plc


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

n = number of patients. N = Number of patients randomized. % = percentage of patients calculated relative to the total number of patients in the All Randomized Analysis Set. Percentage for early discontinuation reasons is calculated based on the number of patients who had early discontinuation data.

Source: Listing 16.2.1.1

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

Verona Pharma plc


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.1.2 Analysis Sets (All Patients Enrolled in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.1.2

Analysis Sets

(All Patients Enrolled in Part A)

| | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | | |
|---|---|---|---|---|---|---|---|
| | Edunt | 30049 | prinna | 300013 | brinna | Flacebo | OVERALL |
| Analysis Set, n (%) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| All Enrolled Analysis Set | × | ×× | ×× | ×× | × | × | × |
| All Randomized Analysis Set | xx (100.0) | xx (100.0) | xx (100.0) | xx (100.0) | xx (100.0) | xx (100.0) | xx (100.0) |
| Safety Analysis Set | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Full Analysis Set | (x.xx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x · xx) xx | (xxxx) xx | (x.x) xx |
| Pharmacokinetics Analysis<br>Set | (xx,x) | (xx.x) | (x · xx) | (xxx) xx | (xx,x) | AN | (xxx) xx |

FEV.: Forced expiratory volume in one second. Na. Not applicable. n = number of patients. N = number of patients randomized. % = percentage of patients calculated relative to the tordal number of patients and the state of the tordal number of patients in the state of the tordal number of patients enrolled. All Randomized Analysis Set: Randomized Analysis Set with sufficient data to compute the pharmacodynamic parameters (FEV, measurement pre-dose and at least one post-dose). Pharmacokinetics Analysis Set: Patients included in the All Randomized Analysis Set who have a blood sampling performed after at least one dose of study medication and pharmacokinetic parameter data.

Source: Listing 16.2.2.1

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


# Version 1.0; 17 May 2021

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.1.3 Critical/Major/Minor Protocol Deviations (ALL Randomised Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.1.3

Critical/Major/Minor Protocol Deviations

(All Randomized Analysis Set in Part A)

| everity/ | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Deviation type | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

| Severity/ | ī | 100µg | 300 | 300µg | 1000µg | r d | 300 | 3000µg | 009 | 6000pg | Plac | Placebo | Overall | all |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Deviation type | Z) | (N=XX) | (N=XX) | (XX | (N=XX) | (X | (N=XX) | (XX | Ä, | (N=XX) | N) | (N=XX) | (N=XX) | (X) |
| Patients with at least one critical/major/minor protocol deviation, n (%) | ×× | xx (xx.x) | ć)<br>XX | x (xx.x) xx | xx (xx.x) | | ×) ×× | : (x.xx) xx | ()<br>(X | xx (xx.x) xx | ()<br>XX | xx (xx.x) xx (xx.x) | ×) | (×.× |
| Critical | × | (xx.x) | xx (xx.x) | | (x.xx) xx | | (x.xx) xx | | C<br>X | xx (xx.xx) | C<br>X | xx (xx.x) | (x.xx) xx | (× :× |
| Type 1 | × | | xx (xx.x) | | xx (xx.x) | | (x.xx) xx | | × | | C)<br>XX | | xx (xx.x) | ×.× |
| Type 2 | × | xx (xx.x) | xx (xx.x) | | xx (xx.x) | | (xx.x) | | × | xx (xx.x) | C XX | xx (xx.x) | (xx.x) | (× · × |
| : | | | | | | | | | | | | | | |

CTMS: Clinical trial management system. n = number of patients. N = Number of patients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. Protocol deviations were obtained from CTMS.

Source: Listing 16.2.3.1

Major

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Deviation types are sorted in descending order of frequency of the Overall column. A patient may have multiple critical/major/minor protocol deviations within and is counted once at each level of summarization.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.1.4.1 Demographic Characteristics (All Randomized Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Page X of Y Part A

(All Randomized Analysis Set in Part A) Demographic Characteristics Table 14.1.4.1

| Variable/ | RPL554<br>100µg | RPL554<br>300µg | RPL554 1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Апе (уеага) | | | | | | | |
| (141) | | | | | | | |
| ч | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| Mean | ××× | ××.× | ××.× | ×.×× | ×.× | ××.× | x.xx |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | x.xx | ×.× | x.xx | x.xx | ×.×× | ×××× | ×. × |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Sex, n (%) | | | | | | | |
| Male | (x.x) xx | (xx.x) | (x.xx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx |
| Female | (x : xx) | (xx.xx) | (xx, xx) | (x.x.) | (xx.x) | (x : xx) | (xx.x) |
| Childbearing potential, n (%) * | | | | | | | |
| Yes | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xxx) xx | (x.x.) | (x.xx) |
| No | (x · xx) | (x · xx) | (x · xx) | (x : xx) | (x : xx) | (x · xx) | (x · xx) |
| Primary race, n (%) | | | | | | | |
| American Indian or Alaska | (xx,x) | (xx.x) | (xx,x) | (xx.x) | (xxx) xx | (xxx) xx | (x, xx) |
| Native Asian | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) |
| Black or African American<br>Native Hawaiian or Other | (x · xx) xx | xx (xx.x) | (x.x) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.x.) xx |
| Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.x.x) | xx (xx.x) |
| White | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx | xx (xx.x) |
| Document: Z:\RPL554\EZAA8488\Bio | statistics\Docum | nentation\SAP\V | EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | 1 TLF Shells v2 | 2.0 - Part A | | |
| Author: Nicholas Roubinis/Jennifer Allsopp | er Allsopp | | | | | | Version: 2.0 Date: 13JAN2021 |
| | 1 | | | | | | |


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Table 14.1.4.1

Part A Page X of Y

> (All Randomized Analysis Set in Part A) Demographic Characteristics

Version: 2.0 Date: 13JAN2021 xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) (xx.xx) xx (xx.x) xx, xx Overall ××.×× xx.x (N=XX) ××× × × xx (xx.x) (xx.x) xx (xx.x) xx (xx.x)  $(x \cdot x \cdot x)$ xx (xx.x) (xxx) xx xx (xx.x) Placebo xx, xx xx.xx x.xx (N=XX) ×.× × × ×× (xxxx) xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) RPL554 6000µg Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A xx, xx xx.xx xx.x (N=XX) x.xx × × xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) (xx.x) RPL554 3000µg xx, xx xx.x (N=XX) ×.× xx.xx × × RPL554 1000µg xx (xx.x) (xx.x) xx (xxx) xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) (N=XX) ××.× xx.xx ××.× × × xx (xx.x) xx (xx.x) xx (xx.x) (xxx) xx xx (xx.x) (x.xx) xx (xx.xx) xx xx (xx.x) RPL554 300µg xx, xx xx.xx ××.× (N=XX) ××.× × × xx (xx.x) (xxx) xx (xxx) xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx, xx 100µg xx.xx ××. (N=XX) ××× × × Author: Nicholas Roubinis/Jennifer Allsopp Asian-Southeast Asian Heritage White-White/Caucasian/European Asian-East Asian Heritage Asian-Central/South Asian African American/African Hispanic or Latino Ethnicity, n (%) Not reported Weight (kg) Height (cm) Category Min, Max Variable/ Median Other Mean SD q


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Table 14.1.4.1

Page X of Y Part A

Demographic Characteristics

(All Randomized Analysis Set in Part A)

| Variable/ | RPL554<br>100µg | RPL554<br>300µg | RPL554 1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| : | | | | | | | |
| Mean | x.xx | xx.x | xx.x | x.xx | x.x. | x.xx | x.x. |
| SD | xx.xx | ××.×× | ××·×× | ××.×× | ××·×× | ××.×× | xx.xx |
| Median | x.xx | x.xx | x.xx | ×.×× | x.xx | ××.×× | x.xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| BMI $(kg/m^2)$ | | | | | | | |
| п | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| Mean | x.xx | ×.× | x.xx | × × × | ×.×x | x.xx | ×.×× |
| SD | xx.xx | ××.×× | xx.xx | ××.×× | xx.xx | ××.×× | xx.xx |
| Median | ×.×× | ×.<br>×. | ××× | × · × × | ×: × | ××× | ×.×. |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

BMI: Body Mass Index. SD: Standard deviation. n = number of patients. N = Number of patients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. % % = Percentage for childbearing potential calculated relative to the total number of female patients in the analysis set. Age (years) = As calculated relative to informed consent date. BMI  $(kg/m^2)$  = weight (kg) / height  $(m)^2$ .

Source: Listing 16.2.4.1

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Print all statistics and categories even if they are empty, except for the row of missings which will only be shown if present and is not shown in the shell here.

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

```
Programming Notes: Print if the number of patients in the SAF analysis set is different to the RWD analysis set.
Table 14.1.4.2 Demographic Characteristics (Safety Analysis Set in Part A)
                                                                                                                                           DM002: This output uses shell DM001 [Table 14.1.4.1]
```

Programming Notes: Print if the number of patients in the SAF analysis set is different to the RND analysis set. Table 14.1.4.3 Demographic Characteristics (Full Analysis Set in Part A) DM003: This output uses shell DM001 [Table 14.1.4.1]

```
Programming Notes:
Print if the number of patients in the SAF analysis set is different to the RND analysis set.
Do not present Placebo treatment group as Placebo is not included for Pharmacokinetics analysis set.
Table 14.1.4.4 Demographic Characteristics (Pharmacokinetics Analysis Set in Part A)
                                                                                                                                                DM004: This output uses shell DM001 [Table 14.1.4.1]
```

Version: 2.0 Date: 13JAN2021 Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc


Table 14.1.5.1 Screening Disease Characteristics (All Randomized Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Part A Page X of Y

(All Randomized Analysis Set in Part A) Screening Disease Characteristics Table 14.1.5.1

| Variable/ | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Pre-bronchodilator ${\tt FEV_1}$ | | | | | | | |
| . ជ | ×× | ×× | ×× | × | × | ×× | ×× |
| Mean | x.xx | ×.× | x.xx | ×.× | ×.×. | x.xx | ×.×. |
| SD | xx.xx | xx · xx | xx ·xx | xx.xx | ××.×× | ××.×× | xx.xx |
| Median | ××.× | ×.×. | x.x.x | x.xx | ×.×× | x.xx | x.xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx 'xx | xx, xx | xx, xx | xx, xx |
| Pre-bronchodilator FEV1 (% of predicted normal) | | | | | | | |
| ц | ×× | × | ×× | × | × | ×× | ×× |
| Mean | ××× | ×.×× | ××× | ××× | ×.×. | ×××× | ××× |
| SD | xx.xx | ××××× | xx.xx | xx.xx | xx.xx | XX.XX | xx.xx |
| Median | x.xx | ×.×× | ×.× | ×.×. | ××× | x.xx | × : × |
| Min, Max | xx, xx | xx, xx | xx, xx | xx 'xx | xx, xx | xx, xx | xx, xx |
| Post-bronchodilator FEV <sub>1</sub> (L) | | | | | | | |
| с | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| Mean | ××. | ×. × | ×.×× | ×.×. | ×.× | ×.×× | ×.×. |
| SD | xx.xx | xx · xx | xx ·xx | xx.xx | ××.×× | ××.×× | xx.xx |
| Median | ×××× | ×.×× | ×××× | ×.×× | x.x. | x.xx | ×.×× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | 188\Biostatisti | cs\Documentation' | SAP\Verona RPL55 | 4-MD-201 TLF Shel | ls v2.0 - Part A | | Version: 2.0 |
| Author: Nicholas Roubinis/Jennifer Allsopp | Jennifer Allso | đơ | | | | | Date: 13JAN2021 |

CONFIDENTIAL Verona Pharma plc

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Table 14.1.5.1

Screening Disease Characteristics (All Randomized Analysis Set in Part A)

| Variable/ | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

| Post-bronchodilator FEV1 (% of predicted normal) | | | | | | | |
|---|---|---|---|---|---|---|---|
| п | ×× | ×× | ×× | ×× | ×× | ×× | ×× |
| Mean | ××.× | ×××× | ×××× | ×.×× | ×××× | ×××× | ×××× |
| SD | ××.×× | xx.xx | ××.×× | ××.×× | xx.xx | ××.×× | xx.xx |
| Median | ××.× | ×××× | ×××× | ×.×× | ×××× | ×××× | ×××× |
| Min, Max | xx, xx | xx 'xx | xx, xx | xx 'xx | xx, xx | xx 'xx | xx, xx |
| FEV1 reversibility (mL) | | | | | | | |
| и | ×× | ×× | ×× | × | ×× | ×× | ×× |
| Mean | ×××× | ×××× | ××.× | ×.× | ××.× | ×××× | ×.×× |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | ×.×× | ×××× | ×·×× | ×.×× | ×.×× | x.xx | ×××× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx 'xx | xx, xx | xx, xx | xx, xx |
| FEV1 reversibility (%) | | | | | | | |
| п | ×× | ×× | ×× | × | ×× | ×× | ×× |
| Mean | × : × | ×××× | ×: ×× | ××.× | ××× | ×.× | ××× |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | ×.×× | ×××× | ×: ×× | ×.×. | ×: ×× | ×××× | ×××× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Table 14.1.5.1

Part A Page X of Y

Screening Disease Characteristics

(All Randomized Analysis Set in Part A)

| Variable/ | RPL554<br>100uq | RPL554<br>300uq | RPL554<br>1000uq | RPL554<br>3000uq | RPL554<br>6000uq | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Statistics | (N=XX) | (N=XX) | (N=XX) | (X=N) | (N=XX) | (N=XX) | (N=XX) |
| Pre-bronchodilator FVC | | | | | | | |
| (T) | × | × | ×× | ×× | ×× | ×× | ×× |
| Mean | ×.× | ×××× | x.xx | ××.× | xx.x | ×.× | x.xx |
| SD | xx.xx | xx.xx | XX.XX | xx.xx | xx.xx | xx.xx | XX.XX |
| Median | × × × | ×.× | ×.× | × × × | ×.× | ×.×× | × · × |
| Min, Max | xx, xx | xx 'xx | xx 'xx | xx 'xx | xx 'xx | xx, xx | xx, xx |
| Post-bronchodilator FVC $(L)$ | | | | | | | |
| r | ×× | ×× | ×× | ×× | ×× | ×× | XX |
| Mean | × × × | ×.× | ×.× | × × × | ×.× | ×.×× | × · × |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX |
| Median | × × × | ×.× | ×.× | × × × | ×.× | ×.×× | × · × |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Pre-bronchodilator<br>FEV1/FVC | | | | | | | |
| ū | × | ×× | ×× | ×× | × | × | ×× |
| Mean | ×.× | ×××× | ×.×× | ×.× | ××× | ×.× | ×.×× |
| SD | ××.×× | xx.xx | xx.xx | ××.×× | xx.xx | ××.×× | xx.xx |
| Median | ×.× | x.xx | ×.× | ×.× | x.xx | x.xx | x.xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Post-bronchodilator<br>FEVI/FVC<br>Promment: 7.NDDISGANDANDANDNDNDNDNDANMENTSHIANNQADNVaxons DDISGALMD-201 mTF challe w2 0 - Dawt A | | 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 7 | E TE TO COMP. | - 0 C++ 0 C | | |
| Author: Nicholas Roubinis/Jennifer Allsopp | Jennifer Allsop | | | | יים | | Version: 2.0<br>Date: 13JAN2021 |


CONFIDENTIAL Verona Pharma plc


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Table 14.1.5.1

Page X of Y Part A

Screening Disease Characteristics

(All Randomized Analysis Set in Part A)

| | K | RPL554 | RPI | RPL554 | RPL554 | K | RPL554 | RPL55 | 4 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable/ | | 100µg | 30 | 300µg | 1000µg | m | 3000µg | 6000рд | מ | Placebo | ebo | Overall | all |
| Statistics | ٥ | (N=XX) | =N) | (N=XX) | (N=XX) | _ | (N=XX) | (N=XX) | ~ | (N=XX) | (X) | (N=XX) | XX) |
| и | | XX | ^ | ×× | ×× | | ×× | × | | × | | × | ×× |
| Mean | | ×.× | × | ×.×× | ×.× | | ×.× | ×.×. | | ××. | × | × | ×.× |
| SD | × | ××.×× | × | xx.xx | XX.XX | ^ | xx.xx | xx.xx | | xx.xx | ×× | xx.xx | XX |
| Median | | × · × | × | ×.× | ×.× | | ××.× | ×.×. | | ××. | × | × | ×.× |
| Min, Max | × | xx, xx | xx, | xx, xx | xx, xx | × | xx, xx | xx, xx | × | xx, xx | ×× | xx, xx | ×× |
| Reversibility assessment performed with four puffs of albuterol, n (%) | | | | | | | | | | | | | |
| Yes | X | (x.xx) xx | ×× | xx (xx.x) | xx (xx.x) | ×× | xx (xx.x) | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | x.x) |
| No | × | xx (xx.x) | ×× | xx (xx.x) | (xx.x) | × | (x.xx) xx | (x.xx) | | (x)<br>xx | (xx.x) | xx (xx.x) | (x · x) |
| Met protocol<br>requirements of<br>reversibility test [a],<br>n (%) | | | | | | | | | | | | | |
| Yes | × | xx (xx.x) | ×× | xx (xx.x) | xx (xx.x) | × | xx (xx.x) | xx (xx.x) | | (xxxx) xx | | xx (xx.x) | (x · x) |
| No | × | xx (xx.x) | ×× | xx (xx.x) | xx (xx.x) | ×× | (xx.x) xx | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | (x.x) |

FEV;. Forced expired volume in 1 second. FVC: Forced vital capacity. SD: Standard deviation. n = number of patients. N = Number of patients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. Prepatients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. Prepatients and reversibility values are the results of the screening reversibility test.

[a] Patients meet the protocol requirements of the reversibility test by demonstatating >=150 mL increase from pre-bronchodilator FEV.

Source: Listing 16.2.4.2

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

# Clinical Study Report

RPL554-MD-201

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Version 1.0; 17 May 2021

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Table 14.1.5.1

Part A Page X of Y

Screening Disease Characteristics

(All Randomized Analysis Set in Part A)

| / o [ de : | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | | |
|---|---|---|---|---|---|---|---|
| T T C T | 100μg | 300µg | 1000µg | 3000µg | 6000pg | Placebo | Overall |
| tatistics | (X=XX) | (N=XX) | (N=XX) | (X=N) | (XX=N) | (N=XX) | (X=XX) |

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Table 14.1.5.2 Screening Disease Characteristics (Safety Analysis Set in Part A)

DM006: This output uses shell DM005 [Table 14.1.5.1]

Programming Notes: Print = P

Table 14.1.5.3 Screening Disease Characteristics (Full Analysis Set in Part A)

DM007: This output uses shell DM005 [Table 14.1.5.1]

Programming Notes: Print = P

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.1.5.4 Screening Disease Characteristics (Pharmacokinetics Analysis Set in Part A)

DM008: This output uses shell DM005 [Table 14.1.5.1]

Programming Notes: Print if the number of patients in the SAF analysis set is different to the RND analysis set. Do not present Placebo treatment group as Placebo is not included for Pharmacokinetics analysis set.


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

Verona Pharma plc


Table 14.1.6 COPD and Smoking History (All Randomized Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Part A Page X of Y

> COPD and Smoking History Table 14.1.6

(All Randomized Analysis Set in Part A)

| Variable/ | 100µg | RPL554<br>300µg | RPL554 1000µg | RPL554 3000µg | RPL554 6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Duration of COPD (years) (time since diagnosis) | | | | | | | |
| ч | ×× | ×× | ×× | ×× | ×× | × | ×× |
| Mean | ×.× | × × × | ×.×× | ×. × | ×. × | ×.× | x.xx |
| SD | xx.xx | xx.xx | XX.XX | xx.xx | ××.×× | xx.xx | xx.xx |
| Median | ×.× | × × × | ×.×× | ×.× | ×. × | ×. × | x.xx |
| Min, Max | xx, xx | xx 'xx | xx 'xx | xx 'xx | xx 'xx | xx, xx | xx 'xx |
| Patient known to have Chronic Bronchitis, n (%) | | | | | | | |
| Yes | (x.xx) xx | (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) |
| Patient known to have Emphysema, n (%)* | | | | | | | |
| ĭes | (x.xx) xx | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NO | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Smoking status, n (%) | | | | | | | |
| Current Smokers | (x.xx) xx | (xxxx) (xx | xx (xx.x) | xx (xx.x) | (x.xx) xx | xx (xx.x) | (x.xx) xx |
| Ex-smokers | xx (xx.x) | ) xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of packs per<br>day | | | | | | | |
| Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part | 48488\Biost | atistics\Documenta | tion\SAP\Verona RPL5 | 54-MD-201 TLF Sh | ells v2.0 - Part A | <i>A</i> 1 | |
| Author: Nicholas Roubinis/Jennifer Allsopp | is/Jennifer | Allsopp | | | | | Version: 2.0 Date: 13JAN2021 |


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Table 14.1.6

Page X of Y Part A

COPD and Smoking History (All Randomized Analysis Set in Part A)

| Variable/ | RPL554<br>100µg | RPL554<br>300µg | RPL554 1000µg | RPL554 3000µg | RPL554 6000µg | Placebo | Overall |
|---|---|---|---|---|---|---|---|
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| ч | ×× | ×× | ×× | ×× | ×× | × | ×× |
| Mean | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | ××××× |
| SD | xx.xxx | xxxxx.xx | xxxxx.xx | xxxxxx | xx.xxx | xxxxx.xxx | xx.xxx |
| Median | xx.xx | xx.xx | xxxx | ×××××× | xx.xx | ××××× | xxx.xx |
| Min, Max | xx.xx, xx.xx | xx.xx, xx.xx | xx.xx, xx.xx | xx.xx, xx.xx | xx.xx, xx.xx | xx.xx, xx.xx | xx.xx, xx.xx |
| Number of years<br>smoking | | | | | | | |
| ជ | ×× | ×× | ×× | XX | ×× | ×× | ×× |
| Mean | xx.xx | xx.xx | ××.×× | ××.×× | XX.XX | XX.XX | xx.xx |
| SD | xx.xx | xx.xxx | XXX.XX | xx.xx | xx.xxx | xx.xx | xx.xx |
| Median | xx.xx | xx.xx | ××.×× | ××.×× | XX.XX | XX.XX | xx.xx |
| Min, Max | x.x, xx.x | x.x, xx.x | x.x, xx.x | x.x, xx.x | x.x, xx.x | x.x, x.x | x.x, x.xx |
| Smoking exposure (pack-years) | | | | | | | |
| ч | ×× | XX | ×× | XX | ×× | ×× | XX |
| Mean | ××.× | ××× | ××× | ××× | ×.× | ×.× | ×.× |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | XX.XX | ××.×× |
| Median | ××× | ×.× | ×.× | ×××× | x.xx | ×.× | ××.× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

COPD: Chronic obstructive pulmonary disease. SD: Standard deviation. n = number of patients. N = Number of patients in the analysis set. set. % = percentage of patients calculated relative to the total number of patients in the analysis set. Number of packs per day = average consumption during their smoking duration. Snoking exposure (pack-years) = number of packs per day x number of packs smoking, for patients with a smoking history or a current smoker. Duration of COPD (years) (time since diagnosis) = Randomization date - first Document: Z:NRPLS54\EZAAA8488\Biostatistics\Documentation\SAP\Verona RPLS54\MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

> COPD and Smoking History Table 14.1.6

(All Randomized Analysis Set in Part A)

| / 0 [ de i x e 1 x | RPL554 | RPL554 | | | | | |
|---|---|---|---|---|---|---|---|
| Valtable/ | 100µg | 300µg | RPL554 1000µg | RPL554 3000µg | RPL554 6000µg | Placebo | Overall |
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

COPD diagnosis date. \* Patients known to have emphysema will potentially overlap with patients known to have chronic bronchitis.

Source: Listing 16.2.4.3

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

 Verona Pharma plc


Document: Z:\RPL554\EZBAB488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

14.2 Efficacy

Secondary Efficacy

Table 14.2.1 FEV1 by Treatment and Timepoint Pre- and Post- Single Dose (Full Analysis Set in Part A)

Verona Pharma

Protocol: RPL554-MD-201

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Table 14.2.1

FEV1 by Treatment and Timepoint Pre- and Post- Single Dose

(Full Analysis Set in Part A)

| | | | | | | Statistics | | |
|---|---|---|---|---|---|---|---|---|
| Timepoint | Treatment group | Category | п | Mean | SD | Minimum | Median | Maximum |
| 1-hour pre-<br>dose | RPL554 100µg (N=xx) | Result | × | ×<br>×<br>× | ××·×× | ××.×× | × : | ××× |
| | RPL554 300µg (N=xx) | Result | × | ×.<br>×. | xx.xx | xx.xx | ××× | × |
| | RPL554 1000µg (N=xx) | Result | XX | x.xx | xx.xx | xx.xx | x.xx | xx.x |
| | RPL554 3000µg (N=xx) | Result | × | ×.×× | ××.×× | xx.xx | ×. ×. | ×.×× |
| | RPL554 6000µg (N=xx) | Result | XX | xx | ××.×× | xx.xx | x.xx | x.xx |
| | Placebo (N=xx) | Result | × | ××× | ××.×× | ××.×× | ××× | × · · × |
| Immediately<br>pre-dose | RPL554 100µg (N=xx) | Result | × | × | xx · xx | xx.xx | × × × | ××× |
| : | 1 | ī | XX | x.xx | xx.xx | xx.xx | x.xx | xx.x |
| 5 minutes<br>post-dose | RPL554 100µg (N=xx) | Result | × | ××. | xx.xx | XX.XX | ×. ×. | ×. |
| | | Pre-dose | ×× | ×. × | xx.xx | xx.xx | ×.× | ×. ×× |
| | | Change from<br>Pre-dose | × | × | ××.×× | ××.×× | × | × |

SD: Standard deviation. FEV:: Forced expired volume in 1 second. n = Number of patients who have an assessment available pre-dose and the relevant post-dose assessment timepoint (Pre-dose and Change from Pre-dose). N = Number of patients in the analysis set. Pre-dose FEV, is defined as the average of the FEV, pre-dose assessment scallected on Day 1 (within 60 and 5 minutes). Change from Pre-dose Post-dose assessment - Pre-dose.

Source: Listing 16.2.6.1

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

FEV1 by Treatment and Timepoint Pre- and Post- Single Dose

(Full Analysis Set in Part A)

| | Maximum |
|------------|-----------------|
| | Median |
| Statistics | Minimum |
| | SD |
| | Mean |
| | и |
| ' | Category |
| | Treatment group |
| | Timepoint |

Programming Notes:

Display for the following days and timepoints, relative to dosing: 1 hour pre-dose and immediately pre-dose, 5 (# 2), 15 (# 5) and 30 minutes (# 10) and 1, 1.5, 2, 4, 8, 11 and 12 hours (the latter assessments all # 15 minutes).

Table 14.2.2 Change from Baseline FEV, to Average FEV, (over 4 hours) After Single Dose (Full Analysis Set in Part A)

EFF006: This output uses shell EFF004 [Table 14.2.4]

ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. FEV: Forced expiratory volume in 1 second. GeoMean. Ratio: Geometric mean ratio to baseline. SD: Standard deviation. N = Number of patients in the analysis set. Baseline: average of the FEV; pre-dose assessments collected on Day 1 (within 60 and 5 minutes). Change from Baseline: Ratio of (Post-dose assessment - Pre-dose), as each assessment will be log-transformed prior to analysis. [a] number of patients with valid values at baseline and timepoints. [b] ANCOVA model is used to model the change from baseline using baseline FEV; as a continuous fixed effect and planned treatment as categorical fixed effects. [c] number of patients with at least one on treatment value who contributed to the model estimation. \* Indicates a significant p-value (<0.05).

Source: Listing 16.2.6.2

Programming Notes

Replace footnotes in original shell with those listed above

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Docusign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.2.3 Change from Baseline FEV1 to Average FEV1 (over 12 hours) After Single Dose (Full Analysis Set in Part A)

EFF007: This output uses shell EFF004 [Table 14.2.4]

GeoMean: GeoMetric mean. GeoMean Ratio: Geometric mean ratio to baseline. SD: Standard deviation. N = Number of patients in the analysis set. Baseline: average of the FEV; pre-dose assessments collected on Day 1 (within 60 and 5 minutes). Change from Baseline: Ratio 6 (Fost-dose assessment - Fre-dose), as each assessment will be log-transformed prior to analysis. [a] number of patients with Ratio 6 (Fost-dose authority. [b] ANCOVA model is used to model the change from baseline using baseline FEV; as a continuous fixed effect and planned treatment as categorical fixed effects. [c] number of patients with at least one on treatment value who contributed to the model estimation. \* Indicates a significant p-value (<0.05). ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. FEV1: Forced expiratory volume in 1 second.

Source: Listing 16.2.6.2

Programming Notes

Replace footnotes in original shell with those listed above

Table 14.2.3a Change from Baseline FEV; to Average FEV; (over 12 hours) After Single Dose - Sensitivity Analysis (Full Analysis Set in Part A)

EFF007: This output uses shell EFF004 [Table 14.2.4]

ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. FEV: Forced expiratory volume in 1 second. GeoMean: GeoMeants. Geometric mean ratio to baseline. SD: Standard devidation. Ne Number of patients in the analysis set. Baseline: average of the FEV; pre-dose assessment sollected on Day 1 (within 60 and 5 minutes). Change from Baseline: Ratio of (Post-dose assessment - Pre-dose), as each assessment will be log-transformed prior to analysis. [a] number of patients with valid values at baseline and timepoints. [b] ANCOVA model is used to model the change from baseline using baseline FEV; as a continuous fixed effect and planned treatment as categorical fixed effects. [c] number of patients with at least one on treatment value who contributed to the model estimation. \* Indicates a significant p-value (<0.05).

Source: Listing 16.2.6.2

Programming Notes

Only include if at least 1 subject has taken rescue medication less than 6 hours prior to spirometry (ANLO2FL="Y") Replace footnotes in original shell with those listed above

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.2.4 Change from Baseline FEV1 to Peak FEV1 (over 4 hours) After Single Dose (Full Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Part A Page X of Y

Table 14.2.4

Change from Baseline FEV1 to Peak FEV1 (over 4 hours) After Single Dose

(Full Analysis Set in Part A)

| | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
|---|---|---|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Baseline FEV1 (L) | | | | | | |
| n [a] | ×× | ×× | XX | ×× | ×× | ×× |
| Mean (SD) | xx.xx (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.xx (xx.xx) |
| Median | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| Min, Max | xx, xx | xx 'xx | ×× ′×× | xx, xx | xx, xx | xx, xx |
| Peak FEV $_1$ (L) | | | | | | |
| Mean (SD) | xx.xx (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.xx (xx.xx) |
| Median | x.xx | ×.× | ×.× | ×××× | ×.× | x.xx |
| Min, Max | xx, xx | xx , xx | xx 'xx | xx, xx | xx, xx | xx, xx |
| CFB FEV1 | | | | | | |
| Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | (xx.xx) | xx.xx) x.xx |
| Median | x.xx | ×.× | ×.×. | ×.×× | ×. ×. | x · · x |
| Min, Max | xx, xx | xx 'xx | xx 'xx | xx, xx | xx, xx | xx, xx |
| Estimates from ANCOVA [b] | | | | | | |
| n [c] | ×× | × | ×× | × | × | × |
| GeoMean | x.xx | x.xx | ×.×. | x.xx | ×.×. | x.xx |
| 95% CI for GeoMean | (xxx, xxxx) | (xxx, xxxx) | (xxx, xx.x) | (xxx, xx.x) | (xxx, xxxx) | (xxx, xxx) |

Comparisons Against Placebo

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Table 14.2.4

Change from Baseline FEV1 to Peak FEV1 (over 4 hours) After Single Dose

(Full Analysis Set in Part A)

| | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
|---|---|---|---|---|---|---|
| | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Treatment Effect - ANCOVA | | | | | | |
| GeoMean Ratio | ×.×× | × · × | × · × | x.xx | ×.×. | |
| 95% CI for GeoMean Ratio | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| p-value | ×××××× | ×. xxxx | ×.××× | x.xxx | x.xxxx | |
| Comparisons Against RPL554 doses | | | | | | |
| Treatment Effect - ANCOVA | | Comparison<br>Against<br>RPL554 100µg | Comparison<br>Against<br>RPL554 300µg | Comparison<br>Against<br>RPL554 1000µg | Comparison<br>Against<br>RPL554 3000µg | |
| GeoMean Ratio | | × . × | × × × | ×.×× | ×.×. | |
| 95% CI for GeoMean Ratio | | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) | |
| p-value | | x.xxxx | ×××××××××××××××××××××××××××××××××××××× | x.xxxx | X.XXXX | |

ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. FEV: Forced expiratory volume in 1 second.
GeoMean: GeoMean Ratio: Geometric mean ratio to baseline. SD: Standard deviation. N = Number of patients in the
analysis set. Baseline: average of the FEV; pre-dose assessments collected on Day 1 (within 60 and 5 minutes). Change from Baseline:
Ratio of (Post-dose assessment - Pre-dose), as each assessment will be log-transformed prior to analysis. [a] number of patients with
valid values at baseline and timepoints. [b] ANCOVA model is used to model the change from baseline using baseline FEV; as a continuous
fixed effect and planned treatment as categorical fixed effects. [c] number of patients with at least one on treatment value who
contributed to the model estimation. \* Indicates a significant p-value (<0.05).

Source: Listing 16.2.6.2

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: Z:/RPL554\EZBA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

# Clinical Study Report

RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

14.3 Safety

Adverse Event

Table 14.3.1 Treatment-emergent Adverse Events Summary (Safety Analysis Set in Part A)

Page X of Y Part A

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Treatment-emergent Adverse Events Summary Table 14.3.1

× (xx.xx)  $\stackrel{\times}{\times}$ xx (xxxx) xx xx (xxxx) xx (xx.xx) xx (xxxx) xx xx (xxxx) xx (xx.x) n (%) E Overall N=XX(xx.x) (xx.x) × × × × × xx (xx.xx) xx xx (xx.xx) xx xx (x.xx) (xx.x) xx (xx.xx) xx xx (xx.xx) xx xx (xxxx) (xx.xx) n (%) E Placebo N=xx (xx.x) × × × × xx (xx.x) xx xx (xx.xx) xx xx (xx.xx) xx xx (xxxx) xx xx (x.xx) xx xx (xx.x) xx xx (x.xx) xx (xx.x) xx xx (xxxx) xx 6000mg n (%) E RPL554 N=XX× xx (xxxx) xx xx (xx.x) xx xx (xxxx) xx xx (xxxx) xx xx (xx.x) xx xx (xxxx) xx xx (xxxx) xx xx (xxxx) xx xx (xxxx) xx n (%) E 3000µg RPL554 N=xx (Safety Analysis Set in Part A) xx (xxxx) xx xx (xx.xx) xx xx (xx.xx) xx xx (xx.xx) xx × (xx.xx) (xx.xx) xx (xxxx) xx xx (xxxx) xx n (%) E RPL554 1000µg N=XX (xx.x) × × × xx (x.xx) xx xx (x.xx) xx xx (xxxx) xx xx (xxxx) xx xx (xxxx) xx xx (xxxx) xx xx (x.xx) xx xx (x.xx) xx xx (xxxx) xx n (%) E RPL554 N=XX300µg xx (xxxx) xx xx (xx.x) xx xx (xx.x) xx xx (xx.x) xx xx (xxxx) xx xx (xxxx) xx xx (xx.x) xx xx (xxxx) xx xx (xxxx) xx n (%) E RPL554 100µg N=XXAny serious TEAE leading Any serious TEAE related to study medication Any TEAEs classified by maximum severity to studydiscontinuation Any TEAE leading to studydiscontinuation Any TEAE related to study medication Any serious TEAE Moderate Category Variable/ Any TEAE Severe Mild

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A Author: Nicholas Roubinis/Jennifer Allsopp

xx (xxxx) xx

xx (xx.xx) xx


xx (xx.xx) xx

xx (xx.x) xx xx (xxxx) xx xx (xxxx) xx

xx (x.xx) xx xx (xxxx) xx

xx (xx.xx) xx xx (xx.x) xx xx (xx.xx) xx

xx (xx.x) xx

xx (xx.xx) xx

xx (xx.xx) xx

xx (xx.xx) xx

classified by maximum

severity

Any serious TEAEs

xx (xxxx) xx

Moderate

Severe

xx (xx.x) xx

xx (x.xx) xx xx (xxxx) xx

xx (xx.xx) xx xx (xx.x) xx

CONFIDENTIAL Verona Pharma plc


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Table 14.3.1

Page X of Y Part A

Treatment-emergent Adverse Events Summary

(Safety Analysis Set in Part A)

| | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | | |
|---|---|---|---|---|---|---|---|
| | 100µg | 300µg | 1000µg | 3000μg | 6000hg | Placebo | Overall |
| Variable/ | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Category | 五 (%) 口 | n (%) E | n (%) E | n (%) E | n (%) E | n (%) E | n (%) E |

xx (xxxx) xx xx (xx.xx) xx xx (xxxx) xx xx (xx.x) xx xx (xx.x) xx xx (xx.xx) xx xx (xx.x) xx Any TEAE leading to death

TEAE: Treatment-emergent adverse event. n = Number of patients with at least one TEAE in each category. E = Number of mentions (events) in each category. N = Number of patients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. TEAE = All AES that started or worsened in severity on or after the single dose of Study medication, based on the investigator assessment of severity. TEAEs with a missing relationship to study medication were regarded as related to study medication. TEAEs starting after the single dose of study medication with a missing severity were classified as

Source: Listing 16.2.7.1

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.2 Treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.2

Treatment-emergent Adverse Events by System Organ Class and Preferred Term

(Safety Analysis Set in Part A)

| System Organ Class | RPL554<br>100µg | RPL554<br>300µg | | RPL554 1000µg | 0µд | 30<br>30 | RPL554<br>3000µg | K 0 | RPL554<br>6000µg | Plac | Placebo |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term [a] | (N=XX) | (N=XX) | | (N=XX) | | N) | (N=XX) | | (N=XX) | (N=XX) | (XX |
| Patients with at least one TEAE | xx (x.x.) xx | xx (x.xx) xx | × | xx (x.xx) xx | | ×)<br>×× | xx (xx.x) xx | ×× | xx (xx.x) xx | ×<br>× | xx (x.xx) xx |
| System Organ Class #1 | xx (xxxx) xx | xx (xxxx) xx | × | xx (xxxx) xx | | xx (xx.x) | x.x) xx | ×× | xx (x.xx) xx | xx (xx.x) | (×. |
| Preferred Term #1 | xx (xx.x) xx | xx (xx.x) | ×× | xx (xx.x) | ×× | xx (xx.x) | xx (x.x | ×× | xx (xx.xx) xx | xx (xx.x) | xx (x. |
| Preferred Term #2 | xx (xx.x) xx | xx (xx.x) xx | ×× | (xxx) xx | × | ×)<br>×× | xx (xx.x) xx | ×× | xx (x.xx) | xx) xx | xx (x.xx) |
| System Organ Class #2 | xx (xx.x) xx | xx (xx.x) xx | ×× | xx (xx.x) xx | | ×) ×× | xx (xx.x) xx | ×× | xx (xx.x) xx | (xxx) xx | .xx (x. |
| Preferred Term #1 | xx (xx.x) xx | xx (xx.x) xx | ×× | xx (xx.x) xx | | ×)<br>×× | xx (xx.x) xx | ×× | xx (xxxx) xx | (x.xx) xx | .xx (x. |
| Preferred Term #2 | xx (x,xx) xx | xx (x.xx) xx | × | xx (x.xx) xx | | ×× | xx (x.xx) xx | ×× | xx (xx,x) xx | (xxx) xx | (×. |

FI: Preferred term. SOC: System organ class. TEAE: Treatment-emergent adverse event. n = number of patients with at least one TEAE in each category. E = Number of mentions (events) in each category. N = Number of patients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. TEAE = All AEs that started or worsened in severity on or after the first dose of study medication, based on the investigator assessment of severity. Each patient is counted once for each applicable specific AE, and a patient with multiple AEs within a SOC is counted once for that SOC. [a] SOCs and PTs are coded using the MedDEA (Version 21.0).

Source: Listing 16.2.7.1

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

SOCs and PTs within each SOC are sorted in descending order of percentage in the highest dose-level group.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.3 Treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part A)

AE003: This output uses shell AE002 [Table 14.3.2]

PT: Preferred term. SOC: System organ class. TEAE: Treatment-emergent adverse event related to study medication. n = number of patients in patients with at least one related TEAE in each category. E = Number of mentions (events) in each category. N = Number of patients in the analysis set. \* = percentage of patients calculated relative to the total number of patients in the analysis set. TEAE = All AEs that started or worsened in severity on or after the first dose of study medication, based on the investigator assessment of related or not. Each patient is counted once for each applicable specific AE, and a patient with multiple AEs within a SOC is counted once for that SOC. [a] SOCs and PTs are coded using the MedDRA (Version 21.0).

Source: Listing 16.2.7.1

Programming Notes:

Replace footnotes in original shell with those listed above

Version: 2.0 Date: 13JAN2021 Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc


Oli 1:0, 17 May 2021 DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Table 14.3.4 Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Analysis Set in Part A)

Page X of Y Part A

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.4

Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity

(Safety Analysis Set in Part A)

| System Organ Class (%) | Maximum | | RPL554<br>100µg | | RPL554<br>300µg | | RPL554<br>1000µg | | RPL554<br>3000µg | | RPL554<br>6000µg | Pl | Placebo |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Preferred Term, n (%) [a] | Severity | | (N=XX) | | (N=XX) | | (N=XX) | | (N=XX) | | (N=XX) | | (N=XX) |
| Patients with at least | C C | | <u>;</u> | ; | | | <u> </u> | | ĵ | ; | <u>;</u> | : | 3 |
| one TEAE, n (%) | ט ארט פר די מיי | × | (x.xx) xx | × | (x.xx) xx | ×× | (x:xx) xx | × | (x.xx) xx | × | (x.xx) xx | × | (x · xx) xx |
| | Moderate | × | (xx.x) | × | xx (xx.x) | )<br>XX | (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xx.x) |
| | Mild | × | (xx.x) | × | (x.xx) xx | ×× | (xx.x) | × | (xx.x) | × | (x.xx) xx | × | (xx.x) |
| System Organ Class #1 | Severe | × | (xxx) xx | × | xx (xx.x) | ×× | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xxx) xx |
| | Moderate | × | (xx.x) xx | × | (x.x.x) | ×× | xx (xx.x) | × | xx (xx.x) | × | (x.x.x) | × | xx (xx.x) |
| | Mild | × | (xx.x) | × | xx (xx.x) | ×× | (xx.x) | × | (xx.x) | × | xx (xx.x) | × | (xx.x) |
| Preferred Term #1 | Severe | × | (xx.x) | × | (xx.x) | ×× | (xx.x) | × | (xx.x) | × | (x.x.x) | × | (xx.x) |
| | Moderate | × | (x.xx) xx | × | (x.x.x) xx | ×× | (x.xx) xx | × | (x · x) | × | (x.xx) xx | × | (x.xx) |
| | Mild | × | (xx.x) | × | (x.x.x) xx | ×× | (x.xx) xx | × | (xx.x) | × | (x.xx) xx | × | (xx.x) |
| Preferred Term #2 | Severe | × | (x.xx) xx | × | (x.xx) xx | ×× | (xx.x) | × | (x · x) | × | (x.xx) xx | × | (x.xx) |
| | Moderate | × | (xx.x) xx | × | (xxxx) xx | ×× | xx (xx.x) | × | xx (xx.x) | × | (xx.x) xx | × | xx (xx.x) |
| | Mild | × | (x.xx) xx | × | (xx.x) xx | ×× | xx (xx.x) | × | xx (xx.x) | × | (xx.x) xx | × | (x.xx) |
| System Organ Class #1 | Severe | × | (xx.x) xx | × | (x.xx) xx | ×× | (x x x) | × | xx (xx.x) | × | (xx.x) xx | × | (x.xx) |
| | Moderate | × | (xx.x) | × | (x.xx) xx | ×× | (xx.x) | × | (xx.x) | × | (xx.x) xx | × | (xx.x) |
| | Mild | × | (x.xx) xx | × | (x.xx) xx | ×× | xx (xx.x) | × | (x.xx) xx | × | xx (xx.x) | × | (x.xx) |
| : | : | : | | : | | : | | : | | : | | : | |

PT: Preferred term. SOC: System organ class. TEAE: Treatment-emergent adverse event. n = number of patients with at least one TEAE in each category. N = Number of patients in the analysis set. % = percentage of patients calculated relative to the total number of patients in the analysis set. TEAE = All AES that started or worsened in severity on or after the first dose of study medication, absed on the investigator assessment of severity. Each patient is counted once for each applicable specific TEAE at the maximum severity and a patient with multiple TEAEs within a SOC is counted once for that SOC at the maximum severity. (a) SOCs and PTS within each SOC are sorted in descending order of percentage of severe AES (then

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

# Version 1.0; 17 May 2021

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler Table 14.3.4

Page X of Y Part A

Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity

(Safety Analysis Set in Part A)

| , 03 | M | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | |
|---|---|---|---|---|---|---|---|
| System Organ Class (%) | Maximum | 100µg | 300µg | 1000µg | 3000μg | 6000pd | Placebo |
| Preferred Term, n (%) [a] | Severity | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

moderate and mild AEs). TEAEs starting after the first dose of study medication with a missing severity will be classified as severe.

Source: Listing 16.2.7.1

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Table 14.3.5 Treatment-emergent Adverse Events Leading to Discontinuation of Study by System Organ Class and Preferred Term (Safety Analysis Set in Part A)

AE005: This output uses shell AE004 [Table 14.3.2]

Programming Notes

Use the same template of table 14.3.2, selecting only the TEAES leading to discontinuation of study and update "Any TEAE" to "Any TEAE leading to discontinuation of study". Update source footnote to "Source: Listing 16.2.7.2".

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Version 1.0; 17 May 2021

Table 14.3.6 Serious treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part A)

AE006: This output uses shell AE002 [Table 14.3.2]

Programming Notes

Replace footnotes in original shell updating "Patients with at least one TEAE" to "Patients with at least one serious TEAE". Update source footnote to "Source: Listing 16.2.7.4".

Table 14.3.7 Serious treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part A)

AE007: This output uses shell AE003 [Table 14.3.3]

Programming Notes

Use the same template of Table 14.3.3, selecting only the serious TEAEs and update "Patients with at least one TEAE" to "Patients with at least one serious TEAE".

Update source footnote to "Source: Listing 16.2.7.4".

Table 14.3.8 Serious treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity (Safety Analysis Set in Part A)

AE008: This output uses shell AE004 [Table 14.3.4]

Programming Notes

Use the same template of Table 14.3.4, selecting only the serious TEAEs and update "Patients with at least one TEAE" to "Patients with at least one serious TEAE".

Update source footnote to "Source: Listing 16.2.7.4".

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.9 Serious treatment-emergent Adverse Events Leading to Discontinuation of Sutdy by System Organ Class and Preferred Term (Safety Analysis Set in Part A)

AE009: This output uses shell AE005 [Table 14.3.5]

Programming Notes

Use the same template of Table 14.3.5, selecting only the serious TEAEs and update "Any TEAE leading to discontinuation of study" to "Any serious TEAE leading to discontinuation of study". Update source footnote to "Source: Listing 16.2.7.4".

Table 14.3.10 Treatment-emergent Adverse Events with Outcome of Death by System Organ Class and Preferred Term (Safety Analysis Set in Part A)

AE010: This output uses shell AE002 [Table 14.3.2]

Programming Notes

Replace footnotes in original shell updating "Patients with at least one TEAE" to "Patients with a TEAE with outcome of death". Update source footnote to "Source: Listing 16.2.7.3".


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Laboratory

Table 14.3.11 Hematology Laboratroy Data at Screening (Safety Analysis Set in Part A) Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.11

Part A Page X of Y

Hematology Laboratory Data at Screening

(Safety Analysis Set in Part A)

| | | 5400c | 1000μg | 3000μα | 6000p | Placebo |
|---|---|---|---|---|---|---|
| Statistics (N=XX) | (X) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Test #1 (unit) | | | | | | |
| xx x | | XX | ×× | XX | ×× | ×× |
| Mean xx.x | × | ××.× | ×.×. | ××.× | × · · × | × × × |
| SD xx.xx | ×× | xx.xx | xx.xx | xx.xx | xx.xx | ×× · ×× |
| Median xx.x | × | ××.× | ×.×. | ××.× | × · · × | × × × |
| Min, Max xx.x, xx.x | ×.×. | xx.x, xx.x | x.x, xx.x | x.x, xx.x | xx.x, xx.x | xx.x, xx.x |

SD: Standard deviation. n = Number of patients with a screening value. N = Number of patients in the analysis set.

Source: Listing 16.2.8.1

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes: At Screening, blood samples will be taken and tested at the laboratory for the following hematology laboratory tests: Hemoglobin, hematocrit, total white cell count, leukocyte differential count and platelet count. Present in alphabetical order.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.12 Biochemistry Laboratroy Data at Screening (Safety Analysis Set in Part A)

LB002: This output uses shell LB001 [Table 14.3.11]

Programming Notes

Repeat 14.3.11 for Biochemistry (includes creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine transaminase, gamma-glutenthyl transferase, lactate dehydrogenase, creatine kinase, thyroid stimulating hormone, trilodothyronine and thyroxine, glucose, potassium, sodium, and calcium. Present in alphabetical order.
Update source footnote to "Source: Listing 16.2.8.2".


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A Author: Nicholas Roubinis/Jennifer Allsopp

erona Pnarma pic


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.13 Urinalysis Laboratroy Data at Screening (Safety Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.13

Urinalysis Laboratory Data at Screening

(Safety Analysis Set in Part A)

| Laboratory Test (unit) | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
|---|---|---|---|---|---|---|
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Test #1 (unit) | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.x.x) | xx (xx.x) |
| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | (x.xx) xx | (xx.x) |
| 2+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.x.x) | (xxx) xx |
| + 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | (x.xx) xx | (xx.x) |
| 4+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | (x.xx) xx | (x.xx) |
| Total | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Test #2 (unit) | 1 | | | | : | : |

n = Number of patients with a Screening value. N = Number of patients in the analysis set. % = Percentage of patients in each category relative to the total number of patients in the analysis set, with assessments at Screening.

Source: Listing 16.2.8.3

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

At Screening, samples will be taken and tested at the laboratory for the following Urinalyis laboratory tests: Leukocytes esterase, blood, ketones, blitubin, urobilinogen, protein and glucose. If urinalysis on Dipstick is positive for leucocytes and/or blood/hemoglobin, a microscopic examination including erythrocytes, leucocytes, bacteria, casts, epithelial cells and crystals). Present in alphabetical order.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.14 Viral Serology Laboratroy Data at Screening (Safety Analysis Set in Part A)

LB008: This output uses shell LB001 [Table 14.3.11]

Programming Notes Repeat 14.3.13 for Viral Sarology (includes [to confirm post-menopausal status where appropriate] follicle-stimulating hormone [FSH]).. Present in alphabetical order.

Update source footnote to "Source: Listing 16.2.8.4".


Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

Verona Pharma plc


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.15 Hematology Laboratroy Data at Soreening - Normal Reference Ranges (Safety Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.15

Hematology Laboratory Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A)

| Laboratory Test/ | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
|---|---|---|---|---|---|---|
| Reference Range | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Test #1 (unit) | | | | | | |
| Low | xx (xx.x) | xx (xx.x) | (xxx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Normal | xx (xx.x) | xx (xx.x) | (xx.x) xx | xx (xx.x) | (xx.x) | xx (xx.x) |
| High | xx (xx.x) | xx (xx.x) | (xxx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Total | xx (xx.x) | xx (xx.x) | (x.xx) xx | xx (xx.x) | (x.xx) xx | (x.x.x) |
| Test #2 (unit) | : | : | : | : | : | : |

LLN: Lower limit of normal. ULN: Upper limit of normal reference range, n = Number of patients with a Screening value. N = Number of patients in the analysis set. % = Percentage of patients in each category relative to the total number of patients in the analysis set, with assessments at Screening. Reference range classification: Low: < LLN. Normal: >= LLN to <= ULN. High: > ULN.

Source: Listing 16.2.8.1

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes: At Screening, blood samples will be taken and tested at the laboratory for the following laboratory tests: Hemoglobin, hematocrit, total white cell count, leukocyte differential count and platelet count. Present in alphabetical order.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.16 Biochemistry Laboratroy Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A)

LB004: This output uses shell LB003 [Table 14.3.15]

Programming Notes

Repeat Table 14.3.15 for Biochemistry. Table should present these parameters only: Creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine transaminase, gamma-glutamyl transferase, lactate dehydrogenase, creatine kinase, thyroid stimulating hormone, triiodothyronine and thyroxine, glucose, potassium, sodium, and. Present in alphabetical order. Update source footnote to "Source: Listing 16.2.8.2".

Table 14.3.17 Urinalysis Laboratroy Data at Screening - Normal Reference Ranges (Safety Analysis Set in Part A)

LB005: This output uses shell LB003 [Table 14.3.15]

Programming Notes

Repeat Table 14.3.15 for Urinalysis, and update category to 'Wegative' if the results are 'Wormal' or 'Negative', to 'Trace' and 'Positive' if the results are equal to '1+', '2+', '3+', 'or '4+'.

Table should present these parameters only: Leukocytes esterase, occult blood, ketones, bilirubin, urobilinogen, protein and glucose. If urinalysis on Dispative for leucocytes and/or blood/hemoglobin, a microscopic examination including erythrocytes, becoeffed, as peithelial cells and crystals. Present in alphabetical order.

Update source footnote to "Source: Listing 16.2.8.3".

Table 14.3.18 Viral Serology Laboratroy Data at Screening (Safety Analysis Set in Part A)

LB009: This output uses shell LB003 [Table 14.3.15]

Programming Notes

Repeat 14.3.13 for Viral Serology (includes human immunodeficiency virus, hepatitis B and hepatitis C serology). Present in alphabetical order. Note: Patients who received a hepatitis B vaccination and are positive for hepatitis B surface antibody, but are negative for both hepatitis B surface antigen and hepatitis B core antibody, do not need to be excluded from the study. Update source footnote to "Source: Listing 16.2.8.4".

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


OII 1.0; 1 / IMIAY ZUZ1 DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Table 14.3.19 Hematology Laboratroy Data at Screening - Markedly Abnormal Values (Safety Analysis Set in Part A)
Verona Pharma
Protocol: RPL554-MD-201

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Table 14.3.19
Biochemistry Laboratory Data - Markedly Abnormal Values

(Safety Analysis Set in Part A)

| | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
|---|---|---|---|---|---|---|
| Laboratory Test, n (%) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Alanine Aminotransferase (ALT) | | | | | | |
| > 3 x ULN | (xxx) xx | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Alkaline Phosphatase (ALP) | | | | | | |
| > 3 × ULN | xx (xx.x) | xx (xx.x) | (x.xx) xx | (xx.x) | (x.xx) xx | xx (xx.x) |
| Aspartate Aminotransferase (AST) | | | | | | |
| > 3 × ULN | xx (xx.x) | (x.x.x) | xx (xx.x) | xx (xx.x) | (xxx) xx | xx (xx.x) |
| Creatinine | | | | | | |
| > 221 µmol/L | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gamma Glutamyl Transferase (GGT) | | | | | | |
| > 3 × ULN | xx (xx.x) | xx (xx.x) | (xx.x) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bilirubin (TBL) | | | | | | |
| > 3 x ULN | (x.xx) xx | (x.xx) xx | (x.xx) xx | xx (xx.x) | (xxx) xx | xx (xx.x) |

ULN: Upper limit of normal reference range. n = Number of patients with at least one markedly abnormal value. N = Number of patients in the analysis set. % = percentage of patients with at least one markedly abnormal value relative to the total number of patients in the analysis set.

Source: Listing 16.2.8.2

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Table 14.3.20 12-Lead Electrocardiogram Data by Timepoint (Safety Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Page X of Y Part A

12-Lead Electrocardiogram Data by Timepoint (Safety Analysis Set in Part A) Table 14.3.20

| Parameter (Unit) | | | | | | |
|---|---|---|---|---|---|---|
| Timepoint | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Parameter #1 (unit) | | | | | | |
| Pre-dose | | | | | | |
| c | XX | ×× | ×× | ×× | ×× | ×× |
| Mean | x.xx | ×.×× | xx.x | ×.×× | ×.×× | × · · × |
| SD | xx.xx | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | xx.x | x.xx | x.xx | x.xx | x.x. | × |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xxx, xxxx | x.x, xx.x |
| Observed | | | | | | |
| Observed | | | | | | |
| ក [a] | ×× | × | ×× | ×× | ×× | × |
| Mean | xx.x | x.xx | x.xx | x.xx | ×.×. | ×××× |
| SD | xx.xx | xx.xx | xx.xx | ××.×× | xx.xx | xx.xx |
| Median | xx.x | xx | xx.x | xx | x.x. | x . x x |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xxx, xx.x | x.x, xx.x | xx.x, xx.x |
| Change from Pre-dose | | | | | | |
| Mean | xx.x | xx | xx.x | xx | x.x. | x . x x |
| SD | xx.xx | XX.XX | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | x.x. | xx | xx.x | xx | x.x. | xx |
| Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | ostatistics\Documenta | tion\SAP\Verona RE | PL554-MD-201 TLF S | hells v2.0 - Part | A | |
| Author: Nicholas Roubinis/Jennifer Allsopp | fer Allsopp | | | | | Version: 2.0<br>Date: 13JAN2021 |
| | 44-114-114-114-114-114-114-114-114-114- | | | | | |

CONFIDENTIAL Verona Pharma plc

# Clinical Study Report

# RPL554-MD-201

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Version 1.0; 17 May 2021

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Part A Page X of Y

Table 14.3.20

12-Lead Electrocardiogram Data by Timepoint

(Safety Analysis Set in Part A)

| Parameter (Unit) | | | | | | |
|------------------|--------|--------|--------|---------|--------|---------|
| Timepoint | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | - |
| | Биол | Suopg | Биолот | Brinnns | brinne | Flacebo |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

xxx, xxxx

xxx, xxxx

xxxx, xxxx

xx.x, xx.x

xx.x, xx.x

xxx, xxxx

Min, Max

Parameter #2 (unit)

ED: Standard deviation. n = Number of patients who have an assessment available. N = Number of patients in the analysis set. Change from Pre-dose: (Post-dose assessment - Pre-dose assessment).

Source: Listing 16.2.9.2

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes: ECG quantitative assessments include: QTcF Interval (msec), QRS Interval (msec), PR Interval (msec), RR (msec), Heart rate (bpm). Present in alphabetical order. Display for the following timepoints: Pre-dose, 1, 1.5, 2, 4 and 8 hours (all ± 10 minutes)

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Page X of Y Table 14.3.21 12-Lead Electrocardiogram - Shifts from Pre-Dose ECG Assessment by Timepoint (Safety Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

Part A

Table 14.3.21

RPL554 pressurised Metered Dose Inhaler

12-Lead Electrocardiograms - Shifts from Pre-Dose ECG Assessment by Timepoint

Safety Analysis Set

| Timepoint Timepoint Normal Nor | | | | | Category at Timepoint | | |
|---|---|---|---|---|---|---|---|
| xxx Normal xx (xx.x) xx (xx.x) Abnormal NCS xx (xx.x) xx (xx.x) Abnormal CS xx (xx.x) xx (xx.x) xxx xx.xx xx (xx.x) xxx xx (xx.x) xx (xx.x) Abnormal CS xx (xx.x) xx (xx.x) Abnormal CS xx (xx.x) xx (xx.x) Total xx (xx.x) xx (xx.x) Total xx (xx.x) xx (xx.x) | Timepoint<br>Treatment group | z | Pre-dose<br>Category | Normal<br>n (%) | Abnormal NCS<br>n (%) | Abnormal CS<br>n (%) | Total<br>n (%) |
| xxx Normal xx xx.xx xx xx.xx Abnormal CS xx xx.xx xx.xx xx.xx xx.xx Total xx xx.xx xx xx.xx Abnormal NCS xx xx.xx xx xx.xx Abnormal CS xx xx.xx xx xx.xx Total xx xx.xx xx xx.xx Total xx xx xx xx.xx | 1-hour post-dose | | | | | | |
| Abnormal NCS | RPL554 100µg | ××× | Normal | xx (xx.x) | (x.xx) xx | xx (xx.x) | xx (xx.x) |
| Abnormal CS | | | Abnormal NCS | xx (xx.x) | (xx.x) | xx (xx.x) | (xx.x) |
| Total xx (xx.x) xx (xx.x | | | Abnormal CS | xx (xx.x) | (xx.x) | xx (xx.x) | (xx.x) |
| xxx Normal xx xx. (xx.x) xx (xx.x) Abnormal NCS xx (xx.x) xx (xx.x) Abnormal CS xx (xx.x) xx (xx.x) Total xx (xx.x) xx (xx.x) | | | Total | xx (xx.x) | xx (xx.x) | (xx.x) | (xxxx) xx |
| xxx Normal xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx xx <t< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td></t<> | | | | | | | |
| mal NCS xx (xx.x) xx (xx.x) mal CS xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | RPL554 300µg | XXX | Normal | (xx.x) xx | (xxxx) xx | (xx.x) | xx (xx.x) |
| mal CS $xx (xx.x)$ $xx (xx.x)$ $xx (xx.x)$ $xx (xx.x)$ | | | Abnormal NCS | xx (xx.x) | (x.xx) xx | (x.xx) xx | (x.xx) xx |
| xx (xx.x) xx (xx.x) | | | Abnormal CS | xx (xx.x) | (xx.x) | (x.xx) xx | xx (xx.x) |
| | | | Total | (xx.x) xx | (x.xx) xx | xx (xx.x) | (x.xx) xx |

NCS: Not clinically significant, CS: Clinically significant. n = Number of patients in each category with a pre-dose and post-dose assessment. N = Number of patients in the analysis set. % = Percentage of patients in each category relative to the total number of patients in the analysis set, with assessments pre-dose and at the relevant timepoint.

Source: Listing 16.2.9.1

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes: ECG quantitative assessments include: QTcF Interval (msec), QRS Interval (msec), PR Interval (msec), RR (msec), Heart rate (bpm). Display for timepoints: 1, 1.5, 2, 4 and 8 hours (all ± 10 minutes).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Version 1.0; 17 May 2021

Table 14.3.22 Change from Baseline Heart Rate to peak Heart Rate (over 4 hours) After Single Dose (Safety Analysis Set in Part A)

This output uses shell Table 14.2.4

ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. LSMean: Least square mean. LSMean Diff: Least square mean difference. SD: Standard deviation. N = number of patients in the analysis set. Baseline: Pre-dose heart rate. Change from Baseline: Post-dose assessment. — Pre-dose. [a] number of patients with valid values at baseline and timepoints. [b] ANCOVA model is used to model the change from baseline heart rate using baseline heart rate as a continuous fixed effect and actual treatment as categorical fixed effects. [c] number of patients with at least one on treatment value who contributed to the model estimation. \* Indicates a significant p-value (<0.05).

Source: Listing 16.2.9.4

Replace footnotes in original shell with those listed above

Version: 2.0 Date: 13JAN2021 Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Verona Pharma plc


Table 14.3.23 Vital Sign Data - Change from Pre- to Post- dose by Timepoint (Safety Analysis Set in Part A) Verona Pharma Protocol: RPL554-MD-201 Vital Signs

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Table 14.3.23

Vital Sign Data - Change from Pre- to Post- dose by Timepoint

(Safety Analysis Set in Part A)

| N=XX | Parameter (Unit) | | | | | | |
|---|---|---|---|---|---|---|---|
| N=XX | Timepoint | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
| XX | Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| XX | ( ) | | | | | | |
| XX.X XX.X XX.X XX.X XX.XX XX. | Pre-dose | | | | | | |
| XXXX XXXXX XXXXX XXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ជ | ×× | ×× | ×× | ×× | × | ×× |
| XXXXX XXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Mean | × : × × | ××× | ××× | × × × | ×.× | ××× |
| xx | SD | xx.xx | xx.xx | xx.xx | ××.×× | xx.xx | ××.×× |
| xx | Median | × : × × | ×××× | × | ××× | ×.×× | ×××× |
| XX | Min, Max | xxx, xxx | x.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | x.x, xx.x |
| xx | Observed | | | | | | |
| XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX XX.XX <th< td=""><td>п</td><td>××</td><td>××</td><td>××</td><td>××</td><td>××</td><td>××</td></th<> | п | ×× | ×× | ×× | ×× | ×× | ×× |
| x.xx | Mean | xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| xx.x | SD | ××.×× | ×× · × | ××.×× | xx.xx | xx.xx | ××. ×× |
| <pre>c, xx.x</pre> | Median | × × | x.xx | × | x. x. | x . x x | x.xx |
| XX.X XX.X XX.XX XX.X X | Min, Max | xxx, xxx | xx.x, xx.x | x.x, xx.x | xxx, xx.x | x.x, xx.x | x.xx ,x.xx |
| x.xx | Change from Pre-dose | | | | | | |
| x.xx | Mean | × | ×.×. | × × | ×.×. | ×.×. | ×. ×. |
| xx.x xx.x xx.x xx.x xx.x xx.x xx.x xx. | SD | xx.xx | ××. ×× | xx.xx | xx.xx | xx.xx | ××.×× |
| \Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | Median | ×.×. | x.xx | ××.× | x.x.x | ××.× | x.x. |
| | cument: Z:\RPL554\EZAA8488\Bios | tatistics\Documenta | tion\SAP\Verona I | RPL554-MD-201 TLF | Shells v2.0 - Part | A | |
| | Author. Nicholse Bombinis /Jannifar Alleonn | ממספוות אי | | | | | Version: 2.0 |

CONFIDENTIAL Verona Pharma plc

# Clinical Study Report

RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3 Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Table 14.3.23

Part A Page X of Y

Vital Sign Data - Change from Pre- to Post- dose by Timepoint

(Safety Analysis Set in Part A)

| Parameter (Unit) | | | | | | |
|---|---|---|---|---|---|---|
| Timepoint | RPL554<br>100µg | RPL554<br>300µg | RPL554<br>1000µg | RPL554<br>3000µg | RPL554<br>6000µg | Placebo |
| Statistics | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Min, Max | xxx, xx.x | x.x, xx.x | x.x, xx.x | x.x, xx.x | xx.x, xx.x | x.x, xx.x |
| 2-hours post-dose | | | | | | |

SD: Standard deviation. n = Number of patients who have an assessment available. N = Number of patients in the analysis set. Change from Pre-dose: (Post-dose assessment - Pre-dose assessment).

Source: Listing 16.2.9.3

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes: Vital signs assessments include: Systolic blood pressure, diastolic blood pressure and pulse rate. Present in alphabetical order. Display for the following timepoints: Pre-dose, 1, 1.5, 2, 4, 8, 12 and 24 hours (all ± 10 minutes).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Table 14.3.24 Vital Sign Data - Markedly Abnormal Values (Safety Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Part A Page X of Y

> Vital Sign Data - Markedly Abnormal Values Safety Analysis Set Table 14.3.24

| | RPL554<br>100µg | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | RPL554 6000µg | Placebo |
|---|---|---|---|---|---|---|
| Vital Sign Parameter | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| Systolic Blood Pressure (mmHg), n (%) | | | | | | |
| n [a] | ×× | ×× | ×× | ×× | ×× | ×× |
| Value <=90 | xx (xx.x) | (x.xx) | xx (xx.x) | (xx.x) | xx (xx.x) | (xx.x) |
| A decrease from baseline of >=40 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.x.) xx |
| Value >=180 | xx (xx.x) | (x.x.x) | xx (xx.x) | (xx.x) | xx (xx.x) | (xx.x) |
| An increase from baseline of >=40 | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) |
| Diastolic Blood Pressure (mmHg), n (%) | | | | | | |
| n [a] | ×× | ×× | ×× | ×× | ×× | ×× |
| Value <=50 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| A decrease from baseline of $>=20$ | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Value >=105 | xx (xx.x) | xx (xx.x) | (x.x.x) xx | (xx.x) | (xx.x) | (x.xx) xx |
| An increase from baseline of $>=20$ | (x.xx) xx | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) | (xx.x) |
| Pulse Rate (bpm), n (%) | | | | | | |
| n [a] | ×× | ×× | ×× | ×× | ×× | ×× |
| Value <=50 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| A decrease from baseline of $>=30$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Value >=110 | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) xx | xx (xx.x) | xx (xx.x) |
| An increase from baseline of >=30 | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) |
| Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part | tics\Documenta | tion\SAP\Verona I | RPL554-MD-201 TLF | Shells v2.0 - Par | t A | |
| Author: Nicholas Roubinis/Jennifer Allsopp | ddos | | | | | Version: 2.0<br>Date: 13JAN2021 |


Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

Table 14.3.24

Vital Sign Data - Markedly Abnormal Values Safety Analysis Set

| | RPL554 | | | | | |
|---|---|---|---|---|---|---|
| | 100µg | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | RPL554 6000µg | Placebo |
| /ital Sign Parameter | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

bpm: beats per minute. mmHg: millimeters mercury. [a] n = Number of patients with a baseline value and post-baseline value. Baseline and post-baseline value would be needed for criteria relating to an increase/decrease from baeline. N = Number of patients in the analysis set. % = percentages are based on n.

Source: Listing 16.2.9.3

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

 Verona Pharma plc

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Table 14.3.25 Change from Baseline Pulse Rate to Peak Pulse Rate (over 4 hours) After Single Dose (Safety Analysis Set in Part A)

This output uses shell Table 14.2.4

ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. LSWean: Least square mean. LSWean Difference: Leat square mean difference. SD: Standard deviation. N = number of patients in the analysis set. Baseline: Per-dose pulse rate. Change from Baseline mean dimepoints. Pb] ANCOVA model is used to model the change from baseline pulse rate using baseline pulse rate as a continuous fixed effect and actual treatment as categorical fixed effects. [c] number of patients with at least one on treatment value who contributed to the model estimation. \* Indicates a significant p-value (<0.05).

Source: Listing 16.2.9.4

Programming Notes:

Replace footnotes in original shell with those listed above

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

## Version 1.0; 17 May 2021

## DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Physical Examination

Table 14.3.26 Physical Examination Data by Timepoint (Safety Analysis Set in Part A)

Page X of Y Part A

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.26

Physical Examination Data by Timepoint

(Safety Analysis Set in Part A)

| Physical Examination: <full brief=""></full> | | | | | | |
|---|---|---|---|---|---|---|
| Assessment | | | | | | |
| + \$ | RPL554 | RPL554 | RPL554 | RPL554 | RPL554 | |
| TIMEDOTING | 100µg | 300µg | 1000µg | 3000µg | 6000pg | Placebo |
| Category | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) | (N=XX) |

Abdomen (liver and spleen)

xx (xx.x) (xx.x) xx Abnormal NCS Abnormal CS Pre-dose Normal

(xxxx) xx xx (xx.x) xx (xx.x)

xx (xx.x) xx (xx.x) xx (xx.x)

xx (xx.x) xx (xx.x) xx (xx.x)

Cardiovascular system

Pre-dose

CS = Clinically significant. NCS = Not clinically significant. n = Number of patients who have an assessment available at the relevant timepoint. N = Total number of patients in the analysis set.

Source: Listing 16.2.9.5 and 16.2.9.6

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

• Full Physical Examination assessments include: Abdomen [liver and spleen], Cardiovascular system, Extremities, Lymph nodes, Neurological system, Nose, Throat, Respiratory system, Skin, Thyroid gland. Present in alphabetical order.

• Brief Physical Examination assessments include: Abdomen (liver and spleen), Cardiovascular system, Respiratory system, Skin. Present in alphabetical order.

• Display for the following timepoints: Full Physical Examination: Screening and Brief Physical Examination: Pre-dose.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

#### Figures

Figure 14.2.1 Geometric Mean of ratios of Average FEV, (over 4 hours) to pre-dose FEV, by Treatment (Full Analysis Set in Part A)

EFF09: This output uses shell EFF008 [Figure 14.2.3]

Programming Notes

Use template of figure 14.2.3, adjusting for Average  ${\it FEV}_1$  (over 4 hours).

Figure 14.2.2 Geometric Mean of ratios of Average FEV; (over 12 hours) to pre-dose FEV; by Treatment (Full Analysis Set in Part A)

EFF10: This output uses shell EFF008 [Figure 14.2.3]

Programming Notes

Use template of figure 14.2.3, adjusting for Average  $\ensuremath{\operatorname{FEV}}_1$  (over 12 hours).

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


## Version 1.0; 17 May 2021

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Page X of Y Figure 14.2.3 Geometric Mean of ratios to Peak FEV; (over 4 hours) to pre-dose FEV; by Treatment (Full Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Part A

Geometric Mean of ratios of Peak FEV1 (over 4 hours) to pre-dose FEV1 by Treatment (Full Analysis Set in Part A) Figure 14.2.3



FEVI: Forced expiratory volumn in 1 second. Pre-dose FEVI: Average of pre-dose FEVI assessed immediately pre-dose (within 5 minutes) and 1 hour pre-dose (within 5 minutes). Bottom and top whiskers: 95% lower confidence limit and 95% upper confidence limit. Bar: Geometric means of the ratio to pre-dose. ANCOVA model is used to model the change from pre-dose FEVI using pre-dose FEVI as a continuous fixed effect and planned treatment as categorical fixed effects.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Above is an example. Display for all treatment groups in Part A in ascending order (RPL554 100µg, RPL554 300µg, RPL554 1000µg, RPL554 6000µg) and then placebo. For each treatment group present the LSMean and SEM (standard error of the mean).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Figure 14.2.4 Mean Change from pre-dose FEV; during spirometry over Time by Treatment (Full Analysis Set in Part A)
Portocol: PEP5554-MD-201
RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Mean Change from pre-dose FEV, during spirometry over Time by Treatment (Full Analysis Set in Part A)



Means are calculated on the observed data.

Pre-dose: the highest FEV1 result collected immediately pre-dose (within 5 minutes).

Source: Listing 16.2.6.1

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Above is an example. Display for all treatment groups and placebo. For each treatment group present the Mean change from baseline. Display for the following time points on Day 1: 5 minutes, 15 minutes, 10 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 8 hours, 11 hours and 12 hours. On the x-axis present actual time scale (in spacing of timepoints).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

## Clinical Study Report

Version 1.0; 17 May 2021 RPL554-MD-201

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Figure 14.2.5 Change from Pre-dose FEV1 over Time by Treatment by Subject (Full Analysis Set in Part A)

EFF09: This output uses shell EFF009 [Figure 14.2.4]

Programming Notes

Use template of figure 14.2.4.
Update to have 1 page per treatment group with "Planned Treatment:" displayed above the figure on the left.
Present each partient for that treatment. Do no include a legend so that unblinding does not occur on a subject-level.
Update y-axis tills to "Change from pre-dose FEVI (L)".
Include the following footnote: "Pre-dose: the average of the FEVI pre-dose assessments collected on Day I (within 60 and 5 minutes)."


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Figure 14.3.1 Mean Change from Pre-dose Heart Rate to Peak Heart Rate (over 4 hours) by Treatment (Safety Analysis Set in Part A)

This output uses shell Figure 14.2.1

Pre-dose heart rate: The heart rate value assessed immediately before administration. Bottom and top whiskers: 95% lower confidence and 95% upper confidence limit. Bar: Results on orginal scale. ANCOVA model is used to model the change from pre-dose heart rate using pre-dose heart rate as a continuous fixed effect, and actual treatment as categorical fixed effects.

Programming Notes

Use template of figure 14.2.1, adjusting for ECG assessment = heart rate. Update source footnote to "Source: Listing 16.2.9.4". Replace footnotes in original shell with those listed above

Figure 14.3.2 Mean Change from Pre-dose in Heart Rate over Time by Treatment (Safety Analysis Set in Part A)

This output uses shell Figure 14.2.4

Means are calculated on the observed data. Pre-dose: the pre-dose assessment collected of day 1.

Programming Notes

Display for all treatment groups and placebo. For each treatment group present the Mean change from baseline. Display for the following time points on Day 1: 1 hour, 2 hours, 4 hours and 8 hours. Update source footnote to "Source: Listing 16.2.9.2". Replace footnotes in original shell with those listed above

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Figure 14.3.3 Mean Change from Pre-dose Pulse Rate to Peak Pulse Rate (over 4 hours) by Treatment (Safety Analysis Set in Part A)

This output uses shell Figure 14.2.1

Pre-dose pulse rate: The pulse rate value assessed immediately before administration. Bottom and top whiskers: 95% lower confidence and 95% upper confidence limit. Bar: Results on orginal scale. ANCOVA model is used to model the change from pre-dose pulse rate using pre-dose pulse rate as a continuous fixed effect, and actual treatment as categorical fixed effects.

Programming Notes:

Use template of figure 14.2.1, adjusting for vital sign assessment = pulse rate. Update source footnote to "Source: Listing 16.2.9.4". Replace footnotes in original shell with those listed above

Figure 14.3.4 Mean Change from Pre-dose in Pulse Rate over Time by Treatment (Safety Analysis Set in Part A)

This output uses shell Figure 14.2.4

Programming Notes:

Display for all treatment groups and placebo. For each treatment group present the Mean change from baseline. Bisplay for the following time points on Day 1: 1 hour, 2 hours, 4 hours, 8 hours, 12 hours, Day 2: 24 hours. Update source footnote to "Source: Listing 16.2.9.3".
Replace footnotes in original shell with those listed above

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

 $\textbf{Listings} \\ \textbf{Listing 16.2.1.1 Completed/Discontinued Patients (All Randomized Analysis Set in Part A)} \\$ Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y

Part A

Listing 16.2.1.1

Completed/Discontinued Patients

(All Randomized Analysis Set in Part A)

Treatment group: <PPL554 100hg/RPL554 300hg/RPL554 1000hg/RPL554 300hg/RPL554 6000hg/PPLacebo>

| Date of completion/discontinuation/Study day | DDMMYYYY/xx |
|--------------------------------------------------------|-------------|
| Discontinued<br>between Part A<br>and Part B | ×× |
| Part A<br>Treatment<br>discontinued | ×× |
| Completed Part<br>A/Primary reason<br>if not completed | No/XXXXXX |
| Randomization<br>date/Study day | DDMMYYYY/xx |
| Informed<br>consent<br>date/Study<br>day | DDMMYYYY/xx |
| Patient ID | XXXXXXX |

Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:NM

Programming Notes Order by treatment group (as per shell) and within group by patient ID.

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.2.1 Protocol Deviations (All Randomized Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.2.1

Protocol Deviations

(All Randomized Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| | ı |
|--------------------------|---------------|
| Severity | XXXXXXXXXX |
| Type of<br>deviation | XXXXXXXXXX |
| Protocol<br>deviation | XXXXXXXXXX |
| Deviation date/Study Day | DDMMMYYYY/xx |
| Age/Sex/Race | XXXXXXX/X/XX |
| Patient ID | XXXXXXXXXXXXX |

As: Native Asian. B1: Black or African American. F: Female. Ia: American Indian or Alaskan. M: Male. Ot: Other. PI: Native Hawaiian or Pacific Islanders. Un: Unknown. W: White. Age (years): As calculated relative to informed consent date. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell) and within group by patient ID and then the deviation date.


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.3.1 Patients Excluded from Analysis Sets (All Randomized Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

(All Randomized Analysis Set in Part A) Patient Excluded from Analysis Sets Listing 16.2.3.1

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| XXXXXXX 47/M/W PK XXXXXXX 67/M/B1 SAF | Patient ID | Age/Sex/Race | Affected analysis set |
|---|---|---|---|
| 67/M/B1 | XXXXXXXX | 47 / M/W | PK |
| | XXXXXXX | 67/M/B1 | SAF |

As: Native Asian. Bl: Black or African American. eCRF: Electronic case report form. F: Female. Ia: American Indian or Alaskan. M: Male. Ot: Other. PI: Native Hawaiian or Pacific Islanders. Un: Unknown. W: White. Age (years): As calculated relative to informed consent date. All measurements listed above are measured at Screening on the Demography eCRF.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell) and within group by patient ID. Print "No patient excluded from any analysis set" if the listing has no observations.


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.4.1 Demographic Characteristics (All Randomized Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.4.1

Demographic Characteristics

(All Randomized Analysis Set in Part A)

| | Childbearing<br>potential | × | NA |
|---|---|---|---|
| | Re-<br>screened<br>patient | × | × |
| | BMI<br>(kg/m²) | XX. | × |
| 10µg/Placebo> | Height<br>(cm) | ×× | XXX |
| 10µg/RPL554 600 | Weight<br>(kg) | ×× | × |
| Treatment group: <rpl554 1000µg="" 100µg="" 3000µg="" 300µg="" 6000µg="" placebo="" rpl554=""></rpl554> | Ethnicity | White-<br>White/Caucasian/European<br>Heritage | White-<br>White/Caucasian/European<br>Heritage |
| 100µg/RPL554 3 | Country Age/Sex/Race | 62/F/W | M/W/L9 |
| roup: <rpl554< td=""><td>Country</td><td>USA</td><td>USA</td></rpl554<> | Country | USA | USA |
| Treatment g | Patient ID | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXX |

As: Native Asian. B1: Black or African American. BMI: Body mass index. eCRF: Electronic case report form. F: Female. Ia: American Indian or Alaska. M: Male. NA: Not applicable. Ot: Other. Pi: Native Hawaiian or Pacific Islanders. Un: Unknown. W: White. Age (years): As calculated relative to informed consent date. BMI (kg/m²) = Weight (kg) / Height (m)². All measurements listed above are measured at Screening on the Demography eCRF.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Order by treatment group (as per shell) and within group by patient ID.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.4.2 Screening Disease Characteristics (All Randomized Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

(All Randomized Analysis Set in Part A) Screening Disease Characteristics Listing 16.2.4.2

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/Placebo>

| Patient | Bi | Bronchodilator FEV <sub>1</sub> | lator | FEV1 | FVC (L) | (L) | FEV | FEV1/FVC | Reversibility FEV1 | 1<br>1 | Assessment<br>performed<br>with four<br>puffs of | Met<br>reversibility |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age/Sex/Rad | ce (I) | (L) | (%) | (%) | Pre | Post | Pre | Post | mT | 9/0 | albuterol | test criteria? |
| XXX/X/XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XXX | XXX |

As: Native Asian. Bl: Black or African American. eCRF: Electronic case report form. F: Female. FEV; Forced expired volume in 1 second. FVC: Forced vital capacity. Ia: American Indian or Alaskan. Ot: Other. PI: Native Hawaiian or Pacific Islanders. Un: Unknown. W: White. Age (years): As calculated relative to informed consent date. Pre-, post-bronchodilator and reversibility values are the results of the screening reversibility test.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell) and within group by patient  $\ensuremath{\mathsf{ID}}.$ 


Verona Pharma plc


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.4.3 COPD and Smoking History (All Randomized Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.4.3 COPD and Smoking History

(All Randomized Analysis Set in Part A)

Smoking History

| ı | |
|------------------------------------------------------|-------------|
| Smoking exposure (pack-years) | XX |
| Number of<br>Years<br>smoking | XX |
| Number of<br>packs<br>per day | XX |
| Smoking<br>category | Current |
| Bronchiti<br>s?/<br>Emphysema<br>? | Yes/Yes |
| Date of most<br>recent<br>exacerbation/S<br>tudy day | DDMMYYYY/xx |
| Duration of COPD (years) (time since diagnosis) | XX.X |
| Date of COPD<br>first<br>diagnosed | DDMMMYYYY |
| Patient ID | XXXXXXX |

COPD: Chronic Obstructive Pulmonary Disease. Smoking exposure (pack-years) = Number of packs per day \* Number of years smoking, for patients with a smoking history or a current smoker. Study day: Day relative to day of the first dose of study medication. Duration of COPD (years) (time since diagnosis) = Randomization date - date COPD first diagnosed.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Order by treatment group (as per shell) and within group by patient ID.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.4.4 Medical History (All Randomized Analysis Set in Part A)
Verona Pharma
Protocol: RPL554-MD-201
RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Listing 16.2.4.4

Medical History

(All Randomized Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/RPL554 6000µg/Placebo>

| Study day | DDMMMYYYY/xx |
|---------------------------|----------------------------------------|
| Study day | DDMMMYYYY/xx |
| SOC/PT | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| Medical history diagnosis | XXXXXXXXXXXXXX |
| Patient ID | XXXXXXXX |

End date/

Start date/

MedDRA: Medical Dictionary for Regulatory Activities. PT: Preferred Term. SOC: System Organ Class. Medical history: Coded using MedDRA (Version 21.0). Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Order by treatment group (as per shell) and within group by patient ID.


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.4.5 Surgical Procedure History (All Randomized Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

> Surgical Procedure History Listing 16.2.4.5

(All Randomized Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| End date of<br>procedure/<br>Study day | DDMMYYYY/xx |
|------------------------------------------|------------------|
| Start date of<br>procedure/<br>Study day | DDMMMYYYY/xx |
| Purpose of procedure | XXXXXXXXXXXX |
| Reported name of procedure | XXXXXXXXXXXXXXXX |
| Patient ID | XXXXXXXXX |

Surgical procedure history: Coded using MedDRA (Version 21.0). Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes:

Order by treatment group (as per shell) and within group by patient ID.

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.4.6 Prior and Concomitant Medications (All Randomized Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

(All Randomized Analysis Set in Part A) Prior and Concomitant Medications Listing 16.2.4.6

Treatment group: <PPL554 100ug/RPL554 300ug/RPL554 100ug/RPL554 3000ug/RPL554 600ug/PPL554 600ug/Placebo>

| Patient ID | Start date<br>(Study day)/<br>End date<br>(Study day) | Prior?[a]/<br>Concomitant?[b] | System organ class/<br>Preferred term/<br>Reported term | Indication | Dose<br>(Unit) | Frequency | Route |
|---|---|---|---|---|---|---|---|
| XXXXX | DDMMMYYYYY (xx) / (xx) / | Prior | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | ×××××× | (xx)<br>(xx) | × | ××× |
| | DDMMMYYYY<br>(xx)/<br>ongoing | Prior/Concomitant | /************************************* | ×××××× | (xx) | × | ×× |
| | DDMMMYYYY (xx)/ | Concomitant | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | ×××××× | (xx) | × | ××× |

[a] Medications which started and stopped in the 3 months prior to the single dose of study medication [b] Medication with onset date on or after the single dose of study medication and ended on or after the single dose of study medication or were organing at the end of Part A. A patient can report more than one concomitant medication with the same preferred term. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.5.1 Drug Exposure and Accountability (All Randomized Analysis Set in Part A)
Verona Pharma
Protocol: RPL554-MD-201
RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Listing 16.2.5.1

Drug Exposure and Accountability
(All Randomized Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/RPL554 6000µg/RPL6000

| Date of Part A completion/<br>discontinuation/Study day | DDMMYYYY/xx |
|---------------------------------------------------------|--------------|
| Start time<br>of inhalations | нн:мм |
| Dosing date/<br>Study day | DDMMMYYYY/xx |
| Patient ID | XXXXXXXX |

Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.6.1 Spirometry: FEV1 Results (Full Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Listing 16.2.6.1

(Full Analysis Set in Part A) Spirometry: FEV1 Results

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/Placebo>

| | | Assessment | | | | |
|---|---|---|---|---|---|---|
| | | performed/ | | Capable of | | |
| | | Date and | Refrained | withdrawing from | | |
| | | time/ | from | long acting | FEV1 measurement | |
| Patient ID | Timepoint | Study day | smoking | bronchodilators | (L) | Predicted FEV1 (%) |
| XXXXX | XXXXXX | XX/DDMMYYY<br>HH:MM/xx | XX | XX | X.XXX | XX.X |
| | XXXXXX | | | | | |

FEV: Forced expiratory volume in 1 second. FEV; pre-dose assessment (-5 minutes) collected at visit of interest. Study day: Day relative to day of the first dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes
The assessment timepoints can be Pre PFT, Post PFT, Pre PFT -60 min, Immediately Predose, Post PFT 5min, 15min, 30min, 1h, 1.5h, 2h, 4h, 8h, 11h, 12h and EOS: The minutes from dosing is the difference between the Date/Time of assessments (from dataset CDM.I.SSW/CDM.R.SSW) and the Date/Time of Dosing (from dataset CDM.EX). Order by treatment group (as per shell) and within group by patient ID.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.6.2 Spirometry: FEV1 Derived Measurements (Full Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Spirometry: FEV1 Derived Measurements (Full Analysis Set in Part A) Listing 16.2.6.2

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/Placebo>

| XXX X XXX X XXX X XXX X XXX X XXX X XXX X |
|-------------------------------------------|
| XX/DDMMXYY/xx |

AUC: Area under the curve. FEV1: Forced expiratory volume in 1 second. FEV1 pre-dose assessment (-5 minutes) collected at visit of interest. Peak FEV1 = Maximum post-dose value among the values collected up to timepoint of interest hours. Average FEV1 AUC: AUC of the FY1 values divided by the length of the time (in hours) interval of interest (per visit). Study day: Day relative to day of the rising dose of study medication. \* when a subject has taken rescue medication less than 8 or 6 hours (for protocol version 1 or 2 respectively) prior to study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

The assessment timepoints can be Pre PFT, Post PFT, Pre PFT -60 min, Immediately Pre-dose, Post PFT 5min, 15min, 10min, 11.5h, 2h, 4h, 8h, 11h, 12h and EOS. The minutes from dosing is the difference between the Date/Time of assessments (from dataset CDM.SPIRO) and the Date/Time of Dosing (from dataset CDM.EX) Order by treatment group (as per shell) and within group by patient ID. In the "Average FEM! (over 12 hours)" \* any results where a subject has taken rescue medication less than 8 or 6 hours (for protocol version 1 or 2 respectively) prior to study medication. Programming Notes

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.6.3 Rescue Medications Taken at Site (All Randomized Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

> (All Randomized Analysis Set in Part A) Rescue Medications Taken at Site Listing 16.2.6.3

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

Number of Albuterol or Salbuterol puffs taken/ Number of Ipratropium puffs taken XX/YY Date/time of administration/ Study day DDMMMYYYY/ HH:MM/xx Medication name Patient ID XXXX/XXXX

Rescue medications = Short acting bronchodilators used to relieve i.e., rescue symptoms immediately. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:NM

Programming Notes

Order by treatment group (as per shell) and within group by patient ID and visit.

CONFIDENTIAL Verona Pharma plc


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

### Clinical Study Report

Version 1.0; 17 May 2021 RPL554-MD-201

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.6.4 Rescue Medication Taken between Visits (All Randomized Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Rescue Medications Taken between Visits (All Randomized Analysis Set in Part A) Listing 16.2.6.4

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/RPL6000

| | Dispensed rescue | medication weight | / (b) | Collected weight | (b) | XX.X/ | XX.XX |
|---|---|---|---|---|---|---|---|
| | | | | | iispensed/collected Reason canister not dispensed/collected | XXXXXXX/ | XXXXXXX |
| | | | Date and time | canister | dispensed/collected | DDMMMYYYY/HH:MM/ | DDMMMYYYY/HH:MM |
| Rescue | medication | canister | dispensed?/ | collected? | (X/N) | X/X | |
| | | | | Inhaler | number | XX | |
| | | | | | Patient ID | | |

Rescue medications = Short acting bronchodilators used to relieve i.e., rescue symptoms immediately.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell) and within group by patient ID and visit.


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.7.1 All Adverse Events (Safety Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

> All Adverse Events Listing 16.2.7.1

(Safety Analysis Set in Part A)

Treatment group: <PPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/Placebo>

| , | ı |
|-------------------------------------------------------|-------------------|
| Blind<br>broken | Yes |
| Discontinued from study | Yes |
| Treatmen<br>t<br>given | Yes |
| Chronicit<br>Y<br>[h] | X/X/XX |
| Out<br>[g] | Rslv |
| Ser<br>[f] | N |
| Act<br>[e] | NC |
| Rel<br>[d] | Y |
| Sev<br>[c] | IM |
| start/End<br>date<br>or ongoing<br>(Study<br>day) [b] | AXXXXMMMQQ |
| SOC/PT/Reported<br>term [a] | XXXXX/XXXXX/XXXXX |
| Study day<br>of first<br>treatment | XX |
| Patient<br>ID | XXXXX |

PT: Preferred term. SOC: System organ class.

[a] An asterisk "\*" indicates a non-treatment-emergent adverse event.

[b] Study day: Day relative to day of the single dose of study medication.

[c] Severity: MI=Mild, MO=Moderate, SE=Severe.

[d] Related to study drug.

[e] Action taken with respect to study drug: NC = Dose not changed, DI = Drug Interrupted DW = Drug withdrawn, OT = Other, NA = Not

Applicable.

[f] Serious AE.

[g] Outcome: Fatal = Fatal, NRslv = Not recovered/not resolved, Rslv = Recovered/Resolved, RslvS = Recovered/Resolved with sequelae, Recovering/Resolving = RslvG, Unk = Unknown.

[h] S = Single Occasion, I = Intermittent, P = Persistent. SOCs and PTs are coded using the MedDRA (Version 21.0).

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment by patient ID, adverse event start date and adverse event end date (in that order).

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.7.2 Treatment-emergent Adverse Events Leading to Study Discontinuation (Safety Analysis Set in Part A)

L017: This output uses shell L016 [Listing 16.2.7.1]

Listing 16.2.7.3 Treatment-emergent Adverce Events Leading to Death (Safety Analysis Set in Part A)

L018: This output uses shell L016 [Listing 16.2.7.1]

Listing 16.2.7.4 Serious Treatment-emergent Adverse Events (Safety Analysis Set in Part A)

L019: This output uses shell L016 [Listing 16.2.7.1]

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.7.5 Serious Treatment-emergent Adverse Events - Details (Safety Analysis Set in Part A) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Page X of Y Part A

> Serious Treatment-emergent Adverse Events - Details (Safety Analysis Set in Part A) Listing 16.2.7.5

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/RPL6000

| Patient ID | SOC/PT/<br>Reported Term | SAE details | Answer |
|---|---|---|---|
| XXXXXXXXXX | XXXXXX/XXXXXX/XXXXXX | Date Investigator became aware of SAE | DDMMMYYYY |
| | | Death | XXXXX |
| | | Life-threatening | XXXXX |
| | | Initial or prolonged hospitalization | XXXXX |
| | | Date of admission (DD MMM YYYY) | DDMMMYYYY |
| | | Date of discharge (DD MMM YYYY) | DDMMMYYYY |
| | | Persistent or significant disability/incapacity | XXXXX |
| | | Congenital anomaly/birth defect | XXXXX |
| | | Occurred with overdose | XXXXX |
| | | Other medically important event | XXXXX |
| | | Was the SAE caused by other medication? (e.g. Concomitant medication, background medication, rescue medication) | XXXXX |
| | | If Yes, Please Specify | XXXXX |
| | | Was the SAE caused by study procedure(s)? | XXXXX |
| | | If Yes, Please Specify | XXXXX |
| | | Describe treatment for event including medications (1) | XXXXX |
| | | Describe treatment for event including medications (2) | XXXXX |
| | | Describe treatment for event including medications (3) | XXXXX |
| | | List all diagnostic tests that were done to confirm event (1) | XXXXX |
| | | List all diagnostic tests that were done to confirm event (2) | XXXXX |
| | | List all diagnostic tests that were done to confirm event (3) | XXXXX |
| | | Description of SAE/narrative | XXXXX |
| | | Additional information | XXXXX |
| Document: Z:\RPL554' | | EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A | |
| Author: Nicholas Rol | Author: Nicholas Roubinis/Jennifer Allsopp | | Date: 13JAN2021 |


Verona Pharma plc


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Verona Pharma Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Listing 16.2.7.5

Serious Treatment-emergent Adverse Events - Details

(Safety Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/PPLeebo>

| Answer |
|--------------------------|
| SAE details |
| SOC/PT/<br>Reported Term |
| Patient ID |

PT: Preferred Term. SAE: Serious Adverse Event. SOC: System Organ Class. SOCs and PTs are coded using the MedDRA (Version 21.0).

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.


Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.8.1 Hematology (Safety Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

Listing 16.2.8.1

(Safety Analysis Set in Part A) Hematology

Treatment group: <PPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/Placebo>

| Change<br>from<br>Baseline | XX.X |
|-----------------------------------------|-----------------------|
| Value (unit)<br>L/H [a] | XX (unit) |
| Date/Time of assessment/<br>Study day | DDMMYYYY/HH:MM/<br>xx |
| Timepoint | Scr |
| Reference<br>Range<br>(Lower-<br>Upper) | XXX - XXX |
| Parameter | Hemoglobin |
| Patient ID | XXXXXXXXXXX |

Scr: Screening. [a] L = Below low normal range. H = Above high normal range. \* = Markedly abnormal values. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Add a symbol '\*' next to the value to identify markedly abnormal values. Order by treatment group (as per shell), hematology parameter (in alphabetical order) and by patient ID.

Listing 16.2.8.2 Biochemistry (Safety Analysis Set in Part A)

L022: This output uses shell L021 [Listing 16.2.8.1]

Scr: Screening. [a] L = Below lower limit of reference range. H = Above upper limit of reference range. Study day: Day relative to day of the single dose of study medication.

\* = Markedly abnormal value (refer to section 16.2.1 of the statistical analysis plan for the markedly abnormal criteria).

Programming Notes

Replace footnotes with those above.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.8.3 Urinalysis (Safety Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

> Listing 16.2.8.3 Urinalysis

(Safety Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/Placebo>

| Result [a] | NEGATIVE (N) | TRACE (T) | 1+ (P) |
|---|---|---|---|
| Date/Time of assessment/<br>Study day | DDMMMYYYY/HH:MM/xx | DDMMMYYYY/HH:MM/xx | DDMMMYYYY/HH:MM/xx |
| Timepoint | Screening | 1 | į |
| Parameter | Bilirubin | | |
| Patient ID | XXXXXXXXXXX | | |

Scr: Screening. [a] Category assigned and used in the shift table: N = Normal or 'Negative'; T = '"race' P = '1+','2+','3+',' or '4+'.

The flag appears only for the following parameters: Leucocyte Esterase, Bilirubin, Glucose, Ketones, Occult blood, Protein and Urobilinogen. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell), urinalysis parameter (in alphabetical order) and by patient ID.

Listing 16.2.8.4 Viral Serology (Safety Analysis Set in Part A)

L022: This output uses shell L021 [Listing 16.2.8.3]

Programming Notes

Replace footnotes with those related to Viral Serology

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

## Version 1.0; 17 May 2021

# DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.1 Electrocardiogram Local Reading Overall Evaluation (Safety Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Electrocardiogram Local Reading Overall Evaluation (Safety Analysis Set in Part A) Listing 16.2.9.1

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| Abnormal | Significant | X |
|--------------|----------------------|-------------------|
| Overall ECG | Evaluation | Normal |
| Date/Time of | assessment/Study day | DDMMYYYY/HH:MM/xx |
| | Day/Timepoint | XXXX/XXXX |
| | Patient ID | XXXXXXXXXXX |

EGG: Electrocardiogram. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell), within group by patient ID and then by timepoint.

Version: 2.0 Date: 13JAN2021 Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.2 12-Lead ECG (Safety Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

> (Safety Analysis Set in Part A) Listing 16.2.9.2 12-lead ECG

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| ay/Timepo<br>XXX | Date/Time of int assessment/Study day ECG parameter (unit) Result Baseline CFB | DDWMMYYY/HH:MM/xx HR (bpm) XX.X XX.X | RR interval (msec) XX.X XX.X XX.X | PR interval (msec) XX.X XX.X XX.X | QRS duration (msec) XX.X XX.X XX.X | QT interval (msec) XX.X XX.X XX.X | Bazett's QTc (msec) XX.X XX.X XX.X | Fridericia's QTc (msec) XX.X XX.X XX.X |
|---|---|---|---|---|---|---|---|---|
| 2 0 | Date/Time of assessment/Study da | | | | | | | |

bpm: beats per minute. CFB: Change from baseline. ECG: Electrocardiogram. HR: Heart rate. QTcB: QT interval using Bazett's correction formula. msec: milliseconds. QTcF: QT interval using Fridericia's correction formula. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell), within group by patient ID and then by timepoint.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.3 Vital Signs (Safety Analysis Set in Part A) Verona Pharma Protocol: RPLS54-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Listing 16.2.9.3

Vital Signs

(Safety Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/Placebo>

| Markedly<br>abnormal | Y | | $\forall$ | : |
|---|---|---|---|---|
| CFB | x.xx | x.x. | XX.X H | ÷ |
| Baseline | xx.x | XX.X | x.xx | i |
| Result | XX.X L | ×.× | ×.× | : |
| Vital sign<br>parameter (unit) | SBP (mmHg) | DBP (mmHg) | Pulse (beats/min) | Ē |
| Date/Time of<br>assessment/Study<br>day | DDMMMYYYY/HH:MM/xx SBP (mmHg) | | | DDMMMYYYY/HH:MM/xx |
| Day/Timepoint | XXXXX | | | XXXXX |
| Patient ID | XXXXXXXXXX | | | |

CFB: Change from baseline. Study day: Day relative to day of the single dose of study medication. Baseline: Defined as the assessment performed pre-dose. L and H represents marked decrease or increase from baseline.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell), within group by patient ID, and then timepoint.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-WD-201 ILF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.4 Derived Safety Measurements (Safety Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Derived Safety Measurements Listing 16.2.9.4

(Safety Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/Placebo>

| Peak<br>Pulse Rate (bpm) (over 4 hours) | | |
|-----------------------------------------|--------------|---|
| Peak<br>Pulse Rate (b) | XXXX.X | : |
| Peak<br>Heart Rate (bpm) (over 4 hours) | X.XXX | : |
| Date/<br>Study day | DDMMMYYYY/xx | : |
| Patient ID | XXXXX | : |

Peak = Maximum post-dose value among the values collected up to timepoint of interest hours. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell), within group by patient ID, and then  ${\sf date/time}$ .


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.5 Brief Physical Examination (Safety Analysis Set in Part A) Verona Pharma

Page X of Y Part A

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.5

Brief Physical Examination

(Safety Analysis Set in Part A)

Treatment group: <RPL554 150µg/RPL554 500µg/RPL554 1500µg/RPL554 3000µg/RPL554 6000µg/Placebo>

| Patient ID | Date/Time of examination/Study day | Body system | Result<br>If Abnormal, clinical significant, Specify |
|---|---|---|---|
| 8 | DMMMYYYY/HH: | XXXXXXXXXXXX | XXXXXXXXXXXXXX |

Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell), within group by patient ID and then alphabetically by body system. Only include patients with at least one markedly abnormal clinically significant finding.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.6 Full Physical Examination (Safety Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.6

Full Physical Examination

(Safety Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 3000µg/RPL554 6000µg/RPL6000

| | 1 | |
|---------|-----------|----------|
| | Specify | |
| | nificant, | |
| | ical sign | |
| | al, clin | XXXX |
| Result | Abnorma. | XXXXXXX |
| Re | ΙĮ | XX |
| | | XX |
| | system | XXXXXXX |
| | Body | XXXX |
| | ıdy day | 1/xx |
| me of | tion/Str | YY/HH:M |
| Date/Ti | examina | DDMMMYY |
| | | × |
| | atient ID | XXXXXXXX |
| | Pat | × |

CFB: Change from baseline. Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell), within group by patient ID and then alphabetically by body system. Only include patients with at least one markedly abnormal clinically significant finding.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.7 Chest X-ray (All Randomized Analysis Set in Part A) Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part A

Listing 16.2.9.7

Chest X-ray

(All Randomized Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| Result of X-ray/<br>Specification (eCRF) | Abnormal clinically significant/please specify | Consistent with COPD |
|---|---|---|
| Date of X-ray/<br>Study day | DDMMWYYY/xx | DDMMYYYY / xx |
| Chest X-ray<br>performed | New | Historical |
| Patient ID | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXX |

eCRF: Electronic case report form. Study day: Day relative to day of the single dose of study medication. Chest X-ray is assessed at Screening. Patient performs either a new X-ray ("New") or if an X-ray was performed in the last 12 months, this is acceptable ("Historical").

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order by treatment group (as per shell) and within group by patient ID. Specification (eCRF) refers to result "Abnormal clinically significant" where free text could be required to be concatenated.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.8 Inhalation Training (All Randomized Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

> Inhalation Training Listing 16.2.9.8

(All Randomized Analysis Set in Part A)

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/Placebo>

| Date of inhalation training/ | Study day | DDMMMYYY / xx |
|------------------------------|------------|---------------|
| Inhalation training | given? | XXXXXXX |
| | Timepoint | XXXX/XXXX |
| | Patient ID | XXXXXXX |

Study day: Day relative to day of the single dose of study medication.

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.

Document: 2:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp
#### Clinical Study Report RPL554-MD-201

### Version 1.0; 17 May 2021

# DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.9 Pregnancy Serum and Urine Test at Screening (All Randomized Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

> Pregnancy Serum and Urine Test at Screening (All Randomized Analysis Set in Part A) Listing 16.2.9.9

Treatment group: <RPL554 100µg/RPL554 300µg/RPL554 1000µg/RPL554 300µg/RPL554 6000µg/PPL3cebo>

| Urine<br>pregnancy<br>test result | XXXXXXX |
|---|---|
| Urine pregnancy test<br>performed/Date of<br>test/Study day | XX/DDMMYYYY/xx |
| Serum pregnancy test<br>result | XXXXXXX |
| Serum pregnancy test<br>performed/Date of test/Study<br>day | XX/DDMMMYYYY/xx |
| Patient ID | XXXXXXX |

Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes Order group (as per shell) and within group by patient ID. Consider only female patients.

Consider only female patients.

Multiple pregnancy risk factors and multiple relevant family history will be presented as one result per row, as these are not presented separately in Pregnancy report eCRF.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201


DocuSign Envelope ID: 5C5B89F7-2E1F-48F2-BC37-30CD3E98C5D3

Listing 16.2.9.10 Pregnancy Report at Screening (All Randomized Analysis Set in Part A) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part A

Listing 16.2.9.10

(All Randomized Analysis Set in Part A) Pregnancy Report at Screening

Treatment group: <RPL554 100ug/RPL554 300ug/RPL554 300ug/RPL554 6000ug/PPL3600>

| Patient ID | Pregnancy report item | Results |
|--------------|-----------------------------------------|--------------|
| XXXXXXXXXXXX | Date of last menstrual period/Study day | DDMMYYYY/xx |
| | Date of expected delivery/Study day | DDMMWYYYY/xx |
| | Overall number of previous pregnancies | XX |
| | Number of normal deliveries | XX |
| | Number of spontaneous miscarriages | XX |
| | Number of other previous pregnancies | XX |
| | Relevant pregnancy risk factors | XXXXXXXXX |
| | Relevant family history | XXXXXXXXX |

Study day: Day relative to day of the single dose of study medication.

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Programming Notes
Order by treatment group (as per shell) and within group by patient ID.
Consider only female patients.
Multiple pregnancy risk factors and multiple relevant family history will be presented as one result per row, as these are not presented separately in Pregnancy report eCRF.

Document: Z:\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part A

Author: Nicholas Roubinis/Jennifer Allsopp


CONFIDENTIAL Verona Pharma plc



# TABLES, LISTINGS AND FIGURES SHELLS - PART B

RPL554-MD-201

Single and Repeat Doses of RPL554 Administered by Pressurised Metered Dose Inhaler in Patients A Phase II, Randomized Study to Assess the Pharmacokinetics, Safety and Pharmacodynamics of with COPD

AUTHOR: JENNIFER ALLSOPP

VERSION NUMBER AND DATE: V2.0, 22JAN2021

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

# TABLES, LISTINGS AND FIGURES SHELLS – PART B SIGNATURE PAGE

Tables, Listings and Figures Shells V2.0 - Part B (Dated 22JAN2021) for Protocol RPL554-MD-201.

| | Name | Signature | Date |
|-----------|------------------------|-----------|------|
| Author: | Jennifer Allsopp | | |
| Position: | Senior Biostatistician | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Tables, Listings and Figures Shells – Part B, authorizing that the content is acceptable for the reporting of this study.

| fame our reference or remaining | | | |
|---|---|---|---|
| | Name | Signature | Date |
| Approved by: | Mark Shaw | | |
| Position: | Associate Director | | |
| Company: | IQVIA | | |
| Approved by: | Tara Rheault | | |
| Position: | VP, R&D Operations and Project Management | anagement | |
| Company: | Verona Pharma | | |
| Approved by: | Thomas Bengtsson | | |
| Position: | Statistical Consultant to Verona | | |
| Company: | StatMind | | |

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

# Modification History

| Unique Identifier for this Version Date of the Document Version Author | Date of the Document Version | Author | Significant Changes from Previous Authorized |
|---|---|---|---|
| | | | Version |
| 1.0 | 13JAN2021 | Jennifer Allsopp | Not Applicable – First Draft Version |
| 2.0 | 22JAN2021 | Jennifer Allsopp | Update treatment sequences from blinded sequences |
| | | | to unblinded sequences in output footnotes. |

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

# Table of Contents

| Tables |
|---|
| 14.1 Demographic Data |
| Table 14.1.7 Patient Disposition by Treatment Sequence (Part A Completers) |
| Table 14.1.8 Patient Disposition by Treatment Group (All Randomized Analysis Set in Part B) |
| Table 14.1.9 Analysis Set by Treatment Sequence (All Randomized Analysis Sets in Part B) |
| Table 14.1.10 Analysis Set by Treatment Group (All Randomized Analysis Sets in Part B) |
| Table 14.1.11 Major/Critical Protocol Deviations (All Randomized Analysis Sets in Part B) |
| Table 14.1.12 Demographic Characteristics (All Randomized Analysis Sets in Part B) |
| Table 14.1.13 Screening Disease Characteristics (All Randomized Analysis Sets in Part B) |
| Table 14.1.14 COPD and Smoking History (All Randomized Analysis Sets in Part B) |
| Table 14.1.15 Drug Exposure and Accountability (Safety Analysis Sets in Part B) |
| 14.2 Efficacy |
| Primary Efficacy |
| Table 14.2.5 FEV, by Treatment and Timepoint (Full Analyis Set in Part B) |
| Table 14.2.6 Change from Baseline FEV1 to Peak FEV1 (over 4 hours) on Day 7 (Full Analysis Set in Part B) |
| Table 14.2.6a Change from Baseline FEV; to Peak FEV; (over 4 hours) on Day 7 - Sensitivity Analysis (Completers Analysis Set in Part B) |
| Secondary Efficacy |
| Table 14.2.7 Average FEV1 by Day and Treatment Group (Full Analysis Set in Part B) |
| Table 14.2.8 Change from Baseline FEV; to Average FEV; (over 4 hours) on Day 7 (Full Analysis Set in Part B) |
| Table 14.2.9 Change from Baseline FEV1 to Average FEV1 (over 12 hours) on Day 7 (Full Analysis Set in Part B) |
| Table 14.2.9a Change from Baseline FEV; to Average FEV; (over 12 hours) on Day 7 - Sensitivity Analysis (Full Analysis Set in Part B) |
| Table 14.2.10 Change from Baseline FEV; to Morning Trough FEV; on Day 7 (Full Analysis Set in Part B) |
| Table 14.2.11 Change from Baseline FEV; to Peak FEV; (over 4 hours) on Day 1 (Full Analysis Set in Part B) |
| Table 14.2.12 Change from Baseline FEV; to Average FEV; (over 4 hours) on Day 1 (Full Analysis Set in Part B) |
| Table 14.2.13 Change from Baseline FEV; to Average FEV; (over 12 hours) on Day 1 (Full Analysis Set in Part B) |
| Table 14.2.14 Time to Onset of Action (>10% Increase in FEV;) on Day 1 (Full Analysis Set in Part B) |
| Table 14.2.15 Rescue Medication Use (Full Analysis Set in Part B) |
| Exploratory Efficacy |
| Table 14.2.16 Dyspnea Scale by Day and Timepoint (Full Analysis Set in Part B) |
| Table 14.2.17 Comparison of Change from Baseline Dyspnea Score by Day and Timepoint (Full Analysis Set in Part B) 41 |
| 14.3 Safety |
| Adverse Event |
| Document: \\ieedc-vnasc01\\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 |
| Version: 2.0 Date: 22JAN2021 |

| Table 14.3.27 Treatment-emergent Adverse Events Summary (Safety Analysis Set in Part B) |
|---|
| Table 14.3.28 Treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part B) 46 |
| Table 14.3.29 Treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part B) |
| Table 14.3.30 Treatment-emergent Adverse Events by System Organ Class and Preferred Term and Maximum Severity (Safety Analysis Set in Part B) 49 |
| Table 14.3.31 Treatment-emergent Adverse Events Leading to Discontinuation of Study by System Organ Class and Preferred Term (Safety Analysis Set in Part B) |
| Table 14.3.32 Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part B) 51 |
| Table 14.3.33 Serious Treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part B) |
| Table 14.3.34 Serious Treatment-emergent Adverse Events by System Organ Class, and Preferred Term and Maximum Severity (Safety Analysis Set in Part B) |
| Table 14.3.35 Serious Treatment-emergent Adverse Events Leading to Discontinaution of Study by System Organ Class and Preferred Term (Safety Analysis Set in Part B) |
| Table 14.3.36 Treatment-emergent Adverse Events with Outcome of Death by System Organ Class and Preferred Term (Safety Analysis Set in Part B) |
| Laboratory 53 |
| Table 14.3.37 Hematology Laboratory Data by Day (Safety Analysis Set in Part B) |
| Table 14.3.38 Biochemistry Laboratory Data by Day (Safety Analysis Set in Part B)55 |
| Table 14.3.39 Urinalysis Laboratory Data by Day (Safety Analysis Set in Part B) |
| Table 14.3.40 Hematology Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B) 56 |
| Table 14.3.41 Biochemistry Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B) 58 |
| Table 14.3.42 Urinalysis Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B) 58 |
| Table 14.3.43 Biochemistry Laboratory Data - Markedly Abnormal Values (Safety Analysis Set in Part B) 59 |
| BCG |
| Table 14.3.44 12-Lead Electrocardiogram Data by Day and Timepoint (Safety Analysis Set in Part B) |
| Table 14.3.45 12-Lead Electrocardiogram - Shifts from Baseline by Day and Timepoint (Safety Analysis Set in Part B) |
| Vital Signs |
| Table 14.3.46 Vital Sign Data - Change from Baseline to Post-dose by Day and Timepoint (Safety Analysis Set in Part B) 63 |
| Table 14.3.47 Vital Sign Data - Number and Percentage of Markedly Abnormal Values (Safety Analysis Set in Part B) |
| Table 14.3.48 Change from Baseline Pulse Rate to Peak Pulse Rate (over 4 hours) (Safety Analysis Set in Part B) 67 |
| Physical Examination |
| Table 14.3.49 Physical Examination Data by Treatment Period and Timepoint (Safety Analysis Set in Part B) |
| Table 14.3.50 Physical Examinations - Shifts from Baseline by Treatment Period and Timepoint (Safety Analysis Set in Part B) 70 |
| igures72 |
| Figure 14.2.6 Geometric Mean of ratios of Peak FEV; (over 4 hours) to pre-dose FEV; by Treatment (Full Analysis Set in Part B) 72 |
| ocument: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 |

Author: Jennifer Allsopp

| Figure 14.2.7 Mean Change from pre-dose FEV; to Peak FEV; (over 4 hours) by Treatment (Full Analysis Set in Part B) | . 73 |
|---|---|
| Figure 14.2.8 Mean Change from Pre-dose FEV, during spirometry over Time by Treatment and Day (Full Analysis Set in Part B) | . 74 |
| Figure 14.2.9 Kaplan-Meier plot of Time to Onset of Action (>10% Increase in FEV;) on Day 1 (Full Analysis Set in Part B) | . 75 |
| Figure 14.3.5 Mean Change from Pre-dose Pulse Rate to Peak Pulse Rate (over 4 hours) by Treatment (Safety Analysis Set in Part B) 7 | 97 ( |
| Figure 14.3.6 Mean Change from Pre-dose in Pulse Rate over Time by Treatment and Day (Safety Analysis Set in Part B) | . 76 |
| Listings | . 77 |
| Listing 16.2.1.2 Completed/Discontinued Patients (All Randomized Analysis Set in Part B) | . 77 |
| Listing 16.2.2.2 Protocol Deviations (All Randomized Analysis Set in Part B) | . 78 |
| Listing 16.2.3.2 Patient Included in Analysis Sets (All Randomized Analysis Set in Part B) | . 79 |
| Listing 16.2.4.7 Demographic Characteristics (All Randomized Analysis Set in Part B) | . 80 |
| Listing 16.2.4.8 Screening Disease Characteristics (All Randomized Analysis Set in Part B) | . 81 |
| Listing 16.2.4.9 COPD and Smoking History (All Randomized Analysis Set in Part B) | . 82 |
| Listing 16.2.4.10 Medical History (All Randomized Analysis Set in Part B) | . 83 |
| Listing 16.2.4.11 Surgical Procedure History (All Randomized Analysis Set in Part B) | . 84 |
| Listing 16.2.4.12 Prior and Concomitant Medications (All Randomized Analysis Set in Part B) | . 85 |
| Listing 16.2.4.13 Prior COPD Medications (All Randomized Analysis Set in Part B) | . 86 |
| Listing 16.2.5.2 Drug Exposure and Accountability (All Randomized Analysis Set in Part B) | . 87 |
| Listing 16.2.6.5 Spirometry: FEV1 Results (Full Analysis Set in Part B) | œ<br>œ |
| Listing 16.2.6.6 Spirometry: FEV1 Derived Measurements (Full Analysis Set in Part B) | 68 |
| Listing 16.2.6.7 Spirometry: FEV1 Time to First Occurrence of Onset of Action (Full Analysis Set in Part B) | 06. |
| Listing 16.2.6.8 Dyspnea Scale Score (Full Analysis Set in Part B) | . 91 |
| Listing 16.2.6.9 Rescue Medications (All Randomized Analysis Set in Part B) | . 92 |
| Listing 16.2.6.10 Rescue Medications Canister Dispensed, Weight and Collection Information (All Randomized Analysis Set in Part B) | B) |
| Listing 16.2.7.6 List of All Adverse Events (Safety Analysis Set in Part B) | . 94 |
| Listing 16.2.7.7 Treatment-emergent Adverse Events Leading to Study Discontinutation (Safety Analysis Set in Part B) | . 95 |
| Listing 16.2.7.8 Treatment-emergent Adverse Events Leading to Death (Safety Analysis Set in Part B) | . 95 |
| Listing 16.2.7.9 Serious Treatment-emergent Adverse Events (Safety Analysis Set in Part B) | . 95 |
| Listing 16.2.7.10 Serious Treatment-emergent Adverse Events - Details (Safety Analysis Set in Part B) | 96. |
| Listing 16.2.8.5 Hematology (Safety Analysis Set in Part B) | 80 |
| Listing 16.2.8.6 Biochemistry (Safety Analysis Set in Part B) | 80 |
| Listing 16.2.8.7 Urinalysis (Safety Analysis Set in Part B) | 66. |
| Listing 16.2.9.11 Electrocardiogram Local Reading Overall Evaluation (Safety Analysis Set in Part B) | 100 |
| Listing 16.2.9.12 12-lead ECG (Safety Analysis Set in Part B) | 101 |
| Listing 16.2.9.13 Vital Signs (Safety Analysis Set in Part B) | 102 |
| Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 | 0. |
| Version:<br>Date: 22JAN2 | 2.0 |

| Listing 16.2.9.14 Vital Signs - Patients with at Least One Markedly Abnormal Finding (Safety Analysis Set in Part B) | Listing 16.2.9.15 Derived Safety Measurements (Safety Analysis Set in Part B) | Listing 16.2.9.16 Brief Physical Examination (Safety Analysis Set in Part B) | Listing 16.2.9.17 Full Physical Examination (Safety Analysis Set in Part B) | 10. | Listing 16.2.9.19 Pregnancy Urine Test Results (All Randomized Analysis Set in Part B) | Listing 16.2.9.20 Pregnancy Report Results (All Randomized Analysis Set in Part B) |
|---|---|---|---|---|---|---|
| Ξ. | Ξ. | Ξ. | Ξ. | Ξ. | Ξ. | Ξ. |
| - : | - : | : | - : | : | : | : |
| - 1 | - : | - : | - 1 | : | - : | : |
| - : | - : | - : | - : | : | - : | - : |
| - : | - : | - : | - : | : | - : | - : |
| - 1 | : | : | - 1 | - : | : | : |
| m | | : | - 1 | : | : | : |
| μ. | - 1 | - : | - 1 | - 1 | - : | - : |
| ar | | | - 1 | | | : |
| щ | : | : | - 1 | : | : | : |
| 귀 | : | | - 1 | : | | : |
| 4 | : | : | - : | : | : | : |
| Ω | - : | - : | - 1 | - : | - : | - : |
| ٠H<br>دی | | | | | | |
| Z S | : | : | - 1 | : | : | : |
| al | : | : | - 1 | : | : | : |
| Ar | : | : | - 1 | : | : | : |
| > | : | : | - 1 | : | : | : |
| fe t | - : | | - : | ÷ | | |
| ςς<br>α | - 1 | - : | - 1 | - 1 | : | - : |
| | | | - 1 | | B | : |
| n.g | : | : | - 1 | : | ± | • |
| ğ | : | : | - 1 | : | Par | B |
| 11 | : | | - : | : | - | r, |
| 7 | B | · | - : | B | ÷ | Pai |
| ma | ₽ | Щ | B | ц | e<br>T | g |
| Or | ar | rt | щ | ar | Ω | H |
| h | П | Б | ar | Щ | -1 | et |
| A | H | Е. | щ | Ή | Lys | m (I) |
| d. | (I) | ٠. | ÷ | 0 | ng. | 91.5 |
| ķ | Ω | Se | et<br>Ct | Ŋ | A | 17 |
| ar | -H | (C) | Ω | -H | eq | пa |
| Σ | ΥS | Si | -13 | ΥS | ijΣ | ×. |
| )ne | la] | 117 | 7.5 | la] | lon | eq |
| 1) | A | Į, | la] | A | ng<br>Out | Βį |
| α<br>Ω | 7 | > | A | ď | ĸ | dor |
| Le | Œ<br>H | et | ťΣ | j. | H | ano |
| ц | Ω<br>Q | а£ | E<br>E | E O | A) | ĸ |
| σ_ | | 8 | Sa | ng | Ø | 큠 |
| Ę. | ıt s | п | _ | E, | ıl t | (4) |
| × | ner | Ę. | ior | d. | e Si | S |
| t s | r ei | ď | at | Ø | ĸ | 급 |
| en | Su | jd. | in | מ | st | 0 |
| ţį | lea | × | am | ij | Ð | <u>m</u> |
| Ра | 2 | 国 | Ä | in | 9 | ort |
| 1 | et. | ďa | 근 | Pra | ŗ. | de |
| S | afe | Sic | Ö | g | Ď | Ä |
| эg | cΩ | μV | ΣS | .н<br>О | ς | Ç |
| Ω. | eq | D4 | Ph | at | nan | lan |
| al | Ş. | ef | d | lal | gu | gu |
| Vit | Der | 3ri | En | II. | Pre | Pre |
| 4 | 5 | 9 | 7 | 00 | 0 | 0 |
| ÷. | ÷. | ď. | $\vdash$ | ď. | Η. | 2 |
| 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| . 2 | 5.2 | . 2 | . 2 | . 2 | . 2 | 2.2 |
| 16 | 16 | 16 | 16 | 16 | 16 | 16 |
| ng | ng | пg | ng | ng | пg | ng |
| ţį | ţį | ţij | ţį | Listing 16.2.9.18 Inhalation Training (All Randomized Analysis Set in Part B) | ţij | ţį |
| -H | ٠ <del>٠</del> | -H | -H | -H | -H | ٠.<br>ا |
| Н | Н | н | Н | Н | н | H |

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B Author: Jennifer Allsopp

#### Tables

14.1 Demographic Data Table 14.1.7 Patient Disposition by Treatment Sequence (Part A Completers) Verona Pharma Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Part B

Page X of Y

 $\label{eq:Treatment Sequence}$  Patient Disposition by Treatment Sequence

(Part A Completers)

| | 02 | Seq 1 | w | Seg 2 | S | Seq 3 | Se | Seg 4 | Õ | Overall |
|---|---|---|---|---|---|---|---|---|---|---|
| Description, n (%) | | N=XX | 4 | N=XX | Ż | N=XX | Ż | N=XX | _ | N=XX |
| Number of patients conmpleted Part A | | | | | | | | | | × |
| Number of patients to withdrew between Part A and Part B | | | | | | | | | | × |
| Number of patients randomized (n) | | ×× | | ×× | | ×× | | ×× | | ×× |
| Number of patients treated in: | | | | | | | | | | |
| Treatment Period 1 | ×× | xx (xx.x) | × | (xx.x) xx | ×× | xx (xx.x) | × | (x.xx) xx | × | (xx.x) xx |
| Treatment Period 2 | × | (xx.x) | × | xx (xx.x) | ×× | xx (xx.x) | × | xx (xx.x) | × | (xx.x) xx |
| Treatment Period 3 | ×× | xx (xx.x) | × | (xx.x) xx | ×× | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) |
| Treatment Period 4 | × | xx (xx.x) | × | (x.xx) xx | × | xx (xx.x) | × | (xx.x) xx | × | xx (xx.x) |
| Number of patients who completed the study | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xxxx) xx | × | (xx.x) |
| Number of patients who discontinued the study in: | | | | | | | | | | |
| Treatment Period 1 | × | xx (xx.x) | × | xx (xx.x) | ×× | xx (xx.x) | × | (xx.xx) xx | × | xx (xx.x) |
| Treatment Period 2 | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xx.x) xx |
| Treatment Period 3 | × | (xx.x) | × | xx (xx.x) | ×× | xx (xx.x) | × | xx (xx.x) | × | (xx.x) xx |
| Treatment Period 4 | × | (xx.x) | × | (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) |
| Overall | × | xx (xx.x) | × | xx (xx.x) | ×× | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) |

Primary reason for early study discontinuation

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA84488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Protocol: RPL554-MD-201 Verona Pharma

Part B

Page X of Y

RPL554 pressurised Metered Dose Inhaler

Patient Disposition by Treatment Sequence (Part A Completers)

| | Seg 1 | 1 | Seq 2 | Seq 3 | Seq 4 | Overall |
|---|---|---|---|---|---|---|
| Description, n (%) | N=XX | × | N=XX | N=XX | N=XX | N=XX |
| Adverse event | (x.xx) xx | | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) |
| Death | (x.xx) xx | | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xxx) xx |
| Lost to follow-up | (x.xx) xx | | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) |
| Pregnancy | xx) xx | x (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol violation | (x.xx) xx | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | xx) xx | x (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal by patient | (x.xx) xx | | xx (xx.x) | (xxx) xx | (xxx) xx | (xxxx) |

xx (xx.x)

(xx.x) xx

xx (xx.x)

xx (xx.x)

xx (xx.x)

Other

n = Number of patients. N = Number of patients randomized in Part B. % = Percentage of patients calculated relative to the total number of patients in the analysis Set.

Patients who completed the study excludes patients who withdrew from the study and patients who did not complete all treatment periods i.e. a patient who receives a first and last dose intake plus 1 day for all 4 treatment periods per schedule of events.

Percentages for early discontinuation reasons is calculated based on the number of patients who had early discontinuation data.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 1000 mcg/RPL554 3000 mcg. Seq 2 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg. Seq 9 = Placebo/RPL554 3000 mcg/RPL554 300

Source: Listing 16.2.1.2

Output ID: DS001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.1.8 Patient Disposition by Treatment Group (All Randomized Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Part B

Page X of Y

RPL554 pressurised Metered Dose Inhaler

Table 14.1.8

(All Randomized Analysis Set in Part B) Patient Disposition by Treatment Group

| | RPLS | RPL554 300µg | Z 7 | RPL554<br>1000µg | RP<br>30 | RPL554<br>3000µg | Pla | Placebo | Ove | Overall |
|---|---|---|---|---|---|---|---|---|---|---|
| Description, n (%) | | N=XX | 1 | N=XX | N | N=XX | N | N=XX | N<br>= | N=XX |
| Number of patients treated | × | (x.xx) xx | × | (x.xx) xx | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) |
| Number of patients who completed the study | × | xx (xx.x) | × | (xx) xx | × | xx (xx.x) | × | (xx.x) | × | (xx.x) |
| Number of patients who discontinued the study | × | (x.xx) xx | × | (x.xx) xx | × | (x.x.x) | × | (x.xx) xx | × | (x.xx) xx |
| Primary reason for early study discontinuation | | | | | | | | | | |
| Adverse event | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xx.x) | ×× | xx (xx.x) |
| Death | × | (xx.x) | × | (xx.x) xx | × | xx (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Lost to follow-up | ×× | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Pregnancy | × | xx (xx.x) | × | (xx.x) | × | xx (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Protocol violation | × | xx (xx.x) | × | xx (xx.x) | × | xx (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Physician decision | × | xx (xx.x) | × | (xx.x) | × | xx (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Study terminated by sponsor | × | xx (xx.x) | × | (xx.x) xx | × | (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Withdrawal by patient | × | xx (xx.x) | × | (xx.x) | × | xx (xx.x) | × | (xx.x) | ×× | (xx.x) |
| Other | × | (x.xx) xx | × | (x.xx) xx | × | xx (xx.x) | × | (x.xx) xx | ×× | (x.xx) xx |

N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis Set.

Patients who completed the study excludes patients who withdrew from the study and patients who did not complete all treatment periods i.e. a patient who receives a first and last dose intake plus 1 day for all 4 treatment periods per schedule of events. Percentages for early discontinuation reasons is calculated based on the number of patients who had early discontinuation data.

Source: Listing 16.2.1.2

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp


Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

#### Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Part B

Page X of Y

Patient Disposition by Treatment Group

(All Randomized Analysis Set in Part B)

| | Overall | N=XX |
|--------|--------------|----------------|
| | Placebo | X=N |
| RPL554 | 3000µg | X=XX |
| RPL554 | 1000µg | XX=N |
| | RPL554 300µg | XX=N |
| | | (%) u |
| | | Description, 1 |

Output ID: DS002

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Table 14.1.9 Analysis Set by Treatment Sequence (All Randomized Analysis Sets in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

Analysis Sets by Treatment Sequence Table 14.1.9

(All Randomized Analysis Set in Part B)

| | Seq 1 | Seq 2 | Seq 3 | Seq 4 | Overall |
|---|---|---|---|---|---|
| Analysis set, n (%) | N=XX | N=XX | N=XX | N=XX | N=XX |
| Randomized Analysis Set | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx | xx (xx.x) |
| Safety Analysis Set | (x.xx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx |
| Full Analysis Set | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) |
| Completers Analysis Set | (xx.x) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pharmacokinetics Analysis Set | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n = Number of patients. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients. Set in Part B.

All Randomized Analysis Set in Part B.

All Randomized Analysis Set set: Randomized patients.

Safety Analysis Set: Randomized patients who received at least one dose of study medication.

Full Analysis Set: Patients included in the Safety Analysis Set with sufficient data to compute the pharmacodynamic parameters on at least two treatment periods.

Full Analysis Set: Patients included in the Safety Analysis Set who complete all treatment periods i.e. a patient who receives a first and last dose intake plus I day for all 4 treatment periods per schedule of events.

Pharmacokinetics Analysis Set: Patients included in the All Randomized Analysis Set who have a blood sampling performed after at least one dose of study medication and pharmacokinetic parameter data.

Seq 1 = RPL554 300 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 2 = RPL554 3000 mcg/RPL554 300 mcg. RPL554 300 mcg.

Source: Listing 16.2.3.2

Output ID: DS003

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.1.10 Analysis Set by Treatment Group (All Randomized Analysis Sets in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.1.10

(All Randomized Analysis Set in Part B)

Analysis Sets by Treatment Group

| | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo | Overall |
|---|---|---|---|---|---|
| Analysis set, n (%) | N=XX | N=XX | N=XX | N=XX | N=XX |
| Randomized Analysis Set | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Safety Analysis Set | xx (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Full Analysis Set | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.x) xx | xx (xx.x) |
| Completers Analysis Set | xx (xx.x) | (x.xx) xx | xx (xx.x) | (xxx) xx | xx (xx.x) |
| Pharmacokinetics Analysis Set | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n = Number of patients. N = Number of patients randomized. % = Percentage of patients calculated relative to the total number of patients in All Randomized Analysis Set in Part B.
All Randomized Analysis Set: Randomized patients.
Safety Analysis Set: Randomized patients.
In Part B.
In It analysis Set: Randomized patients who received at least one dose of study medication.
Full Analysis Set: Randomized patients who received at least two treatment periods completers analysis Set: Patients included in the Safety Analysis Set who complete all treatment periods a first and last dose inteake plus I day for all 4 treatment periods per schedule of events.
Pharmacokinetics Analysis Set: Patients included in the All Randomized Analysis Set who have a blood sampling performed after at least one dose of study medication and pharmacokinetic parameter data.

Source: Listing 16.2.3.2

Output ID: DS004

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.1.11 Major/Critical Protocol Deviations (All Randomized Analysis Sets in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Major/Critical Protocol Deviations

(All Randomized Analysis Set in Part B)

| Severity/ | RPL554 300µg | RPL554 1000µg | RPL554 300µg RPL554 1000µg RPL554 3000µg | Placebo | Overall |
|---|---|---|---|---|---|
| Deviation type | N=XX | N=XX | N=XX | N=XX | N=XX |
| Patients with at least one critical/major protocol deviation, n (%) | (xx.x) | (xx.x) | (xx.x) | (x.xx) xx | xx (xx.x) |
| Critical | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type 1 | (x.xx) | xx (xx.x) | (xx.x) | (xx.x) | xx (xx.x) |
| Type 2 | (xxx) xx | (x.xx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Major | | | | | |

CTMS: Clinical trial management system. n = Number of patients. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis set. Protocol deviations were obtained from CTMS.

Source: Listing 16.2.2.2

Programming Notes

Deviation types are sorted in descending order of frequency of the Overall column. A patient may have multiple critical/major protocol deviations within and is counted once at each level of summarization.

Output ID: DV001

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Table 14.1.12 Demographic Characteristics (All Randomized Analysis Sets in Part B) Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.1.12

Demographic Characteristics
(All Randomized Analysis Set in Part B)

| N=XX | N=XX | N=XX | N=XX |
|---|---|---|---|
| ×× | ×× | ×× | × |
| x. xx | xx.xx | xx.x | x.xx |
| XX.XX | xx.xx | xx.xx | xx.xx |
| xx.x | xx.x | xx.x | xx.x |
| xx, xx | xx, xx | xx, xx | xx, xx |
| xx (xx.x) | (xx.x) xx | (xx.x) | (x.xx) xx |
| (xxxx) xx | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| xx (xx.x) | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| xx (xx.x) | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| xx (xx.x) | (xx.x) xx | (xx.x) xx | xx (xx.x) |
| xx (xx.x) | (xxxx) xx | xx (xx.x) | xx (xx.x) |
| xx (xx.x) | (xx.xx) xx | (xx.x) | xx (xx.x) |
| xx (xx.x) | (xx.x) xx | (xx.x) xx | xx (xx.x) |
| xx (xx.x) | (x.xx) | (xx.x) | xx (xx.x) |
| | XX.XX | | XX. XX XX. XX XX, XX XX, XX XX (XX. X) XX (X |


Verona Pharma plc

Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler Verona Pharma

Part B Page X of Y

(All Randomized Analysis Set in Part B) Demographic Characteristics Table 14.1.12

| Characteristic / | RND | SAF | FAS | CAS | PK |
|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| * 0 d + 0 | | | | | |
| Cried | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | | | |
| Hispanic or Latino | xx (xx.x) | (xx.x) | (xx.x) | (x.xx) xx | xx (xx.x) |
| African American/African Heritage | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) |
| Asian-Central/South Asian Heritage | xx (xx.x) | (xx.x) | (xxx) xx | (xx.x) xx | (x.xx) xx |
| Asian-East Asian Heritage | xx (xx.x) | xx (xx.x) | (xxx) xx | (xxxx) xx | xx (xx.x) |
| Asian-Southeast Asian Heritage | xx (xx.x) | xx (xx.x) | (xxx) xx | (xxxx) xx | xx (xx.x) |
| White/Caucasian/European Heritage | xx (xx.x) | xx (xx.x) | (xx.x) | (xx.x) xx | xx (xx.x) |
| Not reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Weight (kg) | | | | | |
| u | ×× | ×× | ×× | ×× | ×× |
| Mean | × × × | ×.×. | ××× | × · × × | ×.×× |
| SD | XX.XX | xx.xx | XX.XX | XX.XX | xx.xx |
| Median | ×. ×. | ×.×× | ×.×× | ×.×× | ×××× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Height (cm) | | | | | |
| ់ ជ | × | × | × | × | × |
| Mean | ×. ×× | ×.×. | ×.×× | ××× | x.xx |
| SD | ××××× | xx.xx | ××·×× | xx.xx | xx.xx |
| Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 | \RPL554\EZAA8488\I | 3iostatistics\Docume | ntation\SAP\Verona ] | RPL554-MD-201 TLF S | hells v2.0 |
| anthore Januifer alleonn | | | | , +<br>e | Version: 2.0 |
| pacific ocilitate prescipi | | | | a d | C. ZZOMNZOZI |

Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Demographic Characteristics Table 14.1.12

(All Randomized Analysis Set in Part B)

| Characteristic / | RND | SAF | FAS | CAS | PK |
|------------------|--------|---------|--------|--------|--------|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| Median | x.xx | xx | xx.x | x. xx | xx.x |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| $BMI (kg/m^2)$ | | | | | |
| n | ×× | ×× | ×× | ×× | ×× |
| Mean | x.xx | xx.x | xx.xx | xx.x | xx.x |
| SD | XX.XX | XX.XX | xx.xx | XX.XX | xx.xx |
| Median | x.xx | x · x × | x. xx | x. xx | x.xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

BMI: Body Mass Index. SD: Standard deviation.

n = Number of patients. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis set.

v \* 8 = Percentage for childbearing potential calculated relative to the total number of female patients in the analysis set.

All Randomised Analysis Set (SAF): Randomized patients in Part B.

Safety Analysis Set (SAF): Randomized patients in Part B.

Full Analysis Set (SAF): Patients included in the Safety Analysis Set with sufficient data to compute the pharmacodynamic parameters on at least two treatment periods.

Completers Analysis Set (CAS): Patients included in the Safety Analysis Set who complete all treatment periods i.e. a patient who receives a first and last dose intake plus I day for all 4 treatment periods per schedule of events.

Pharmacokinetics Analysis Set (RAF): Patients included in the All Randomized Analysis Set who have a blood sampling performed after at least one dose of study medication and pharmacokinetic parameter data.

Source: Listing 16.2.4.7

Programming Notes

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

(All Randomized Analysis Set in Part B) Demographic Characteristics Table 14.1.12

| PK | N=XX |
|------------------|------------|
| CAS | N=XX |
| SI | N=XX |
| FAS | |
| SAF | N=XX |
| RND | N=XX |
| Characteristic / | Statistics |

Print all statistics and categories even if they are empty, except for the row of missings which will only be shown if present and is not shown in the shell here. This will not be relevant for ethnicity as there is a category noted as not reported. Therefore, no reason why missing should occur.

Output ID: DM001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Author: Jennifer Allsopp

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

Page X of Y Part B Table 14.1.13 Screening Disease Characteristics (All Randomized Analysis Sets in Part B) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

(All Randomized Analysis Set in Part B) Screening Disease Characteristics Table 14.1.13

| Statistics | N=XX | N=XX | N=XX | N=V | |
|---|---|---|---|---|---|
| | | | | IV—VI | N=XX |
| Pre-bronchodilator FEV $_1$ (L) | | | | | |
| ч | × | × | × | × | × |
| Mean | xx.x | ××× | ×.×. | ×.× | ×. × |
| SD | XX.XX | XX.XX | xx.xx | xx.xx | xx.xx |
| Median | XX.X | ×.×× | ×.× | x.xx | ×.× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Post-bronchodilator FEV $_1$ (L) | | | | | |
| а | XX | ×× | ×× | ×× | × |
| Mean | *** | ×.× | xx.x | x.xx | x.x |
| SD | ×××× | ××××× | XX.XX | ××.×× | ×××× |
| Median | *** | ××× | xx.x | ×××× | ×. × |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| FEV1 reversibility (mL) | | | | | |
| п | ×× | ×× | XX | ×× | × |
| Mean | ××× | ××.× | ××.× | xx.x | × × × |
| SD | ××××× | XX.XX | xx.xx | xx.xx | ××.×× |
| Median | X.XX | x.xx | ×.× | x.xx | x.xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc

Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part B

(All Randomized Analysis Set in Part B) Screening Disease Characteristics Table 14.1.13

| Characteristic / | RND | K SS | RAR | CAS | PK |
|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| FEV <sub>1</sub> reversibility (%) | | | | | |
| r | ×× | ×× | ×× | ×× | XX |
| Mean | ×.× | ×.× | ×.× | ×.×× | ×.× |
| SD | ××.×× | XX.XX | xx.xx | xx.xx | xx.xx |
| Median | ×.× | × · × × | ×.× | ×.× | ×.× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Pre-bronchodilator FVC (L) | | | | | |
| п | ×× | ×× | ×× | ×× | ×× |
| Mean | xx.x | x.xx | x.x | x.xx | ×.×. |
| SD | ××.×× | xx · xx | xx.xx | xx.xx | xx.xx |
| Median | ×.× | x . x x | ×.× | x.xx | ×.×× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Post-bronchodilator FVC (L) | | | | | |
| n | × | ×× | ×× | ×× | ×× |
| Mean | ×.× | x.x. | ×.× | ××.× | ×.× |
| SD | ××.×× | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | ×.× | ×.×× | ×.× | ×.×× | ×.× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B Pre-bronchodilator FEV1/FVC

Version: 2.0 Date: 22JAN2021 Author: Jennifer Allsopp

Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part B

(All Randomized Analysis Set in Part B) Screening Disease Characteristics Table 14.1.13

| Characteristic / | RND | SAF | FAS | CAS | PK |
|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| п | XX | ×× | ×× | ×× | ×× |
| Mean | ×××× | x.xx | x.xx | x.xx | x.xx |
| SD | ××.×× | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | ×.× | ××× | x.xx | x.xx | ×××× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Post-bronchodilator FEV;/FVC | | | | | |
| n | XX | ×× | ×× | ×× | ×× |
| Mean | ××.× | ×××× | xx.x | ××.× | x.xx |
| SD | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx |
| Median | ×.×× | ××× | ×××× | x.xx | × · × × |
| Min, Max | xx, xx | xx 'xx | xx, xx | xx, xx | xx 'xx |
| Post-bronchodilator FEV1 (% of predicted normal) | | | | | |
| n | ×× | ×× | ×× | ×× | ×× |
| Mean | ×.×× | ××× | ×××× | x.xx | × · × × |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx |
| Median | ×××× | ×××× | x.xx | x.xx | ×××× |
| Min, Max | xx, xx | xx 'xx | xx 'xx | xx 'xx | xx 'xx |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Version: 2.0 Date: 22JAN2021 Author: Jennifer Allsopp

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Page X of Y Part B

Table 14.1.13

Screening Disease Characteristics

(All Randomized Analysis Set in Part B)

| Cigracocorpio | RND | SAF | FAS | CAS | 전자 |
|---|---|---|---|---|---|
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| Reversibility assessment performed with four puffs of albuterol, n $(\$)$ | | | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx | xx (xx.x) |
| No | xx (xx.x) | (x.x.) xx | xx (xx.x) | xx (xx.x) | (x.xx) xx |
| Met protocol requirements of reversibility test [a], n $(\$)$ | | | | | |
| Yes | xx (xx.x) | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx |
| No | xx (xx.x) | (xxxx) xx | xx (xx.x) | xx (xx.x) | (xxxx) xx |

Pre-, post-bronchodilator and reversibility values are the results of the screening reversibility test.

[a] Patients meet the protocol requirements of the reversibility test by demonstrating >=150 mL increase from pre-bronchodilator FEV.

FEV.

All Romomised Analysis Set in Part B (RND): Randomized patients in Part B.

Salety Analysis Set (SAF): Randomized patients who received at least one dose of study medication.

Full Analysis Set (FAS): Patients included in the Safety Analysis Set with sufficient data to compute the pharmacodynamic parameters on at least two treatment periods.

Completers Analysis Set (CAS): Patients included in the Safety Analysis Set who complete all treatment periods i.e. a patient who receives a first and last dose intake plus 1 day for all 4 treatment periods per schedule of events.

Pharmacokinetics Analysis Set (FK): Patients included in the All Randomized Analysis Set who have a blood sampling performed after at least one dose of study medication and pharmacokinetic parameter data.

Source: Listing 16.2.4.8

Output ID: DM005

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

Page X of Y Part B Table 14.1.14 COPD and Smoking History (All Randomized Analysis Sets in Part B) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

(All Randomized Analysis Set in Part B) COPD and Smoking History Table 14.1.14

| | ××=N | X=N | XX=N | >-IN |
|---|---|---|---|---|
| N=XX | **** | | | VV-N |
| × | × | ×× | ×× | × |
| x.xx | ×.× | x.xx | x.xx | ××× |
| ××.×× | ××.×× | xx.xx | xx.xx | ××.×× |
| x.x. | x.xx | ××.× | ×.×× | x.xx |
| xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| xx (xx.x) | (x.xx) xx | (xx.x) | (x.xx) xx | xx (xx.x) |
| xx (xx.x) | (x.xx) xx | (x.x.x) xx | (x.xx) xx | xx (xx.x) |
| (xx.x) | (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) |
| (x.xx) xx | (xx.x) xx | xx (xx.x) | (xx.x) xx | xx (xx.x) |
| (xx.x) | (xx.x) | (xx.x) | (xx.x) | xx (xx.x) |
| (x.xx) xx | xx (xx.x) | (x.xx) xx | xx (xx.x) | (x.xx) xx |
| ×× | ×× | ×× | ×× | ×× |
| AA8488\Biostat | istics\Documenta | ation\SAP\Verona | RPL554-MD-201 T | LF Shells v2.0 |
| | | | | Version: 2.0<br>Date: 22JAN2021 |
| | xx | XX | XX XX XX XXX XX.XX (XX.XX) (XX.XX) XX (XX.XX) XX | xx |

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y

Part B

Table 14.1.14

COPD and Smoking History

(All Randomized Analysis Set in Part B)

| Variable/ | RND | SAF | FAS | CAS | PK |
|-----------|--------|--------|--------|--------|--------|
| Category | N=XX | N=XX | N=XX | N=XX | N=XX |
| Mean | ××.× | ×. ×. | ×.×× | ×. × | ×.× |
| SD | ××.×× | ××.×× | xx.xx | xx.xx | xx.xx |
| Median | x.xx | ×.×× | x.xx | x.x. | ××.× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

COPD: Chronic obstructive pulmonary disease. SD: Standard deviation. n = Number of patients calculated relative to the total number of patients. N = Number of patients in the analysis set.

Smoking exposure (pack-years) = Number of packs per day x Number of years smoking, for patients with a smoking history or a current

Duration of COPD (years) (time since diagnosis) = (Randomization date - first COPD diagnosis date) / 365.25.

All Randomized Analysis Set in Part B (RND): Randomized patients in Part B.

Safety Analysis Set (SRF): Randomized patients who received at least one dose of study medication.

Full Analysis Set (RAS): Patients included in the Safety Analysis Set with sufficient data to compute the pharmacodynamic

parameters on at least two treatment periods. Completes and treatment periods i.e. a patient who completers Analysis Set (CAS): Patients included in the Safety Analysis Set who complete all treatment periods i.e. a patient who receives a first and last dose intake plus I day for all 4 treatment periods per schedule of events.

Pharmacokinetics Analysis Set (PK): Patients included in the All Randomized Analysis Set who have a blood sampling performed after at least one dose of study medication and pharmacokinetic parameter data.

Source: Listing 16.2.4.9

Output ID: MH001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.1.15 Drug Exposure and Accountability (Safety Analysis Sets in Part B) Verona Pharma

Protocol: RPL554-MD-201

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Drug Exposure and Accountability (Safety Analysis Set in Part B) Table 14.1.15

| Variable/ | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo | Overall |
|---|---|---|---|---|---|
| Category | N=XX | N=XX | N=XX | N=XX | N=XX |
| Duration of exposure (days) [a] | | | | | |
| п | × | ×× | ×× | ×× | ×× |
| Mean | ×.×. | x.xx | ×. ×× | ×. × | ×. ×. |
| SD | xx.xx | xx.xx | xx · xx | xx.xx | xx.xx |
| Median | x.xx | x.xx | ×.× | ×. × | ×. ×. |
| Min, Max | xx 'xx | xx 'xx | xx 'xx | xx, xx | xx, xx |
| Drug accountability (weight of pMDI used (g)) | | | | | |
| п | ×× | × | ×× | ×× | ×× |
| Mean | x.xx | x.xx | ×. ×× | ×.×. | ×. ×. |
| SD | XX.XX | XX.XX | XX.XX | xx.xx | xx.xx |
| Median | x.x. | x.xx | ×. ×× | ×. ×. | ×. ×. |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

SD: Standard deviation.
Study medication administration and accountability data are from the Drug Accountability eCRF page.

Study medication of exposure per period (days) = (Date of last study medication administration - date of first study medication administration + 1).

[b] Drug accountability (weight of pMDI used (g)) = Weight of pMDI dispensed - weight of pMDI returned, including those dispensed and taken on site.

Source: Listing 16.2.5.2

Output ID: DA001

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

14.2 Efficacy

Primary Efficacy Table 14.2.5 FEV, by Treatment and Timepoint (Full Analyis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

Table 14.2.5 FEV1 by Treatment and Timepoint (Full Analysis Set in Part B)

| Day 1 Timepoint 1-hour pre- dose Immediately pre-dose 5 mins post- dose | Treatment ground | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | treatment group | Category | п | Mean | SD | Minimum | Median | Maximum |
| Immediately pre-dose 5 mins post- dose | RPL554 300µg (N=XX) | Result | ×× | x.xx | xx.xx | xx.xx | × | ×. ×. |
| Immediately pre-dose 5 mins post- dose | RPL554 1000µg (N=XX) | Result | × | ×. × | xx.xx | xx.xx | ×. ×. | ×.<br>×. |
| Immediately pre-dose 5 mins post- dose | RPL554 3000µg (N=XX) | Result | × | ×. ×. | xx.xx | xx.xx | × × × | ×. ×. |
| Immediately pre-dose 5 mins post- dose | Placebo (N=XX) | Result | × | ×.<br>×. | xx · xx | xx.xx | × × × | ×.<br>×. |
| pre-dose 5 mins post-dose | | | | | | | | |
| <br>5 mins post-<br>dose | RPL554 300µg (N=XX) | Result | ×× | x.xx | xx.xx | xx.xx | ×. ×. | ×.×× |
| 5 mins post-<br>dose | I | I | ı | ŧ | I | Ī | i | i |
| 5 mins post-<br>dose | | | | | | | | |
| | RPL554 300µg (N=XX) | Result | × | ××× | xx.xx | xx · xx | × | ×. × |
| | | Pre-dose | × | x.x.x | xx.xx | xx.xx | ×. ×. | ××.× |
| | | Change from Pre-dose | × | × · · × | xx.xx | xx.xx | ×. ×. | ×. ×. |
| 1 | 1 | | 1 | ŧ | i | i | 1 | 1 |

SD: Standard deviation. FEV;: Forced expiratory volume in 1 second.

n = Number of patients who have an assessment available at the relevant post-dose assessment timepoint (Result). n = Number of patients who have an assessment available at Pre-dose and the relevant post-dose assessment timepoint (Pre-dose and Change from Pre-dose). N = Number of patients in the analysis set.

Pre-dose, N = Number of patients in the analysis set.

Pre-dose, highest FEV; result collected immediately pre-dose (within 5 minutes). Change from Pre-dose: Post-dose assessment - Baseline.

Source: Listing 16.2.6.5

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Display for the following days and timepoints, relative to dosing:

Day 1-1 hour pre-dose and immediately pre-dose, 5 ( $\pm$  2), 15 ( $\pm$  5) and 30 minutes ( $\pm$  10) and 1, 1.5, 2, 4, 8 and 12 hours (the latter assessments all  $\pm$  15 minutes).

Day 7-1 hour pre-dose and immediately pre-dose, 30 minutes ( $\pm$  10) and 1, 1.5, 2, 4, 8, 11 and 12 hours (the latter assessments all  $\pm$  15 minutes). Programming Notes

Output ID: EFF003

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.2.6 Change from Baseline FEV; to Peak FEV; (over 4 hours) on Day 7 (Full Analysis Set in Part B) Verona Pharma Protocol: RPL554-MD-201

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

Change from Baseline FEV1 to Peak FEV1 (over 4 hours) on Day 7 Table 14.2.6

(Full Analysis Set in Part B)

| | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo |
|---|---|---|---|---|
| Day 7 | N=XX | N=XX | N=XX | N=XX |
| Baseline FEV1 (L) | | | | |
| n [a] | ×× | XX | ×× | ×× |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | x.xx | x.xx | ×.×. | ×.×× |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Peak FEV1 (L) | | | | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | ×.×. | x.xx | ×.×. | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Change from Baseline ${\rm FEV_1}$ | | | | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | ×.×. | XX.XX |
| Min, Max | xx, xx | xx, xx | xx, xx | xx 'xx |
| Estimates from ANCOVA [b] | | | | |
| n [c] | ×× | XX | XX | ×× |
| GeoMean | x.xx | x.xx | ×.×× | ×. ×. |
| 95% CI for GeoMean | (xx, x, xx) | (xxx, xxxx) | (xxx, xxxx) | (xxx, xx.x) |

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp


Verona Pharma plc

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Part B

Page X of Y

Change from Baseline FEV1 to Peak FEV1 (over 4 hours) on Day 7

(Full Analysis Set in Part B)

| | RPL554 300µg | RFL554 1000µg | RPL554 3000µg | Placebo |
|---|---|---|---|---|
| Day 7 | N=XX | N=XX | N=XX | N=XX |
| Comparisons Against Placebo | | | | |
| Treatment Effect - ANCOVA [c] | | | | |
| GeoMean Ratio | xx.x | xx.x | XX.X | |
| 95% CI for GeoMean Ratio | (xx.x, xx.x) | (xx.x, xx.x) | (xxx, xx.x) | |
| p-value | x.xxx | x xxxx x | X . X X X X | |
| Comparisons Against RPL554 doses | | | | |
| Treatment Effect - ANCOVA [c] | | Comparison Against<br>RPL554 300µg | Comparison Against<br>RPL554 1000µg | |
| GeoMean Ratio | | xx.x | XX.X | |
| 95% CI for GeoMean Ratio | | (xxx, xxxx) | (xxx, xx.x) | |
| p-value | | X.XXX | XXXXX.X | |

ANCOVA: Analysis of covariance. CI: Confidence interval. FEV;: Forced expiratory volume in 1 second. GeoMean: Geometric mean atio. SD: Standard deviation.

Na Number of patients in the analysis set.

Ratio: Geometric mean ratio. SD: Standard deviation.

Na Number of patients in the analysis set.

Baseline: average of the FEV; pre-dose assessments collected on Day 1 (within 60 and 5 minutes).

[a] number of patients with valid values at baseline and peak.

[b] ANCOVA model is used to model the change from baseline using baseline FEV; as a continuous fixed effect and planned treatment and treatment period as categorical fixed effects.

[c] number of patients with at least one on treatment value who contributed to the model estimation.

\* Indicates a significant adjusted p-value (<0.05).

Source: Listing 16.2.6.6

Output ID: EFF004

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc Table 14.2.6a Change from Baseline FEV, to Peak FEV, (over 4 hours) on Day 7 - Sensitivity Analysis (Completers Analysis Set in Part B)

EFF005: This output uses shell EFF004 [Table 14.2.6]

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Version: 2.0 Date: 22JAN2021 Author: Jennifer Allsopp

Table 14.2.7 Average FEV; by Day and Treatment Group (Full Analysis Set in Part B) Secondary Efficacy

EFF006: This output uses shell EFF003 [Table 14.2.5]

AUC: Area under the curve. SD: Standard deviation.

In a Number of patients who have an assessment available at the relevant post-dose assessment timepoint (Result). In a Number of patients who have an assessment available pre-dose and the relevant post-dose assessment timepoint (Pre-dose and Change from Pre-dose). In Number of patients in the analysis set.

Pre-dose: average of the FEV; pre-dose assessments (-60 minutes and -5 minutes). Change from Pre-dose: Post-dose assessment - Pre-dose. Apatient misses' the last two assessments in the time interval measured, or does not have any pre-dose assessments the AUC is set to missing.

Source: Listing 16.2.6.6

Replace footnotes in original shell with tha listed above. Amend the presentation to AUC. To be presented for both AUC<sub>0-13</sub>, and AUC<sub>0-13</sub>, on Day 1 and Day 7, respectively. Programming Notes

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Version: 2.0 Date: 22JAN2021 Author: Jennifer Allsopp

```
ANCOVA: Analysis of covariance. AUC: Area under the curve. CI: Confidence interval. FEV: Forced expiratory volume in 1 second. GeoMean: GeoMean Ratio: Geometric mean ratio. SD: Standard deviation.

N = Number of patients in the analysis set.

Baseline: average of the FEV; pre-dose assessments collected on Day 1 (within 60 and 5 minutes).

[a] number of patients with valid values at baseline and average.

[b] ANCOVA model is used to model the change from baseline AUCo-t using baseline FEV; as a continuous fixed effect and actual treatment pariod as categorical fixed effects.

[c] number of patients with at least one on treatment value who contributed to the model estimation.

* Indicates a significant adjusted p-value (<0.05).
Table 14.2.8 Change from Baseline FEV; to Average FEV; (over 4 hours) on Day 7 (Full Analysis Set in Part B)
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                            Replace footnotes in original shell with those listed above.
                                                                                                                                                                                              EFF007: This output uses shell EFF004 [Table 14.2.6]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             Source: Listing 16.2.6.6
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                  Programming Notes
```

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B Author: Jennifer Allsopp

```
Version: 2.0
Date: 22JAN2021
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                     Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0
- Part B
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        Table 14.2.9a Change from Baseline FEV1 to Average FEV1 (over 12 hours) on Day 7 - Sensitivity Analysis (Full Analysis Set in Part B)
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                  Baseline: average of the FEV; pre-dose assessments collected on Day 1 (within 60 and 5 minutes).

[a] number of patients with valid values at baseline and average.

[b] ANCOVA model is used to model the change from baseline AUC0-t using baseline FEV; as a continuous fixed effect and actual treatment period as categorical fixed effects.

[c] number of patients with at least one on treatment value who contributed to the model estimation.

* Indicates a significant adjusted p-value (<0.05).
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                         [a] number of patients with valid values at baseline and average.

[b] ANCOVA model is used to model the change from baseline AUG. tusing baseline FEV, as a continuous fixed effect and actual treatment and treatment period as categorical fixed effects.

triangular to fine patients with at least one on treatment value who contributed to the model estimation.

* Indicates a significant adjusted p-value (<0.05).
                                                                                                                                                                                                                                                                                                                                                                                           ANCOVA: Analysis of covariance. AUC: Area under the curve. CI: Confidence interval. FEV; Forced expiratory volume in 1 second. GeoMean: Geometric mean. GeoMean Ratio: Geometric mean ratio. SD: Standard deviation.

N = Number of patients in the analysis set.
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        ANCOVA: Analysis of covariance. AUC: Area under the curve. CI: Confidence interval. FEV1: Forced expiratory volume in 1 second. GeoMean: Geometric mean. Geometric mean ratio. SD: Standard deviation.
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                    Replace footnotes in original shell with those listed above Only include if at least 1 subject has taken rescue medication less than 6 hours prior to spirometry (ANLO2FL="Y")
Table 14.2.9 Change from Baseline FEV; to Average FEV; (over 12 hours) on Day 7 (Full Analysis Set in Part B)
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                           N = Number of patients in the analysis set. Baseline: average of the \rm FEV_1 pre-dose assessments collected on Day I (within 60 and 5 minutes). Includes subjects who took rescue medication less than 6 hours prior to spirometry.
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      Replace footnotes in original shell with those listed above
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          EFF009: This output uses shell EFF004 [Table 14.2.6]
                                                                                                                                                                                                           EFF008: This output uses shell EFF004 [Table 14.2.6]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                     Source: Listing 16.2.6.6
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        Source: Listing 16.2.6.6
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                      Author: Jennifer Allsopp
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                       Programming Notes
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          Programming Notes
```

```
ANCOVA: Analysis of covariance. CI: Confidence interval. FEV: Forced expiratory volume in 1 second. GeoMean: Geometric mean. Ratio. So Standard deviation.

Ratio: Geometric mean ratio. SD: Standard deviation.

N = Number of patients in the analysis set.

Baseline: average of the FEV; pre-dose assessments collected on Day I (within 60 and 5 minutes).

Morning trough FEV; is the average of the FEV; pre-dose assessments (-60 minutes and -5 minutes) on Day 7.

[a] number of patients with valid values at baseline and morning trough FEV; using baseline FEV; as a continuous fixed effect, actual treatment and treatment begind as categorical fixed effects.

[c] number of patients with at least one on treatment value who contributed to the model estimation.

* Indicates a significant p-value (<0.05).
Table 14.2.10 Change from Baseline FEV; to Morning Trough FEV; on Day 7 (Full Analysis Set in Part B)
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             Replace footnotes in original shell with those listed above
                                                                                                                                                                                                    EFF0010: This output uses shell EFF004 [Table 14.2.6]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               Source: Listing 16.2.6.6
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          Programming Notes
```

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc
```
Version: 2.0
Date: 22JAN2021
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                              Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                  Table 14.2.13 Change from Baseline FEV, to Average FEV, (over 12 hours) on Day 1 (Full Analysis Set in Part B)
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                             Table 14.2.12 Change from Baseline FEV, to Average FEV, (over 4 hours) on Day 1 (Full Analysis Set in Part B)
Table 14.2.11 Change from Baseline FEV, to Peak FEV, (over 4 hours) on Day 1 (Full Analysis Set in Part B)
                                                                                                                                           EFF11: This output uses shell EFF004 [Table 14.2.6]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               EFF12: This output uses shell EFF006 [Table 14.2.8]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                        EFF13: This output uses shell EFF007 [Table 14.2.9]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                              Footnotes should be the same as Table 14.2.9
                                                                                                                                                                                                                                                                                                                                                                                                                 Footnotes should be the same as Table 14.2.6
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          Footnotes should be the same as Table 14.2.8
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                           Author: Jennifer Allsopp
                                                                                                                                                                                                                                                                                                                                                 Programming Notes
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                               Programming Notes
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                          Programming Notes
```

Table 14.2.14 Time to Onset of Action (>10% Increase in FEV1) on Day 1 (Full Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

Time to Onset of Action (>10% Increase in FEV1) on Day 1 (Full Analysis Set in Part B) Table 14.2.14

| | | RPL554 300µg | RPL554 1000µg | RPL554 3000µg |
|---|---|---|---|---|
| Parameter | Statistics | N=XX | N=XX | N=XX |
| Number of patients with onset of action | n (%) | (x.x) xx | xx (xx.x) | xx (xx.x) |
| Number of patients censored | n (%) | (x.x.x) | xx (xx.x) | xx (xx.x) |
| Time to onset of action (mins) | P25 | × : | ××× | ××× |
| | Median (Min, Max) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| | P75 | × | × | ×.× |
| | Hodges-Lehmann Median difference<br>to RPL554 3000µg | × ; | × ; | |
| | p-value | × ×××× | ×.xxxx | |

n = Number of patients with onset of action. % = Percentage of patients calculated relative to the total number of patients in the mailysis set.

Time to onset of action (mins): Time of onset of action (defined as >10% increase in FEV; from pre-first dose) = Time of onset of action (or censoring time) - time of end of inhalation (mins).

25.5, Median and P75: Patients not experiencing onset of action are censored at 120 mins or at time of premature discontinuation (if withdrawn before 120 minutes).

(if withdrawn before 120 minutes).

Source: Listing 16.2.6.7

Programming Notes

Only present if the number of onset of action cases are sufficient to calculate the statistics presented (2 10% of patients with onset of action). The pre-dose value is inserted at time 0.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

Time to Onset of Action (>10% Increase in FEV;) on Day  $1\,$ 

(Full Analysis Set in Part B)

| RPL554 3000µg | N=XX |
|---------------|------------|
| RPL554 1000µg | N=XX |
| RPL554 300µg | N=XX |
| | Statistics |
| | Parameter |

Output ID: EFF14

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

 Verona Pharma plc


Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.2.15 Rescue Medication Use (Full Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.2.15

(Full Analysis Set in Part B) Rescue Medication Use

| | Maximum | × | ×. ×. |
|------------|-----------------|---------------------|----------------------|
| | Median | ××. | ×. ×. |
| cics | Minimum | ××.×× | xx.xx |
| Statistics | SD | XX.XX | xx.xx |
| | Mean | ×.×. | ×: × |
| | и | ×× | ×× |
| | Category | Result | Result |
| | Treatment group | RPL554 300µg (N=XX) | RPL554 1000µg (N=XX) |

xx.xx xx.xx xx.xx

××.× ××. ×.×

× × ×

Result Result Result

RPL554 3000µg (N=XX)

Placebo (N=XX)

××.×

××.× ×. ×

xx.xx xx.xx

SD: Standard deviation. n = Number of patients who have an assessment available at the relevant post-dose assessment timepoint (Result). N = Number of patients in the analysis set. The average number of puffs of rescue medication taken per day between days 1 and 7 (inclusive) for each treatment period was collected in the patient diaries.

Source: Listing 16.2.6.9

Programming Notes

Use information from the patient diarys (number of puffs). For each treatment period calculate the average of the 7 days. If less than 4 days have results between days 1 and 7 then no result will be presented for that treatment period.

Output ID: EFF15

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

Table 14.2.16 Dyspnea Scale by Day and Timepoint (Full Analysis Set in Part B) Exploratory Efficacy Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

Dyspnea Scale by Day and Timepoint (Full Analysis Set in Part B) Table 14.2.16

| um Median Maximum | x.xx xx.x x | x.xx x x x x | x.xx xx.x | x.xx x x x x x | x.xx | x.xx xx.x | x.xx x x x x x | x x x x x x x x x x x x x x x x x x x | : | × | : |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Minimum | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | : | xx.xx | : |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | xx.xx | : | xx.xx | : |
| n Mean | xx xx.x | xx.xx | xx xx.x | xx xx.x | xx xx.x | xx xx.x | xx xx.x | xx xx x | : | xx.xx | : |
| Category | Result | Result | Result | Result | Result | Baseline x | CFB | Result | | Result x | |
| Treatment group | RPL554 300µg (N=XX) | RPL554 1000µg (N=XX) | RPL554 3000µg (N=XX) | Placebo (N=XX) | RPL554 300µg (N=XX) | | | RPL554 1000µg (N=XX) | : | RPL554 300µg (N=XX) | 1 |
| Timepoint | Pre-dose | | | | 30 mins post-dose | | | | | 1 hour post-dose | |
| Day | Day 1 | | | | | | | | | | |

CFB: Change from Baseline. SD: Standard deviation.

n = Number of patients who have an assessment available at the relevant post-dose assessment timepoint (Result). n = Number of patients who have an assessment available at Baseline and the relevant post-dose assessment timepoint (Baseline and Change from Baseline). N = Number of patients in the analysis set.

Baseline dyspines score is defined as the value of dyspinea assessed prior to dosing on day 1 of treatment period 1.

Change from Baseline: Post-dose assessment - Baseline.

Source: Listing 16.2.6.8

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Table 14.2.16

Part B Page X of Y

Dyspnea Scale by Day and Timepoint

(Full Analysis Set in Part B)

| | Maximum | ×.×× |
|------------|-----------------|---------------------|
| | Median | × × × |
| Statistics | Minimum | ××. |
| | SD | xx.xx |
| | Mean | ××× |
| | и | × |
| | Category | Result |
| | Treatment group | RPL554 300µg (N=XX) |
| | Timepoint | Pre-dose |
| | Day | Day 1 |

Programming Notes Display for the following day and timepoints, relative to dosing: Day 1-30 minutes and 1, 1.5, 2, 4, 8 and 12 hours post-dose Day 7-30 minutes and 1, 1.5, 2, 4, 8, 11 and 12 hours post-dose

Output ID: EFF16

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA84488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B Author: Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Table 14.2.17 Comparison of Change from Baseline Dyspnea Score by Day and Timepoint (Full Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

 $\mbox{Table 14.2.17} \\ \mbox{Comparisons of Change from Baseline Dyspnea Score by Day and Timepoint}$ 

(Full Analysis Set in Part B)

| | | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo |
|---|---|---|---|---|---|
| Day Timepoint | Statistic | N=XX | N=XX | N=XX | N=XX |
| Day 1 Pre-dose | Baseline Dyspnea Score | | | | |
| | n [a] | ×× | ×× | ×× | XX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | x.x. | x.xx | x.x. | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| Day 7 Pre-dose | Dyspnea Score | | | | |
| | и | ×× | ×× | ×× | ×× |
| | Mean (SD) | xx.xx) x.xx | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | ×.× | ×. ×. | × · × × | ×.×× |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| | CFB Dyspnea Score | | | | |
| | Mean (SD) | xx.xx) x.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | x. xx | x. x | x . x x | x.xx |
| | Min, Max | xx, xx | xx, xx | xx, xx | xx, xx |
| | Estimates from ANCOVA [b] | | | | |
| | n [c] | ×× | ×× | ×× | XX |
| | LSMean | ×.×× | ×.×× | × · × × | x. xx |
| | 95% CI for LSMean | (xx.x, xx.x) | (xxx, xxxx) | (xxx, xxxx) | (xxx, xxxx) |

Document: \\ieedc-vnasc01\\biosdata\Verona\_Pharma\RPL554\EZAA8488\\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

Comparisons of Change from Baseline Dyspnea Score by Day and Timepoint

(Full Analysis Set in Part B)

| N=XX | | RPL554 300µg | | | Placebo |
|---|---|---|---|---|---|
| Comparisons Against Placebo Treatment Effect - ANCOVA [c] LSMean Diff Comparisons Against RPL554 doses Comparisons Against RPL554 doses Comparison Treatment Effect - ANCOVA [c] LSMean Diff LSMean Diff Comparison Treatment Diff Comparison Comparison Comparison Against RPL554 Against RPL554 Bology LSMean Diff Comparison Against RPL554 Comparison Comparison Accordance Comparison Against RPL554 Against RPL554 Bology Comparison Comparison Accordance Accordance Comparison Accordance Accordan | Statistic | N=XX | N=XX | N=XX | N=XX |
| Treatment Effect - ANCOVA [c] LSMean Diff (xx.x, xx.x) | Comparisons Against Placebo | | | | |
| LSMean Diff | Treatment Effect - ANCOVA [c] | | | | |
| 95% CI for LSMean Diff | LSMean Diff | x.x. | x. xx | x . x . | |
| D-value X.xxxx X.xxx X.xxxx X. | 95% CI for LSMean Diff | (xx.x, xx.x) | (xx.x, xx.x) | (xxx, xx.x) | |
| Comparisons Against RPL554 doses Comparison Treatment Effect - ANCOVA [c] Sology LSMean Diff xx.x 95% CI for LSMean Diff xx.xx p-value | p-value | x.xxx | x.xxxx | x.xxxx | |
| Treatment Effect - ANCOVA [c] Comparison Comparison Against RPL554 Against RPL554 300µg xx.x 95% CI for LSWean Diff (xx.x, xx.x) p-value x.xxxx x.xxxxx.x.x.x.x.x.x.x.x.x.x.x.x | Comparisons Against Rrioo4 doses | | | | |
| LSMean Diff S5% CI for LSMean Diff (xx.x, xx.x) (xx.x, xx.x) (xx.x, xx.x) (xx.x, xx.x) (xx.x, xx.x) (xx.x, xx.x) | Treatment Effect - ANCOVA [c] | | Comparison<br>Against RPL554<br>300µg | Comparison<br>Against RPL554<br>1000µg | |
| 95% CI for LSMean Diff p-value | LSMean Diff | | ××.×× | x.xx | |
| p-value x.xxxx x.xxxx | 95% CI for LSMean Diff | | (xx.x, xx.x) | (xxx, xx.x) | |
| | p-value | | X.XXXX | x.xxxx | |
| | i | : | : | | |

ANCOVA: Analysis of covariance. CFB: Change from Baseline. CI: Confidence interval. LSWean: Least square mean. LSWean Diff: Least squares mean difference. SD: Standard deviation.

N = Number of patients in the analysis set. n = Number of patients who have an assessment available pre-dose and the relevant post-baseline timepoint. Baseline: Day 1 pre-dose Dyspnea Score.

[a] number of patients with valid values at baseline and post-baseline.

[b] ANCOVA model is used to model the change from baseline using baseline Dyspnea Score as a continuous fixed effect and planned treatment particd as categorical fixed effects.

[c] number of patients with at least one on treatment value who contributed to the model estimation.

\* Indicates a significant adjusted p-value (<0.05).

Source: Listing 16.2.6.8

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp


Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

#### Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

Comparisons of Change from Baseline Dyspnea Score by Day and Timepoint Table 14.2.17

(Full Analysis Set in Part B)

### Placebo N=XX RPL554 3000µg N=XX RPL554 1000µg N=XX RPL554 300µg N=XX Statistic Timepoint

Programming Notes

Display for the following day and timepoints, relative to dosing: Day 1 - Pre-dose (Baseline), 30 minutes and 1, 1.5, 2, 4, 8 and 12 hours post-dose Day 7 - Pre-dose, 30 minutes and 1, 1.5, 2, 4, 8, 11 and 12 hours post-dose

Output ID: EFF17

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

CONFIDENTIAL Verona Pharma plc

14.3 Safety Adverse Event Table 14.3.27 Treatment-emergent Adverse Events Summary (Safety Analysis Set in Part B)

Page X of Y Part B

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Treatment-emergent Adverse Events Summary (Safety Analysis Set in Part B) Table 14.3.27

| | Щ | RPL554 | | RPL554 | | 174 | RPL554 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 300µg | | 1000µg | | ίŋ | 3000µg | | Д | Placebo | 0 | _ | Overall | |
| Variable/ | | N=XX | | N=XX | | | N=XX | | | N=XX | | | N=XX | |
| Category | E E | n (%) E | | n (%) E | | Д | (%) | | ď | (%) | 田 | | I (%) I | 团 |
| Any TEAE | × | xx (xx.x) xx | × | (x.xx) xx | × | ×× | xx (xx.x) x | × | ×× | xx (xxxx) xx | × | × | xx (xx.x) | × |
| Any TEAE related to study medication | × | (xx.x) | × | (xx.x) | × | ×× | xx (xx.x) | ×× | )<br>XX | (xx.x) | ×× | × | (xxx) | × |
| Any TEAE leading to study discontinuation | × | (xx.xx) | × | (x x x) | × | ×× | xx (xx.x) x | × | ×× | xx (xx.x) xx | × | × | (xx.x) | × |
| Any TEAEs classified by maximum severity, n (%) | | | | | | | | | | | | | | |
| Mild | × | xx (xx.x) | × | (xx.x) | | .)<br>XX | (xx.x) | | ×× | xx (xx.x) | | × | xx (xx.x) | |
| Moderate | × | (xx.x) | × | (x.xx) xx | | <br>×× | (xxx) xx | | ×× | xx (xx.x) | | × | (×××) | |
| Severe | × | (xx.x) | × | (xx.x) | | .)<br>×× | (xx.x) | | ×× | xx (xx.x) | | × | (xx.x) | |
| Any TEAE leading to death | ×× | (xx xx) | × | (xx.x) | ×× | ×× | xx (xx.x) x | ×× | ×× | (xx.x) | ×× | × | (xx.x) | × |
| Any serious TEAE | ×× | (x.xx) | × | (x.xx) xx | × | .)<br>×× | xx (xx.x) x | × | ×× | xx (xx.x) | ×× | × | (xx.x) | × |
| Any serious TEAE related to study medication | × | xx (x.xx) | × | (x · xx) xx | × | <br>× | xx (xx.x) x | × | ×× | xx (xx.x) xx | × | × | (xx.x) | × |
| Any serious TEAE leading to study discontinuation | × | (x.x) | × | (x : xx) | × | )<br>×× | xx (xx.x) | × | ×× | (xx.x) | × | × | (xx.x) | × |
| Any serious TEAEs classified by maximum severity, n (%) | | | | | | | | | | | | | | |
| Mild | ×× | (xx.x) | × | (x.xx) xx | | ×× | (xx.x) | | ×× | xx (xx.x) | | × | xx (xx.x) | |
| Moderate | × | (xx.x) | × | (x.xx) xx | | ×× | xx (xx.x) | | ×× | xx (xx.x) | | × | xx (xx.x) | |
| Severe | × | (xx.x) | × | xx (xx.x) | | ×× | xx (xx.x) | | ×× | xx (xx.x) | | × | xx (xx.x) | |
| Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B | ZAA848 | 8\Biostat | istic | s\Docum | entat | ion\9 | SAP\Ve | rona | RPL55 | .4-MD | 201 TL | E SF | ells v | 2.0 |
| Author Tonnifor Alloom | | | | | | | | | | | | > | Version: 2.0 | . 2 |

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Part B Page X of Y

Treatment-emergent Adverse Events Summary

(Safety Analysis Set in Part B)

| | RPL554 | RPL554 | RPL554 | | |
|-----------|---------|---------|---------|---------|---------|
| | 300µg | 1000μg | 3000μg | Placebo | Overall |
| Variable/ | N=XX | N=XX | N=XX | N=XX | N=XX |
| Category | n (%) E | n (%) E | n (%) E | n (%) E | n (%) E |

TEAE: Treatment-emergent adverse event.

TEAE: Treatment-emergent adverse event.

In Number of patients with at least one TEAE in each category. E = Number of mentions (events) in each category. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis set. TEAE = All AEs that started or worsened in severity on or after the first dose of study medication, based on the investigator assessment of severity.

TEAES with a missing relationship to study medication will be regarded as related to study medication.

TEAES starting after the first dose of study medication with a missing severity will be classified as severe.

Overall group TEAEs are independent of treatment group. Overall = Presented for all patients in the Safety Analysis Set.

Source: Listing 16.2.7.6

Output ID: AE001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.3.28 Treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part B)

Part B Page X of Y

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.28

Treatment-emergent Adverse Events by System Organ Class and Preferred Term

(Safety Analysis Set in Part B)

| System Organ Class (%) | RPL554 300µg | RPL554 300µg RPL554 1000µg RPL554 3000µg | RPL554 3000µg | Placebo | Overall |
|---|---|---|---|---|---|
| Preferred Term (%) [a] | N=XX | N=XX | N=XX | N=XX | N=XX |
| Patients with at least one TEAE, n (%) E | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (x.x.) xx |
| System Organ Class #1 | (xx.x) xx | (x · xx) | xx (xx.x) | (xxx) xx | xx (xx.x) |
| Preferred Term #1 | (x.xx) xx | (x.xx) xx | (x.xx) xx | (xx.x) | (x.xx) xx |
| Preferred Term #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | (xx.x) | xx (xx.x) |
| Preferred Term #1 | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Preferred Term #2 | xx (xx.x) | (xx.x) | (xx.x) xx | (xx.x) | (xx.x) |

PT: Preferred term. SOC: System organ class. TEAE: Treatment-emergent adverse event.

n = Number of patients with at least one TEAE in each category. E = Number of mentions (events) in each category. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis set.

TEAE = All ABES that started or worsened in severity on or after the first dose of study medication, based on the investigator assessment of severity.

Each patient is counted once for each applicable specific AE, and a patient with multiple AEs within an SOC is counted once for that

[a] SOCs and PTs are coded using the MedDRA (Version 21.0).

Source: Listing 16.2.7.6

Programming Notes

SOCs and PTs within each SOC are sorted in descending order of percentage in the Overall group.

Output ID: AE002

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp


Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

#### Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

Table 14.3.28

Treatment-emergent Adverse Events by System Organ Class and Preferred Term

(Safety Analysis Set in Part B)

| System Organ Class (%) | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo | Overall |
|---|---|---|---|---|---|
| Preferred Term (%) [a] | N=XX | N=XX | N=XX | N=XX | N=XX |

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

CONFIDENTIAL Verona Pharma plc

Table 14.3.29 Treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part B)

AE003: This output uses shell AE002 [Table 14.3.28]

PT: Preferred term. SOC: System organ class. TEAE: Treatment-emergent adverse event.

n = Number of patients with at least one related TEAE in each category. E = Number of mentions (events) in each category. N = Number of patients in the analysis set.

TEAE = All AED the analysis set.

TEAE = All AED that the analysis set.

TEAE = All AED that started or worsened in severity on or after the first dose of study medication, based on the investigator sassesment of related or not.

Each patient is counted once for each applicable specific AE, and a patient with multiple AES within an SOC is counted once for that SOC.

[a] SOCs and PTs are coded using the MedDRA (Version 21.0).

Source: Listing 16.2.7.6

Programming Notes:

Replace footnotes in original shell with those listed above

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Table 14.3.30 Treatment-emergent Adverse Events by System Organ Class and Preferred Term and Maximum Severity (Safety Analysis Set in Part B)

Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.30

Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity

(Safety Analysis Set in Part B)

| | Maximum | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo | Overall |
|---|---|---|---|---|---|---|
| Preferred Term, n (%) [a] | Severity | N=XX | N=XX | N=XX | N=XX | N=XX |
| Patients with at least one TEAE, n (%) | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | (x.xx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class #1 | Severe | xx (xx.x) | xx (xx.x) | (x.xx) xx | (x.xx) xx | (x.xx) xx |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | (xx.x) xx | xx (xx.x) | xx (xx.x) |
| Preferred Term #1 | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term #2 | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | (xxx) xx | xx (xx.x) | xx (xx.x) |
| System Organ Class #2 | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Moderate | xx (xx.x) | xx (xx.x) | (xx.x) xx | xx (xx.x) | xx (xx.x) |
| | Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ī | 1 | : | : | | : | : |

PT: Preferred term. SOC: System organ class. TEAE: Treatment-emergent adverse event. n = Number of patients with at least one TEAE in each category. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis set.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Part B Page X of Y

Treatment-emergent Adverse Events by System Organ Class, Preferred Term and Maximum Severity

(Safety Analysis Set in Part B)

| N=XX | Severity |
|------|----------|

TEABE = All AES that started or worsened in severity on or after the first dose of study medication, based on the investigator assessment of severity.

Bach patient is counted once for each applicable specific TEAE at the maximum severity and a patient with multiple TEAEs within an SOC is counted once for that SOC at the maximum severity.

[a] SOCs and PTS are coded using MedDRA (Version 21.0).

TEAES starting after the first dose of study medication with a missing severity will be classified as missing.

Versall = Presented for all patients in the Safety Analysis Set. Source: Listing 16.2.7.6

SOCs and PTs within each SOC are sorted in descending order of percentage in the Overall group.> Programming Note Output ID: AE004

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Table 14.3.31 Treatment-emergent Adverse Events Leading to Discontinuation of Study by System Organ Class and Preferred Term (Safety Analysis Set in Part B)

AE005: This output uses shell AE004 [Table 14.3.28]

Use the same template of table 14.3.28, selecting only the TEAEs leading to discontinuation of study medications and update "Any TEAE" to "Any TEAE leading to discontinuation of study".

Update source footnote to "Source: Listing 16.2.7.7". Programming Notes

Table 14.3.32 Serious Treatment-emergent Adverse Events by System Organ Class and Preferred Term (Safety Analysis Set in Part B)

AE006: This output uses shell AE002 [Table 14.3.28]

Replace footnotes in original shell updating "Patients with at least one TEAE" to "Patients with at least one serious TEAE". Update source footnote from to "Source: Listing 16.2.7.9". Programming Notes

Table 14.3.33 Serious Treatment-emergent Adverse Events Related to Study Medication by System Organ Class and Preferred Term (Safety Analysis Set in Part B)

AE007: This output uses shell AE003 [Table 14.3.28]

Use the same template of Table 14.3.28, selecting only the serious TEAEs and update "Patients with at least one TEAE" to "Patients with at least one serious TEAE". Update source footnote from to "Source: Listing 16.2.7.9". Programming Notes

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.3.34 Serious Treatment-emergent Adverse Events by System Organ Class, and Preferred Term and Maximum Severity (Safety Analysis Set in Part B)

AE008: This output uses shell AE004 [Table 14.3.30]

Use the same template of Table 14.3.28, selecting only the serious TEAEs and update "Patients with at least one TEAE" to "Patients with at least one serious TEAE". Update source footnote to "Source: Listing 16.2.7.9". Programming Notes

Table 14.3.35 Serious Treatment-emergent Adverse Events Leading to Discontinaution of Study by System Organ Class and Preferred Term (Safety Analysis Set in Part B)

AE009: This output uses shell AE005 [Table 14.3.28]

Use the same template of Table 14.3.29, selecting only the serious TEAEs and update "Any TEAE leading to discontinuation of study" to "Any serious TEAE leading to discontinuation of study". Also update "n = Number of patients with at least one related TEAE in each category." with at least one serious TEAE leading to discontinuation of study." Update source footnote to "Source: Listing 16.2.7.9". Programming Notes

Table 14.3.36 Treatment-emergent Adverse Events with Outcome of Death by System Organ Class and Preferred Term (Safety Analysis Set in

This output uses shell AE002 [Table 14.3.28] AE010:

Replace footnotes in original shell updating "Patients with at least one TEAE" to "Patients with a TEAE with outcome of death". Update source footnote to "Source: Listing 16.2.7.8". Programming Notes

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

Laboratory Table 14.3.37 Hematology Laboratory Data by Day (Safety Analysis Set in Part B) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Part B

Page X of Y

Hematology Laboratory Data by Day (Safety Analysis Set in Part B) Table 14.3.37

| Laboratory Test | RPL554 | RPL554 | RPL554 | | |
|---|---|---|---|---|---|
| Time Point | 300µg | 1000μg | 3000µg | Placebo | Overall |
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| Test #1 (unit) | | | | | |
| Baseline | | | | | |
| ū | ×× | XX | ×× | ×× | XX |
| Mean | x.x. | ×.×. | XX.X | x. x. | ××.× |
| SD | xx.xx | xx.xx | XX.XX | XX.XX | xx.xx |
| Median | x.xx | x.xx | x.xx | x.xx | xx.x |
| Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| Day 7 | | | | | |
| Observed | | | | | |
| ч | ×× | ×× | ×× | ×× | |
| Mean | ×.×× | ×: ×× | ×××× | ×.×× | |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | |
| Median | ×.×× | ×.×× | ×××× | ×××× | |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | |
| Change from Baseline | | | | | |
| Mean | x.x. | x. x. | x.xx | x. x. | |
| SD | xx.xx | xx.xx | XX.XX | xx.xx | |
| Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 | ata\Verona_Pharma\RPL5 | 54\EZAA8488\Biostatis | tics\Documentation\SAP\ | Verona RPL554-MD-201 | ITLF Shells v2.0 |
| Fair D | | | | | Version: 2.0 |
| Author: Jennifer Allsopp | | | | | Date: 22.JAN2021 |

Date: 22JAN2021 Author: Jennifer Allsopp

Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Table 14.3.37

Part B Page X of Y

Hematology Laboratory Data by Day

(Safety Analysis Set in Part B)

| Laboratory Test | RPL554 | RPL554 | RPL554 | | |
|-----------------|-----------|-----------|-----------|-----------|---------|
| Time Point | 300µg | 1000μg | 3000µg | Placebo | Overall |
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| Median | x.xx | ××.× | ×.×× | ×.×. | |
| Min, Max | x.x, xx.x | x.x, xx.x | x.x, xx.x | x.x, xx.x | |
| Test #2 (unit) | : | | | | |

SD: Standard deviation.

n = Number of patients with a Baseline value and a post-baseline value. N = Number of patients in the analysis set.

Change from Baseline: (Post-baseline assessment - Baseline).

Baseline: Defined as the pre-dose assessment for each treatment period.

Overall: Presented for all patients in the first treatment period in the Safety Analysis Set. Overall n = Number of Baseline values with an assessment available at Baseline and at least one post-dose assessment for treatment period 1.

Source: Listing 16.2.8.5

Programming Notes

Blood samples will be taken and tested at the laboratory for the following hematology laboratory tests: Hemoglobin, hematocrit, total white cell count, leukocyte differential count and platelet count. Present in alphabetical order.

Output ID: LB001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.3.38 Biochemistry Laboratory Data by Day (Safety Analysis Set in Part B)

LB002: This output uses shell LB001 [Table 14.3.37]

Programming Notes

Repeat 14.3.37 for Biochemistry (includes creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine transaminase, gamma-glutamyl transferase, lactate dehydrogenase, creatine kinase, thyroid stimulating hormone, triiodothyronine and thyroxine, glucose, potassium, sodium, calcium. Present in alphabetical order. Update source footnote to "Source: Listing 16.2.8.6".
Add footnote to "A number of missing chemistry labs are due to a processing issues such as hemolyzed samples.".

Table 14.3.39 Urinalysis Laboratory Data by Day (Safety Analysis Set in Part B)

LB007: This output uses shell LB001 [Table 14.3.37]

Repeat 14.3.37 for Urinalysis (includes Leukocytes esterase, occult blood, ketones, bilirubin, urobilinogen, protein and glucose. If urinalysis on Dipstick is positive for leucocytes and/or blood/hemoglobin, a microscopic examination including erythrocytes, leucocytes, bacteria, casts, epithelial cells and crystals). Present in alphabetical order. Update source: Listing 16.2.8.7".

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Page X of Y Table 14.3.40 Hematology Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B)
Verona Pharma

Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Hematology Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B) Table 14.3.40

| | | | | Category at Time Point | ime Point | |
|---|---|---|---|---|---|---|
| Laboratory Test | | | | | | |
| Day | | Baseline | TOW | Normal | High | Total |
| Treatment | N [a] | Category | n (%) | n (%) | n (%) | n (%) |
| Test #1 | | | | | | |
| Day 7 | | | | | | |
| RPL554 300µg | ×× | Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Normal | (xx.x) xx | (x.xx) xx | (x.xx) xx | (xx.x) xx |
| | | High | xx (xx.x) | (x.x.x) | xx (xx.x) | xx (xx.x) |
| | | Total | (x.xx) xx | (x.xx) xx | (x.xx) xx | |
| RPL554 1000µg | ×× | Low | (x.xx) xx | xx (xx.x) | (x.xx) xx | xx (xx.x) |
| | | Normal | (x.xx) xx | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| | | High | (x.xx) xx | xx (xx.x) | (x.xx) xx | (x.xx) xx |
| | | Total | xx (xx.x) | xx (xx.x) | (xx.x) | |
| RPL554 3000µg | × | i | 1 | i | ŧ | i |
| į | | i | Ī | ŧ | i | : |
| | | i | 1 | i | 1 | : |
| | | ŧ | ŧ | į | : | : |
| End of Study | | | | | | |
| Overall | ×× | į | : | į | : | i |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Verona Pharma Protocol: RPL554-MD-201 RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

Table 14.3.40

Hematology Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day

(Safety Analysis Set in Part B)

| | | | | Category at Time Point | Point | |
|---|---|---|---|---|---|---|
| Laboratory Test | | | | | | Ì |
| Day | | Baseline | Low | Normal | High | Total |
| Treatment | N [a] | Category | n (%) | n (%) | n (%) | n (%) |
| | | 1 | 1 | 1 | 1 | 1 |
| | | : | | : | : | : |
| Test #2 | | | | | | |
| I | | | | | | |

LIN: Lower limit of normal reference range. ULN: Upper limit of normal reference range.

n = Number of patients. [a] N = Number of patients with a baseline value and a post-baseline value at the time point. Percentages are based on N.

Reference range classification: Low: < LLN. Normal: >= LLN to <= ULN. High: > ULN.

Baseline: Defined as the pre-dose assessment for each treatment period.

End of Study: Defined as the last available assessment assigned to study. Source: Listing 16.2.8.5

Programming Notes

Blood samples will be taken and tested at the laboratory for the following laboratory tests: Hemoglobin, hematocrit, total white cell count, leukocyte differential count and platelet count. Present in alphabetical order.

Output ID: LB003

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.3.41 Biochemistry Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B)

LB004: This output uses shell LB003 [Table 14.3.40]

Repeat Table 14.3.40 for Biochemistry. Table should present these parameters only: Creatinine, total bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine transaminase, gamma-glutamyl transferase, lactate dehydrogenase, creatine kinase, thyroid stimulating hormone, trilodothyronine and thyroxine, glucose, potassium, sodium, and calcium. Present in alphabetical order. Update source footnote to "Source: Listing 16.2.8.6".
Add footnote "A number of missing chemistry labs are due to a processing issues such as hemolyzed samples.".

Table 14.3.42 Urinalysis Laboratory Data - Shifts from Baseline in Normal Reference Ranges by Day (Safety Analysis Set in Part B)

LB005: This output uses shell LB003 [Table 14.3.40]

Programming Notes

Repeat Table 14.3.40 for Urinalysis, and update category to "Negative' if the results are 'Normal' or 'Negative', to 'Trace' if the results are 'Trace' and 'Positive' if the results are equal to '1+','2+','3+',' or '4+'.

Table should present these parameters only: Leukcoytes esterase, occult blood, ketones, bilirubin, urobilinogen, protein and glucose. If urinalysis on bipstick is positive for leuccoytes and/or blood/hemoglobin, a microscopic examination including erythrocytes, leuccytes, bacteria, casts, epithelial cells and crystals. Present in alphabetical order.

Update source footnote to "Source: Listing 16.2.8.7".

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Table 14.3.43 Biochemistry Laboratory Data - Markedly Abnormal Values (Safety Analysis Set in Part B) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

> Biochemistry Laboratory Data - Markedly Abnormal Values (Safety Analysis Set in Part B) Table 14.3.43

| | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo |
|---|---|---|---|---|
| Laboratory Test, n (%) | N=XX | N=XX | N=XX | N=XX |
| ATTEN CONTRACTOR CONTRACTOR CONTRACTOR | | | | |
| ALGIILIG AMILIOCLAMBLELANG (ALI) | | | | |
| > 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Alkaline Phosphatase (ALP) | | | | |
| > 3 x ULN | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Aspartate Aminotransferase (AST) | | | | |
| > 3 x UIN | (x.xx) xx | xx (xx.x) | xx (xx.x) | (x.x.) xx |
| Creatinine | | | | |
| > 2.5 mg/dL | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Gamma Glutamyl Transferase (GGT) | | | | |
| > 3 x UIN | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Bilirubin (TBL) | | | | |
| > 3 x UIN | (x.xx) xx | (x.xx) xx | (xx.x) | xx (xx.x) |

ULN: Upper limit of normal reference range. n = Number of patients in each category with at least one markedly abnormal value. N = Number of patients in the analysis set. % = Percentage of patients with at least one markedly abnormal value relative to the total number of patients in each treatment group.

Source: Listing 16.2.8.6 Output ID: LB006 [Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Page X of Y ECG Table 14.3.44 12-Lead Electrocardiogram Data by Day and Timepoint (Safety Analysis Set in Part B) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Part B

12-Lead Electrocardiogram Data by Day and Timepoint (Safety Analysis Set in Part B) Table 14.3.44

| Parameter (Unit) | | | | | |
|---|---|---|---|---|---|
| Day | RPL554 | RPL554 | RPL554 | | |
| Time Point | 300µg | 1000μ9 | 3000µg | Placebo | Overall |
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| ECG Parameter #1 (unit) | | | | | |
| Baseline | | | | | |
| п | ×× | ×× | × | ×× | ×× |
| Mean | ×.×. | ×.×. | ×. ×. | ××.× | ×.×. |
| SD | ××.×× | ××.×× | ××.×× | xx.xx | ××.×× |
| Median | ×.×. | x.xx | ×. ×. | x.x. | ×.×. |
| Min, Max | x.x, xx.x | x.x, xx.x | x.x, xx.x | x.x, xx.x | x.x, xx.x |
| Day 7 | | | | | |
| Pre-dose | | | | | |
| Observed | | | | | |
| n | ×× | ×× | ×× | ×× | |
| Mean | ×.×. | ×.×× | ×. ×. | ×.× | |
| SD | ××.×× | xx.xx | xx.xx | xx.xx | |
| Median | ×.× | ×. ×× | ×. ×. | ×.× | |
| Min, Max | x.x, xx.x | x.x, xx.x | xxx, xxxx | xx.x, xx.x | |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Change from Baseline

Author: Jennifer Allsopp


Verona Pharma plc

Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

12-Lead Electrocardiogram Data by Day and Timepoint

(Safety Analysis Set in Part B)

| Parameter (Unit) | | | | | |
|---|---|---|---|---|---|
| Day | RPL554 | RPL554 | RPL554 | | |
| Time Point | 300µg | 1000μg | 3000µg | Placebo | Overall |
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| Mean | x. x. | ×.×× | ×. ×. | ×.×. | |
| SD | xx.xx | xx.xx | xx.xx | xx.xx | |
| Median | x.xx | ×.×× | ×. ×× | x.xx | |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xxx, xxxx | |

ECG Parameter #2 (unit)

SD: Standard deviation.

n = Number of patients with baseline value and a post-baseline value at the time point. N = Number of patients in the analysis set.

Change from baseline: (Pre-dose assessment - baseline assessment).

Baseline: Defined as the pre-dose assessment for each treatment period.

Overall n = Number of patients with a Baseline value at treatment period 1, Day 1.

Source: Listing 16.2.9.12

Programming Notes

ECG quantitative assessments include: QToF Interval (msec), QRS Interval (msec), PR Interval (msec), RR (msec), Heart rate (bpm). Present in alphabetical order. Display for Pre-dose on Day 7.

Output ID: EG001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Part B Page X of Y Table 14.3.45 12-Lead Electrocardiogram - Shifts from Baseline by Day and Timepoint (Safety Analysis Set in Part B) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

| | | | | Category at Timepoint | Timepoint | |
|---|---|---|---|---|---|---|
| Day | | | | | | |
| Time Point | | Baseline | Normal | Abnormal NCS | Abnormal CS | Total |
| Treatment | N | Category | n (%) | n (%) | n (%) | n (%) |
| Day 7 | | | | | | |
| Pre-dose | | | | | | |
| RPL554 300µg | XXX | Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | (x.xx) xx |
| | | Abnormal NCS | xx (xx.x) | xx (xx.x) | (xx.x) | (xx.x) |
| | | Abnormal CS | xx (xx.x) | xx (xx.x) | (xx.x) | (xx.x) |
| | | Total | (x.xx) xx | (xxx) xx | (x.xx) xx | (x.xx) xx |
| RPL554 1000µg | xxx | ï | ŧ | : | : | ; |

NCS = Not clinically significant; CS = Clinically significant.

N = Number of patients with a baseline value and a post-baseline value at the time point. Percentages are based on N. Baseline: Defined as the pre-dose assessment for each treatment period.

Source: Listing 16.2.9.11

Programming Notes

ECG quantitative assessment is Interpretation of results. Display for Pre-dose on Day  $7.\,$ 

Output ID: EG002

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Date: 22JAN2021

Author: Jennifer Allsopp

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Page X of Y Part B Vital Signs Table 14.3.46 Vital Sign Data - Change from Baseline to Post-dose by Day and Timepoint (Safety Analysis Set in Part B) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Table 14.3.46
Vital Sign Data - Change from Baseline to Post-dose by Day and Timepoint (Safety Analysis Set in Part B)

| Time Point Statistics Statistics N=XX N=XX N=XX N=XX N=XX N=XX N=XX N=X | N=XX N=XX XX XX XX | RPL554 3000µg<br>N=XX | | |
|---|---|---|---|---|
| XX | XX | N=XX | Placebo | Overall |
| ×× | × | | N=XX | N=XX |
| XX XX XX | × × × | | | |
| xx | × | | | |
| XXXX<br>XX XX | ×.×× | ×× | ×× | × |
| *** | | × × | ×.× | ×. ×. |
| | ××·×× | xx.xx | xx · xx | ××.×× |
| Median xx.x | ×.×× | × : × | ×.× | ××.× |
| Min, Max xx.x, xx.x xx.x | x.x, xx.x | xx.x, xx.x | x.x, xx.x | xx.x, xx.x |
| 1-hour post-dose<br>Observed | | | | |
| n [a] xx | ×× | ×× | ×× | |
| Mean xx.x > | ×.×. | ×.× | ×.× | |
| x xx.xx x | ××.×× | ××.×× | xx.xx | |
| Median xx.x > | ×.×. | ×.× | ×.× | |
| Min, Max xx.x, xx.x xx. | x.x, xx.x | x.x, xx.x | xx.x, xx.x | |
| Change from Baseline | | | | |

CONFIDENTIAL Verona Pharma plc

Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Vital Sign Data - Change from Baseline to Post-dose by Day and Timepoint Table 14.3.46

(Safety Analysis Set in Part B)

| Parameter (Unit) | | | | | |
|---|---|---|---|---|---|
| Day | | | | | |
| Time Point | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo | Overall |
| Statistics | N=XX | N=XX | N=XX | N=XX | N=XX |
| Mean | ×.×× | ×.× | ×××× | ×.×× | |

2-hour post-dose

Min, Max Median

SD

SD: Standard deviation.

[a] n = Number of patients who have an assessment available at the relevant post-dose assessment timepoint (Observed).

n = Number of patients who have an assessment available at Baseline and the relevant post-dose assessment timepoint (Baseline).

n = Number of patients in the analysis set.

Change from baseline: (Fre-dose assessment for each parameter.

Baseline: Defined as the pre-dose assessment for each parameter.

Baseline: Defined as the practices in the first treatment period in the Safety Analysis Set. Overall n = Number of Baseline values with an assessment available at Baseline and at least one post-dose assessment for treatment period 1, Day 1.

xxx, xx.x

xx.x, xx.x

xxx, xxxx

xxx, xxxx

xx.xx xx.x

> xx.xx ×××

 $\overset{\times}{\times}\overset{\times}{\cdot}$ ××.×

×××

××.×

××.× xx.xx ×××

Source: Listing 16.2.9.13

Programming Notes

Vital signs assessments include: Systolic blood pressure, diastolic blood pressure and pulse rate. Present in alphabetical order. Display for the following timepoints: Day 1 and Day 7: Pre-dose, 1, 2, 4, 8 and 12 hours (all  $\pm$  10 minutes).

Output ID: VS001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Table 14.3.47 Vital Sign Data - Number and Percentage of Markedly Abnormal Values (Safety Analysis Set in Part B) Verona Pharma

Part B Page X of Y

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Vital Sign Data - Number and Percent of Markedly Abnormal Values Table 14.3.47

(Safety Analysis Set in Part B)

| | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo |
|---|---|---|---|---|
| Vital Sign Parameter | N=XX | N=XX | N=XX | N=XX |
| Systolic Blood Pressure (mmHg), n (%) | | | | |
| n [a] | XX | ×× | × | × |
| Value <= 90 | (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) |
| A decrease from baseline of $>=40$ | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Value >= 180 | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| An increase from baseline of $>=40$ | (xx.x) | (x.x.x) | xx (xx.x) | xx (xx.x) |
| Diastolic Blood Pressure (mmHg), n (%) | | | | |
| n [a] | XX | ×× | × | × |
| Value <= 50 | (xxx) xx | (x.x.x) | xx (xx.x) | (x.x) xx |
| A decrease from baseline of $>=20$ | (xxx) xx | (x.x.x) | xx (xx.x) | (x.x) xx |
| Value >= 110 | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| An increase from baseline of $>=20$ | (xxx) xx | (x.xx) xx | xx (xx.x) | xx (xx.x) |
| Pulse Rate (bpm), n (%) | | | | |
| n [a] | XX | XX | ×× | × |
| Value <= 50 | (xxx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| A decrease from baseline of >=30 | (xx.x) | (xx.x) | xx (xx.x) | xx (xx.x) |
| Value >= 110 | (xxx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| An increase from baseline of >=30 | xx (xx.x) | xx (xx.x) | (xxx) xx | xx (xx.x) |

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA84488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0
- Part B

Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Vital Sign Data - Number and Percent of Markedly Abnormal Values

Table 14.3.47

(Safety Analysis Set in Part B)

| Placebo | N=XX |
|---------------|-------------------|
| RPL554 3000µg | N=XX |
| RPL554 1000µg | N=XX |
| RPL554 300µg | N=XX |
| | al Sign Parameter |
| | Vital |

bpm: beats per minute. mmHg: millimeters mercury.
[a] n = Number of patients with a baseline value and a post-baseline value.
Baseline and post-baseline value would be needed for criteria relating to an increase/decrease from baseline.
N = Number of patients in the analysis set. % = Percentages are based on n.

Source: Listing 16.2.9.14

Output ID: VS002

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp


Verona Pharma plc


Author: Jennifer Allsopp

#### Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

```
Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B
                                                                                                                                                                                                                                                                                                                                                                                                                                                          Replace footnotes with:

ANCOVA: Analysis of covariance. CI: Confidence interval. LSMean: Least square mean. LSMean Diff: Least squares mean difference. SD: Standard deviation.

Ancova: Analysis of covariance. CI: Confidence interval. LSMean: Least square mean difference. SD: Standard deviation.

As a number of patients in the analysis set.

Baseline: Pre-dose pulse rate on Day 1 of each treatment period.

Change from Baseline: Post-dose assessment - Pre-dose.

[a] Number of patients with validy values at baseline and timepoint.

[b] ANCOVA model is used to model the change from baseline in pulse rate using baseline assessment as a continuous fixed effect, actual treatment and treatment period as categorical fixed effects.

[c] Number of patients with at least one on treatment value who contributed to the model estimation.

* Indicates a significant p-value (<0.05).
Table 14.3.48 Change from Baseline Pulse Rate to Peak Pulse Rate (over 4 hours) (Safety Analysis Set in Part B)
                                                                                                                                                                               VS005: This output uses shell EFF004 [Table 14.2.6]
                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                                         Source: Listing 16.2.9.15
                                                                                                                                                                                                                                                                                                                                                                                               Programming Notes
```

CONFIDENTIAL Verona Pharma plc

#### Clinical Study Report RPL554-MD-201 Version 1.0; 17 May 2021

Physical Examination Table 14.3.49 Physical Examination Data by Treatment Period and Timepoint (Se

Table 14.3.49 Physical Examination Data by Treatment Period and Timepoint (Safety Analysis Set in Part B) Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.49

Physical Examination Data by Treatment Period and Timepoint

(Safetv Analysis Set in Part B)

| (כמותרא י | (Sarety milarysts Set III Fait B) | ( P) | | |
|---|---|---|---|---|
| Physical Examination: Brief | | | | |
| Assessment | | | | |
| Treatment Period | | | | |
| Time Point | RPL554 300µg | RPL554 1000µg | RPL554 3000µg | Placebo |
| Category | N=XX | XX=N | XX=N | X=N |

xx (xx.x) (xx.x)xx (xx.x) xx (xx.x) (xx.x) xx (xx.x) xx (xx.x) (xxx) xx xx (xx.x) Treatment Period X - Day Y Physical Examination Test #1 Treatment Period X - Day Y Physical Examination Test #2 Abnormal NCS Abnormal NCS Abnormal CS Abnormal CS Pre-dose Normal Pre-dose Normal

CS = Clinically significant. NCS = Not clinically significant. EOS: End of Study.

n = Number of patients who have an assessment available at the relevant timepoint. N = Number of patients in the analysis set. % = Percentage of patients calculated relative to the total number of patients in the analysis set.

Per-chose: Defined as the assessment taken immediately prior to study medication.

End of Study: Defined as the last available assessment assigned to study.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Version: 2.0 Date: 22JAN2021 CONFIDENTIAL Verona Pharma plc

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

Table 14.3.49

Physical Examination Data by Treatment Period and Timepoint

(Safety Analysis Set in Part B)

Physical Examination: Brief

Assessment

Placebo N=XX RPL554 3000µg N=XXRPL554 1000µg N=XX RPL554 300µg N=XX Treatment Period Time Point Category

Source: Listing 16.2.9.16 and 16.2.9.17

Programming Notes

Full/Brief Physical Examination assessments include: For Full: Abdomen [liver and spleen], Cardiovascular system, Extremities, Lymph nodes, Neurological system, Nose, Throat, Respiratory system, Skin, Thyroid gland. For Brief: Abdomen (liver and spleen), Cardiovascular system, Respiratory system, Skin. Present in alphabetical order.

For Full, display for treatment period/timepoints: EOS. For Brief, display for treatment period/timepoints: Treatment period l to 4 - Day l/7 - pre-dose.

Output ID: PE001

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Table 14.3.50 Physical Examinations - Shifts from Baseline by Treatment Period and Timepoint (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Table 14.3.50

Physical Examinations - Shifts from Baseline by Treatment Period and Timepoint

(Safety Analysis Set in Part B)

| Physical Examination: Brief | | | | | | |
|---|---|---|---|---|---|---|
| Assessment | | | | Category a | Category at Timepoint | |
| Treatment Period | | | | | | |
| Time Point | | Baseline | Normal | Abnormal NCS | Abnormal CS | Total |
| Treatment | Z | Category | n (%) | n (%) | n (%) | n (%) |

Physical Examination Parameter #1

Treatment Period X - Day Y

| | (xx.x) | (xx.x) | (xx.x) | | (xx.x) xx | xx (xx.x) | (xx.x) | |
|---|---|---|---|---|---|---|---|---|
| | × | × | × | | × | × | × | |
| | ×.× | ×.× | (x.xx) xx | ×.× | ×.× | xx (xx.x) | ×.× | ×.× |
| | × | × | × | × | (xx.x) | × | xx (xx.x) | xx (xx.x) |
| | × | × | × | × | × | × | × | × |
| | (x.xx) xx | (x.x.) xx | (x.xx) xx | (×.×) | (x.xx) xx | (x.x) | (x.x.) xx | xx (xx.x) |
| | X | ()<br>X | ×× | C)<br>X | "<br>× | X | ()<br>X | X |
| | ~ | ^ | 7 | ~ | ^ | ^ | ^ | ^ |
| | ×.× | ×.× | (x.xx) xx | (×.× | (x.xx) xx | ×.× | ×.× | ×.× |
| | × | × | × | × | × | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | × | × | × | × | × | × | × | × |
| | | NCS | Ω<br>() | | | CS | Ω<br>() | |
| | l<br>I | mal 1 | mal ( | | 1 | mal 1 | mal ( | |
| | Normal | honor | Abnormal CS | otal | lorma | Abnormal NCS | honor | [ota] |
| | 4 | H | A | г | 4 | H | H | г |
| | × | | | | × | | | |
| | )µg | | | | 6 <b>n</b> 00 | | | |
| 1) | 4 300 | | | | 4 100 | | | |
| rre-dose | RPL554 300µg | | | | RPL554 1000µg | | | |
| FL | - | | | | | | | |

CS = Clinically significant. NCS = Not clinically significant. EOS: End of Study.

n = Number of patients. N = Number of patients with a baseline value and a post-baseline value at the time point. Percentages are based on N.

Baseline: Defined as the assessment taken immediately prior to study medication.

End of Study: Defined as the last available assessment assigned to study.

For full physical examination baseline is defined as the screening assessment. Baseline for brief physical examinations is Day 1 of each treatment period. Baseline for full physical examination is screening collected in Part A which is compared to the EOS visit from Part B.

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp
Protocol: RPL554-MD-201 Verona Pharma

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Physical Examinations - Shifts from Baseline by Treatment Period and Timepoint

Table 14.3.50

(Safety Analysis Set in Part B)

Physical Examination: Brief

| | | Total | n (%) |
|----------------------|------------------|--------------|-----------|
| ategory at Timepoint | | Abnormal CS | n (%) |
| Category a | | Abnormal NCS | (%)<br>U |
| | | Normal | n (%) |
| | | Baseline | Category |
| | | | Z |
| Assessment | Treatment Period | Time Point | Treatment |

Source: Listing 16.2.9.16 and 16.2.9.17

Full/Brief Physical Examination assessments include: For Full: Abdomen [liver and spleen], Cardiovascular system, Extremities, Lymph nodes, Neurological system, Nose, Throat, Respiratory system, Skin, Thyroid gland. For Brief: Abdomen (liver and spleen), Cardiovascular system, Respiratory system, Skin. Present in alphabetical order.

For Full, display for treatment period/timepoints: EOS. For Brief, display for treatment period/timepoints: Treatment period 1 to 4 - Day 1/7 - pre-dose.

Output ID: PE002

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

#### Figures

Part B Page X of Y Figure 14.2.6 Geometric Mean of ratios of Peak FEV, (over 4 hours) to pre-dose FEV, by Treatment (Full Analysis Set in Part B) RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Geometric Mean of ratios of Peak  $\operatorname{FEV}_1$  (over 4 hours) to pre-dose  $\operatorname{FEV}_1$  by Treatment Figure 14.2.6



FEV: Forced expiratory volume in 1 second. Pre-dose FEV: The value of FEV: assessed immediately before first administration on each Day 1.

Bottom and top whiskers: 95% lower confidence limit and 95% upper confidence limit.

Bottom and top whiskers: 95% lower confidence limit and 95% upper confidence limit.

Bar: Geometric means on the ratio to pre-dose. ANCOVA model is used to model the change from pre-dose FEV; using pre-dose FEV; as a continuous fixed effect, planned treatment and treatment period as categorical fixed effects. Source: Listing 16.2.6.6

Programming Notes

Above is an example. Display for all treatment groups in Part B in ascending order (RPL554 300pg, RPL554 1000pg and RPL554 3000pg) and then placebo. For each treatment group present the GeoMean and SEM (standard error of the mean).

Output ID: EFF11

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Figure 14.2.7 Mean Change from pre-dose FEV; to Peak FEV; (over 4 hours) by Treatment (Full Analysis Set in Part B) Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Figure 14.2.7

Mean Change from pre-dose FEV1 to Peak FEV1 (over 4 hours) Treatment

(Full Analysis Set in Part B)



FEV: Forced expiratory volume in 1 second. Pre-dose FEV: The value of FEV: assessed immediately before first administration on each Day 1.

Bottom and top whiskers: 95% lower confidence limit and 95% upper confidence limit. Bar: LS Means change from pre-dose. ANCOVA model is used to model the change from pre-dose FEV1 using pre-dose FEV1 as a continuous fixed effect, planned treatment and treatment period as categorical fixed effects.

Source: Listing 16.2.6.6

Programming Notes

Above is an example. Display for all treatment groups in Part B in ascending order (RPL554 300µg, RPL554 1000µg and RPL554 3000µg) and then placebo. For each treatment group present the LSMean and SEM (standard error of the mean). Update y-axis label to "LS Means change from pre-dose (mL)".

Output ID: EFF12

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Page X of Y Part B Figure 14.2.8 Mean Change from Pre-dose FEV, during spirometry over Time by Treatment and Day (Full Analysis Set in Part B) Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Mean Change from Pre-dose FEV; during Spirometry over Time by Treatment and Day

Figure 14.2.8

(Full Analysis Set in Part B)



Means are calculated on the observed data. Pre-dose: the highest FEV1 result collected immediately pre-dose (within 5 minutes) on day 1 for each treatment period.

Source: Listing 16.2.6.5

Programming Notes

Insert a label below the figure for each of the treatment groups, each with a different colour and symbol. Display for all treatment groups in Part B in ascending order (RPLS54 300µg, RPLS54 1000µg and RPLS54 3000µg) and then placebo. Also adjust x-axis for the Repeat figure for Day 7.

Output ID: EFF09

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Page X of Y Figure 14.2.9 Kaplan-Meier plot of Time to Onset of Action (>10% Increase in FEV;) on Day 1 (Full Analysis Set in Part B) Verona Pharma

Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Figure 14.2.9

Kaplan-Meier plot of Time to Onset of Action (>10% Increase in FEV1) on Day 1

(Full Analysis Set in Part B)



Time to first onset of action (mins): Time of first onset of action (defined as >10% increase in FEV; from pre-first dose) = Time of onset of action (or censoring time) - time of end of inhalation (mins).
P25, Median and P75 time to onset of action: Estimated using Kaplan-Meier statistics.
Censored: Patients not experiencing onset of action are censored at 120 mins or at time of premature discontinuation (if withdrawn before 120 minutes).

Source: Listing 16.2.6.7

Programming Notes

Insert a label below the figure for each of the treatment groups, each with a different colour and symbols.

Output ID: EFF10

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Figure 14.3.5 Mean Change from Pre-dose Pulse Rate to Peak Pulse Rate (over 4 hours) by Treatment (Safety Analysis Set in Part B)

VS003: This output uses shell EFF11 [Figure 14.2.6]

Pre-dose pulse rate: The pulse rate value assessed immediately before administration on each Day 1. Bottom and top whiskers: 95% lower confidence and 95% upper confidence limit. Bar: Results on orginal scale. ANCOVA model is used to model the change from predose pulse rate as a continuous fixed effect, and actual treatment as categorical fixed effects.

Update source footnote to "Source: Listing 16.2.9.15". Replace footnotes in original shell with those listed above Programming Notes

Figure 14.3.6 Mean Change from Pre-dose in Pulse Rate over Time by Treatment and Day (Safety Analysis Set in Part B)

VS004: This output uses shell EFF09 [Figure 14.2.6]

Means are calculated on the observed data. Pre-dose: the pre-dose assessment collected on day 1 for each treatment period.

Update source footnote to "Source: Listing 16.2.9.15". Replace footnotes in original shell with those listed above Programming Notes

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


### Listings

Listing 16.2.1.2 Completed/Discontinued Patients (All Randomized Analysis Set in Part B) Protocol: RPL554-MD-201 Verona Pharma

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

> (All Randomized Analysis Set in Part B) Completed/Discontinued Patients Listing 16.2.1.2

> > Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| Mas treatment unblinded by unblinded by Randomiz- the site? If ation yes, provide atter date date and ID Study day reason TP I DDWMYYYY XXX/DDWMYYY DDWM | | | | | | |
|---|---|---|---|---|---|---|
| treatment unblinded by unblinded by the site? If ation yes, provide date, Study day reason DDMMMYYYY, XXX/DDMMMYYY | | | | | Completed study/ | |
| unblinded by Atheritation yes, provide date/ date and Study day reason DDMMMYYYY/ XXX/DDMMMYYY | | | | | Date of | Reason not |
| Randomiz- the site? If ation yes, provide date/ date and Study day reason DDMMMYYYY XXXX/DDMMMYYY | | | | | completion/ | completed, Other |
| ation yes, provide date/ date and Study day reason DDMMMYYYY/ XXX/DDMMMYYY | | | | | discontinuation/ | (specify)/If AE, |
| date/ date and Study day reason DDMMMYYYY/ XXX/DDMMMYYYY | | | | Treatment | Study Day/Primary | specification/If |
| Study day reason DDMMMYYYY/ XXX/DDMMMYYY | | | | period | reason if not | death, date of |
| DDMMMYYYY / XXX/DDMMMYYY | TP 1 TP 2 TP 3 TP 4 | TP 3 | TP 4 | discontinued | completed | death |
| | DDMMMXYYY/ DDMMMYYYY/ DDMMMYYYY/ | /XXXXMMMQQ | /XXXXWMDQ | ******* | No/DDMMMYYYY/xx/ | XXXXXXX/XXXXXXXX |
| | XX XX | ×× | ×× | WWW.WWW.WW | XXXXXX | /DDMMMYYYY |

TP: Treatment Period. Study day: Relative to first dose of study medication (i.e., Treatment period 1, Day 1).

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 1000 mcg/RPL554 300 mcg/RPL554 1000 mcg/RPL554 1000 mcg/RPL554 300 mcg/

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L001

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.2.2 Protocol Deviations (All Randomized Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Protocol Deviations Listing 16.2.2.2

(All Randomized Analysis Set in Part B)

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| | [ |
|---------------------------------|----------------|
| Severity | XXXXXXXXXX |
| Type of deviation | XXXXXXXXXX |
| Protocol<br>deviation | XXXXXXXXXX |
| Deviation date/<br>Relative Day | DDMMYYYY/xx |
| Treatment<br>group | XXXXXXXX |
| Age/Sex/Race | XXXXXXX/X/XX |
| Patient ID | XXXXXXXXXXXXXX |

Seq

As: Native Asian. Bl: Black or African American. CTMS: Clinical trial management system. eCRF: Electronic case report form. F: Female. Is: American Indian or Alaskan. M: Male. Ot: Other. Pi Native Hawaiian or Pacific islanders. Un: Unknown. W: White. Protocol deviations: Defined as deviation types reported in the CTMS log:

Age (years): As reported in the eCRF.

Female and addition per treatment period (i.e., Treatment period X, Day I).

Seq 1 = RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and then the deviation date.

Output ID: L003

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.3.2 Patient Included in Analysis Sets (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.3.2

(All Randomized Analysis Set in Part B) Patient Included in Analysis Sets

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | | | Analysis Sets | Sets | |
|---|---|---|---|---|---|
| Patient ID | Randomized | Safety | Full | Completers | Pharmacokinetic |
| | Yes | Yes | Yes | Yes | Yes |
| XXXXX | Yes | Yes | Yes | No | Yes |

... Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/Placebo/RPL554 300 mcg/ RPL554 300 mcg/RPL554 300

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L002

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Listing 16.2.4.7 Demographic Characteristics (All Randomized Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

Listing 16.2.4.7

Demographic Characteristics

(All Randomized Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| atient ID | Country | Age/Sex/Race | Ethnicity | Weight<br>(kg) | Height (cm) | BMI $(kg/m^2)$ | Re-<br>screened<br>patient | Childbearing potential |
|---|---|---|---|---|---|---|---|---|
| XXXXXXX | UK | 62/F/W | XXXXXXXX | XX | XXX | XX.X | × | × |
| XXXXX | UK | M/W/L9 | ×××××××× | × | XXX | ×.× | × | NA |

As: Native Asian. B1: Black or African American. BMI: Body mass index. eCRF: Electronic case report form. F: Female. Ia: American Indian or Alaska. M: Male. NA: Not applicable. Ot: Other. Pi: Native Hawaiian or Pacific Islanders. Un: Unknown. W: White.

Age (years): As calculated relative to informed consent date.

BMI (kg/m²) = Weight (kg) / Height (m)².

All measurements listed above are measured at Screening on the Demography eCRF.

Seq 1 = RPL554 300 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 3000 mcg. RPL554 3000 mcg. Seq
3 = RPL554 3000 mcg/RPL554 1000 mcg/RPL5

Programming Notes:

Order by treatment group (as per shell) and within group by patient ID.

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.4.8 Screening Disease Characteristics (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.4.8

(All Randomized Analysis Set in Part B) Screening Disease Characteristics

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| | | Bronchod: lator | 11 12+Or | | Brong | ronchod: lator | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | FEV1 (L) | (L) | | É | FVC (L) | | | | Rever | Reversibility |
| | | | | ı | | | | Assessment | | | |
| | | | | | | | Post- | performed | | | |
| | | | | | | | bronchodi- | with four | Met | | |
| Patient | Age/Sex | | | Predicted | | | lator | poffs of | reversibility | | |
| ID | /Race | Pre | Post | FEV1 (%) Pre | Pre | Post | FEV1/FVC | albuterol | test criteria? | o)P | mL |
| 2222 | XX/X/XX | ^^ | >> | | ^^ | ^^ | AA | ^^ | ^^ | > | 222 |
| 7777 | > | \{ | VV | | <b>V</b> V | VV | VV | VV | VV | | 777 |

As: Native Asian. Bl: Black or African American. F: Female. FEV; Forced expired volume in 1 second. FVC: Forced vital capacity. Ia. American Indian or Alaska. M: Male. Ot: Other. Pi: Native Hawaiian or Pacific islanders. Un: Unknown. W: White.

Pre-, post-bornchodilator and reversibility values are the results of the screening reversibility test.

Pag 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 2 = RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 4 = Placebo/RPL554 3000 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L005

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.4.9 COPD and Smoking History (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

COPD and Smoking History Listing 16.2.4.9

(All Randomized Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

Smoking exposure (pack-years) × Number of years smoking × Number of packs per day × Bronchitis/ Emphysema Yes/Yes Date of most recent exacerbation/ Study day DDMMMYYYY/xx Duration of COPD (years) (time since diagnosis) × Date COPD first diagnosed DDMMMYYYY

> Patient ID XXXXXXX

Smoking History

COPD: Chronic Obstructive Pulmonary Disease. Smoking exposure (pack-years) = Number of packs per day \* Number of years smoking, for patients with a smoking history or a current smoker.

Study day: Relative to first dose of study medication (i.e., Treatment period 1, Day 1).

Duration of COPD (years) (time since diagnosis) = (Randomization date - date c COPD first diagnosed)/365.25.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/ RPL554 3000 mcg. Seq 3 = RPL554 3000 mcg/RPL554 1000 mcg/RPL554 3000 mcg. Seq 3 = RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 4 = Placebo/RPL554 3000 mcg/RPL554 1000 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L006

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc

Listing 16.2.4.10 Medical History (All Randomized Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Page X of Y Part B

Listing 16.2.4.10

Medical History

(All Randomized Analysis Set in Part B)

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| End date/ | Study day | **** / ANAMAMATA | DUMMITTI / XX |
|---|---|---|---|
| Start date/ | Study day | / AAAAAAAAA | DDMMINITITY XX |
| | SOC/PT | /XXXXXXXXXXX | ^^^^^^^^ |
| Medical history | diagnosis | 222222222222222222222222222222222222222 | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ |
| | Patient ID | ********** | VVVVVVVV |

MedDRA: Medical Dictionary for Regulatory Activities. PT: Preferred Term. SOC: System Organ Class.

Medical history: Coded using MedDRA (Version 21.0).

Study day: Relative to first dose of study medication (i.e., Treatment period 1, Day 1).

Study day: Relative to First dose of study medication (i.e., Treatment period 1, Day 1).

Study and PREL554 300 mcg/Rel554 3000 mcg/Rel554 3000 mcg/Rel554 1000 mcg/Rel554 1000 mcg/Rel554 3000 mcg. Seq 2 = Rel554 3000 mcg/Rel554 300 mcg. Req.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L007

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Listing 16.2.4.11 Surgical Procedure History (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Surgical Procedure History Listing 16.2.4.11

(All Randomized Analysis Set in Part B)

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| End date of<br>procedure/<br>Study day | DDMMYYYY/xx |
|----------------------------------------|-----------------|
| Start date of procedure/<br>Study day | DDMMMYYYY/xx |
| Purpose of procedure | XXXXXXXXXXXX |
| Reported name of procedure | XXXXXXXXXXXXXXX |
| Patient ID | XXXXXXXX |

Surgical procedure history: Coded using MedDRA (Version 21.0).
Study day: Relative to first dose of study medication (i.e., Treatment period 1, Day 1).
Seq 1 = RFL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 1000 mcg

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L008

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc

Listing 16.2.4.12 Prior and Concomitant Medications (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.4.12

Prior and Concomitant Medications

(All Randomized Analysis Set in Part B)

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| | Frequency/ | Route | /xxxxxxxx | XXXXXXXX |
|---|---|---|---|---|
| | Dose | (Unit) | (XX (XX) | |
| | | Indication | XXXXXX | |
| | ATC Level 1/ | Preferred term | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXX |
| | P?[a]/ | C? [b] | ت<br>ت | |
| Start date (Study day)/ | End date | (Study day) | /(XX) / | DDMMMYYYY (XX) |
| | Treatment | period | XXXXXXXXX | |
| | Treatment | dronb | XXXXXXXXX | |
| | | Patient ID | XXXX/XXXX | |

ATC: Anatomical Therapeutic Chemical. C: Concomitant. P: Prior.

[a] Medication taken between Part A and Part B of the study or prior to the start of study medication.

[b] Medication taken between start and stop of study medication.

[c] Medication taken between start and stop of study medication (i.e., Treatment period 1, Day 1).

Study day Day relative to day of the first dose of study medication (i.e., Treatment period 1, Day 1).

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg, RPL554 300 mcg. Seq 3 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg.

# Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID
'Prior' medications are medications which started and stopped in the time between Part A and Part B (prior to the study medication at TPI, Day 1) and have Started prior to start of study medication? = "Yes" on the Concomitant medications eCRF page.
'Concomitant' medications are medications which:
O'Had an onset date on or after the study medication.

Output ID: L009

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.4.13 Prior COPD Medications (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.4.13

Prior COPD Medications

(All Randomized Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

Frequency/ Route XXXXXXXX/ XXXXXXXX End date (Study day) DDMMMYYYY (XX)/ DDMMMYYYY (XX) Start date (Study day)/ Patient ID

ATC: Anatomical Therapeutic Chemical.
Study day: Day relative to day of the first dose of study medication (i.e., Treatment period 1, Day 1).
Seq 1 = RFL554 3000 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID Prior was a medications which started and stopped in the time between Fart A and Part B (prior to the study medication at TPI, may 1) and have Started prior to start of study medication? = "Ves" on the Concomitant medications eCRF page.

COPD medications are when indication is "Other" and other reason for medication is "COPD".

Output ID: L009

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp


Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

#### Version 1.0; 17 May 2021 Clinical Study Report RPL554-MD-201

Listing 16.2.5.2 Drug Exposure and Accountability (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

(All Randomized Analysis Set in Part B) Drug Exposure and Accountability Listing 16.2.5.2

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | | Weight of | (d) pesn IDWd | XX | ×× |
|---|---|---|---|---|---|
| | Weight of | pMDI returned | (b) | XX | X |
| | Weight of | pMDI dispensed | (6) | XX | ×× |
| | Start time/ | End time | of inhalations | нн:мм/нн:мм | нн:мм/нн:мм |
| Start date and | of study | medication / | Relative day | DDMMMYYYY/xx | DDMMMYYYY/xx |
| | Treatment | period/ | Timepoint | /xxxxxxxxxx | /XXXXXXXXXX |
| | | Treatment | dnozb | | XXXXXXXX |
| | | | Patient ID | XXXXXXXXX | XXXXXXXX |

Relative day: Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/Placebo/RPL554 300 mcg/RPL554 3000 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L010 [Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

CONFIDENTIAL Verona Pharma plc

Listing 16.2.6.5 Spirometry: FEV1 Results (Full Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Part B Page X of Y

RPL554 pressurised Metered Dose Inhaler

Spirometry: FEV1 Results Listing 16.2.6.5

(Full Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | | | Predicted | FEV1 (%) | XX.X | |
|---|---|---|---|---|---|---|
| | | FEV1 | measurement | (T) | X.XXX [a] | |
| Refrained from | smoking/Capable of | withdrawing from long | acting | bronchodilators | XXXXXX/ | |
| | Date and | time/ | Relative | day | DDMMYYY<br>HH:MM/xx | |
| | | Treatment | period/ | Timepoint | /xxxxxx | XXXXXX |
| | | | Treatment | group | XXXXX | |
| | | | Patient | ID | XXXXX | |

FEV: Forced expiratory volume in 1 second. PPT: Pulmonary function test.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/PPL554 1000 mcg/PPL554 1000 mcg/RPL554 300

Programming Notes

The assessment timepoints can be Pre PFT -60 min, Immediately Pre-dose, Post PFT Smin, 15min, 10, 1.5h, 2h, 4h, 8h, 12h and EOS. Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L014

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.6.6 Spirometry: FEV1 Derived Measurements (Full Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Spirometry: FEV1 Derived Measurements (Full Analysis Set in Part B) Listing 16.2.6.6

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| Average FEV <sub>1</sub><br>(AUC) 12h (CFB) | X.XXX (X.XXX) |
|---------------------------------------------|----------------|
| Average FEV1<br>(AUC) 4h (CFB) | X.XXX (X.XXX) |
| Morning<br>trough FEV1 (CFB) | X.XXX (X.XXX) |
| Peak FEV $_1$ 4h (CFB) | X.XXX (X.XXX) |
| Date/<br>Relative day | DDMMYYY/<br>xx |
| Treatment<br>period/<br>Timepoint | /xxxxxxx |
| Treatment<br>group | XXXXXX |
| Patient<br>ID | XXXXX |

AUC: Area under the curve. CFB: Change from Baseline. FEV:: Forced expiratory volume in 1 second.

Peak FEV:: Maximum post-dose value among the values collected up to timepoint of interest hours.

Morning trough FEV:: average of the FEV; pre dose assessments (-60 minutes and -5 minutes) on Day 7.

Average FEV: AUC: AUC of the FEV: values (maximum value of the three assessments at each timepoint) divided by the length of the time

(in hours) interval of interest (per visit).

Relative day, Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 300 mcg/RPL554 3000

Programming Notes

The assessment timepoints can be Pre PFT, Post PFT, Pre PFT -60 min, Immediately Pre-dose, Post PFT 5min, 15min, 10, 11, 1.5h, 2h, 4h, 8h, 11h, 12h and EOS. Order by treatment sequence (as per shell) and within sequence by patient ID and treatment period.

Output ID: L015

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.6.7 Spirometry: FEV; Time to First Occurrence of Onset of Action (Full Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

Part B

Page X of Y

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.6.7

Spirometry: FEV1 Time to First Occurrence of Onset of Action

(Full Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | Time to first | set | of action (mins) (Yes/No)* | XX | XX |
|---|---|---|---|---|---|
| Time of onset | of | | (HH:MM) | HH:MM | HH: MM |
| | Time of | pre-dose | (HH:MM) | HH: MM | HH: MM |
| | | Date/ | Study day | XXXX-MM-DD/XX | YYYY-MM-DD/XX |
| | | Treatment | group | XXXXXX | XXXXXX |
| +<br>4<br>6 | דמרד תור | T T | | XXXXXX | XXXXXX |

Time to first occurrence of onset of action (mins): Time of onset of action (defined as >10% increase in FEV, from pre-first dose) = Time of onset of action (or censoring time) - time of end of inhalation (mins).

\* Patients not experiencing onset of action are censored at 120 mins or at time of premature discontinuation (if withdrawn before 120 minutes).

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg. Seq 3 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg.

Output ID: L032

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Listing 16.2.6.8 Dyspnea Scale Score (Full Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Dyspnea Scale Score Listing 16.2.6.8

(Full Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| Patient<br>ID | Treatment<br>group | Treatment period/<br>Timepoint | Assessment performed/<br>Date and time/<br>Relative day | Dyspnea scale score |
|---|---|---|---|---|
| XXXXXX | XXXXXX | XXXXXX/<br>XXXXXXX | XXX/<br>YYYY-MM-DD/HH:MM/<br>XX | XX |

Dyspnea scale score: Likert scale assessment ranging from 0 to 10, where 10 represents the "worst shortness of breath that you can imagine" and 0 represents "no shortness of breath".

Relative day: Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg RPL554 300 mcg. Se 2 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L033

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Listing 16.2.6.9 Rescue Medications (All Randomized Analysis Set in Part B) Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.6.9

(All Randomized Analysis Set in Part B) Rescue Medications

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | | Number of puffs | × |
|---------|-----------------|-------------------------|-------------|
| | | Rescue Medication Taken | Yes/No |
| Date of | administration/ | Relative day | DDMMMYYYY/x |
| | Treatment | period | XXXXXXX |
| | Treatment | group | XXXXXX |
| | Patient | ID | XXXXXX |

Rescue medications = Short acting bronchodilators used to relieve i.e. rescue symptoms immediately.

Relative day. The first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L034

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Page X of Y Listing 16.2.6.10 Rescue Medications Canister Dispensed, Weight and Collection Information (All Randomized Analysis Set in Part B) Verona Pharma

Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.6.10

Rescue Medications Canister Dispensed, Weight and Collection Information

(All Randomized Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | | | Inh | Inhaler Dispensed | ped | пI | Inhaler Weighed | id | Inh | Inhaler Collected | ed |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Inhaler<br>dispensed? | | | Inhaler<br>weighed? | | | Inhaler<br>collected? | | |
| Patient I | Inhaler | Treatment | If no, | | | If no, | | | If no, | | |
| ID | number | Period | specify | Date/time Weight(g) | Weight(g) | specify | Date/time Weight(g) sp | Weight (g) | ecify. | Date/time Weight(g) | Weight (g) |
| * 252525252525 | *** | 262626262626263 | MANAGEM / M | DDMMYYYY | 75 AA | 22222222 / 25 | DDMMYYYY | 74 7474 | /x/x/x/x/x/ / | DDMMXYYY | W W |
| 7 77777 | VV | 77777777 | V / VVVVV | HH · MM | 77.7 | V / VVVVV | HH · MM | ۷۷.۷۷ | V / VVVVV | HH · MM | ۸۸.۸ |

Rescue medications = Short acting bronchodilators used to relieve i.e. rescue symptoms immediately.
Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/PPlacebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL554 3000 mcg/RPL554 300

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L038

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Listing 16.2.7.6 List of All Adverse Events (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

(Safety Analysis Set in Part B) Listing of All Adverse Events Listing 16.2.7.6

Treatment groups: <RPL554 300µg/RPL554 1000µg/RPL554 3000µg/Placebo>

| | Study day | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | of last | | | Start/End | | | | | | | | | |
| | dose of | | | date | | | | | | | | | |
| | study | | | or ongoing | | | | | | Chronic- | | Disconti- | |
| Patient | medicatio | SOC/PT/Reported | Treatment | (Study day) | Sev | Rel | Act | Ser | Out | ity | Treatment | nued from | Blind |
| ID | n [a] | term [b] | period | [c] | [q] | [e] | [ £ ] | [d] | [h] | [i] | given | study | broken |
| >>>> | >> | /xxxxx/xxxxxx | ^^^^ | VVVVV | TM | > | OIV. | N | Rsl | ^/ ^/ ^^ | 0 | 0 | 0 |
| 00000 | 44 | ^^^^ | 00000 | DOMEST LILL | TIT | 4 | ) 1 | 2 | 4.7 | 4/4/44 | D<br>U | n<br>U | C U |

SOC: System organ class. PT: Preferred Term.

AEs which started within a treatment period are assigned to that treatment period.

[a] Day of last does groupdy medication relative to day of the first dose of study medication (i.e., Treatment period 1, Day 1).

[b] An asterisk "\*" indicates a non-treatment-emergent adverse event.

[c] Study day: Day relative to day of the first dose of study medication (i.e., Treatment period 1, Day 1).

[d] Severity: MI-Mild, MO-Moderate, SE-Severe.

[e] Related to study davig.

[f] Action taken with respect to study drug: NC = Dose Not Changed, DD = Drug Discontinued, DI = Drug Interrupted, O = Other, NA = Not Applicable.

[f] Serious AE.

[g] Serious AE.

[h] Outcome: Fatal = Fatal, NRslv = Not recovered/not resolved, Rslv = Resolved/Recovered, RslvG = Recovering/Resolving, RslvS = Recovering Cocasion, I = Intermittent, P = Persistent.

Socs and PT are coded using the MedDRA (Version 21.0).

Programming Notes

Order by treatment group (as per shell) and within sequence by patient ID, adverse event start date and adverse event end date (in that

Output ID: L016

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.7.7 Treatment-emergent Adverse Events Leading to Study Discontinutation (Safety Analysis Set in Part B)

L017: This output uses shell L016 [Listing 16.2.7.6]

Listing 16.2.7.8 Treatment-emergent Adverse Events Leading to Death (Safety Analysis Set in Part B)

L018: This output uses shell L016 [Listing 16.2.7.6]

Listing 16.2.7.9 Serious Treatment-emergent Adverse Events (Safety Analysis Set in Part B)

L019: This output uses shell L016 [Listing 16.2.7.6]

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Listing 16.2.7.10 Serious Treatment-emergent Adverse Events - Details (Safety Analysis Set in Part B) Verona Pharma RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201

Part B Page X of Y

> Serious Treatment-emergent Adverse Events - Details (Safety Analysis Set in Part B) Listing 16.2.7.10

Treatment groups: <RPL554 300µg/RPL554 1000µg/RPL554 3000µg/Placebo>

| Patient ID | SOC/PT/<br>Reported Term | SAE details | Answer |
|---|---|---|---|
| XXXXXXXXXX | XXXXXX/XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Date Investigator became aware of SAE | DDMMMYYYY |
| | | Death | XXXXX |
| | | Life-threatening | XXXXX |
| | | Initial or prolonged hospitalization | XXXXX |
| | | Date of admission (DD MMM YYYY) | DDMMMYYYY |
| | | Date of discharge (DD MMM YYYY) | DDMMMYYYY |
| | | Persistent or significant disability/incapacity | XXXXX |
| | | Congenital anomaly/birth defect | XXXXX |
| | | Occurred with overdose | XXXXX |
| | | Other medically important event | XXXXX |
| | | Was the SAE caused by other medication? (e.g. Concomitant medication, background medication, rescue medication) | XXXXX |
| | | If Yes, Please Specify | XXXXX |
| | | Was the SAE caused by study procedure(s)? | XXXXX |
| | | If Yes, Please Specify | XXXXX |
| | | Describe treatment for event including medications (1) | XXXXX |
| | | Describe treatment for event including medications (2) | XXXXX |
| | | Describe treatment for event including medications (3) | XXXXX |
| | | List all diagnostic tests that were done to confirm event (1) | XXXXX |
| | | List all diagnostic tests that were done to confirm event (2) | XXXXX |
| | | List all diagnostic tests that were done to confirm event (3) | XXXXX |
| | | Description of SAE/narrative | XXXXX |
| Document: \\ieedc-vnasc<br>- Part B | :01\biosdata\Verona_Pharma\R | Document: \\ieedc-vnasc01\biosdata\Verona_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B | TLF Shells v2.0 |
| | Ω | | Version: 2.0<br>Date: 22JAN2021 |
| | L <sub>4</sub> | | |

RPL554 pressurised Metered Dose Inhaler Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part B

Listing 16.2.7.10

Serious Treatment-emergent Adverse Events - Details

(Safety Analysis Set in Part B)

Treatment groups: <RPL554 300µg/RPL554 1000µg/RPL554 3000µg/Placebo>

| SOC/PT/<br>Reported Term |
|--------------------------|

PT: Preferred Term. SAE: Serious Adverse Event. SOC: System Organ Class. SOCs and PTs are coded using the MedDRA (version 21.0).

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.

Output ID: L020

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Version: 2.0 Date: 22JAN2021 Author: Jennifer Allsopp

Listing 16.2.8.5 Hematology (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.8.5

Hematology

B (Safety Analysis Set in Part

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| Change<br>from<br>Baseline | XX.X |
|---------------------------------------------|------------------------|
| Value<br>(unit)<br>L/H [a] | XX (unit) |
| Date/Time of<br>assessment/<br>Relative day | DDMMMYYYY/HH:MM/<br>** |
| Treatment<br>period/<br>Timepoint | /xxxxxxx/ |
| Treatment<br>group | XXXXXXX |
| Reference<br>Range<br>(Lower-<br>Upper) | XX.X - XX.X |
| Parameter | Hemoglobin |
| Patient ID | XXXXXXXXXXX |

[a] L = Below low normal range. H = Above high normal range.

Baseline: Defined as the pre-dose assessment for each treatment period.

Relative day: Relative to day of the first dose of study medication in each treatment period.

Bed Study: Defined as the last available assessment assigned to study.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 2 = RRL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg. RPL554 300 mcg. RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell), hematology parameter (in alphabetical order), patient ID and treatment period.

Output ID: L021

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Listing 16.2.8.6 Biochemistry (Safety Analysis Set in Part B)

L022: This output uses shell L021 [Listing 16.2.8.5]

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.8.7 Urinalysis (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.8.7

Urinalysis

(Safety Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| Patient<br>ID | Parameter | Treatment<br>group | Treatment<br>period | Date/Time of assessment/<br>Relative day | Result [a] |
|---|---|---|---|---|---|
| XXXXXXXXXX | Ketones | XXXXXX | XXXXXX | DDMMMYYYY/HH:MM/xx | NEGATIVE (N) |
| | Leukocyte Esterase | | | DDWMMYYYY/HH:MM/xx | TRACE (T) |
| | Occult Blood | | | DDMMMYYYY/HH:MM/xx | 1+ (P) |
| | 1 | | | | |

[a] Category assigned and used in the shift table: N = Normal or 'Negative'; T = 'Trace' P = '1+','2+','3+',' or '4+'. The flag appears only for the following parameters: Leucocytte Esterase, Bilitubin, Glucose, Retones, Occult blood, Protein and Urobilinogen. Relative day: Relative to day of the first dose of study medication in each treatment period.

Baseline: Defined as the pre-dose assessment for each treatment period.

End of Study: Defined as the last available assessment assigned to study.

Seq 1 = RPL554 300 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 2 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg. Seq 3 = RPL554 3000 mcg/RPL554 300 mcg. Reg.

Programming Notes

Order by treatment sequence (as per shell), urinalysis parameter (in alphabetical order) and by patient ID and treatment period.

Output ID: L023

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.9.11 Electrocardiogram Local Reading Overall Evaluation (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.11

Electrocardiogram Local Reading Overall Evaluation

(Safety Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

Abnormal Significant/ Specify X/XXXXXX Overall ECG Evaluation Normal Normal Date/Time of assessment/Relative DDMMMYYYY/HH:MM/xx DDMMMYYYY/HH:MM/xx day Treatment Period/Day /Timepoint XXXX/XXXX XXXX/XXXX Treatment XXXXXXXXX XXXXXXXX XXXXXXXXXXX XXXXXXXXXXX Patient

ECG: Electrocardiogram.

Relative day: Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 1000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 1000 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 1000 mcg/RPL554 1000 mcg/RPL554 1000 mcg/RPL554 300 mcg/RPL5

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L024

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc

Listing 16.2.9.12 12-lead ECG (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.12

(Safety Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| CFB | xx.x | х. х | x x | х.х | х.х | XX.X | : |
|---|---|---|---|---|---|---|---|
| Baseline | XX.X | XX.X | XX.X | XX.X | x.xx | x.xx | ŧ |
| Result | x.xx | xx.x | x.xx | xx.x | x.xx | x.xx | i |
| ECG parameter (unit) Result | HR (bpm) | PR interval (msec) | QRS duration (msec) | QT interval (msec) | QTCF | RR interval (msec) | 1 |
| Date/Time of assessment/Relative day | DDMMMYYY/HH:MM/xx | | | | | | DDMMMYYY/HH:MM/xx |
| Treatment<br>Period/Day<br>/Timepoint | XXXXX | | | | | | XXXXX |
| Treatment<br>Group | XXXXX | | | | | | XXXXX |
| Patient ID | XXXXXXXXXXXX | | | | | | |

bpm: beats per minute. CFB: Change from baseline. ECG: Electrocardiogram. HR: Heart rate. QTCF: QT interval using Fridericia's correction formula.

Baseline: Defined as the assessment performed pre-dose for each treatment period.

Relative day: Relative to day of the first dose of study medication in each treatment period.

Relative to day of the grat dose of study medication seen the second precipe of the first dose of study medication in each treatment period.

Relative to day of the first dose of study medication in each treatment period.

Relative to day of the first dose of study medication in each treatment period.

Relative to day of the first dose of study medication in each treatment period.

Relative day: Relative to day of the first dose of study medication in each treatment period.

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.

Output ID: L025

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc

Listing 16.2.9.13 Vital Signs (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.13

Vital Signs

(Safety Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| CFB | x.xx | xx.x | x.xx | : |
|---|---|---|---|---|
| Baseline | XX.X | ×.×. | ×.×x | : |
| Result | xx.x | x.xx | x.xx | : |
| Vital sign<br>parameter (unit) | SBP (mmHg) | DBP (mmHg) | Pulse (beats/min) | : |
| Date/Time of assessment/Relative day | ррмммүүүү нн:мм/хх | | | DDMMMYYYY/HH:MM/xx |
| Treatment<br>period/<br>Timepoint | XXXXX | | | XXXXX |
| Treatment<br>group | XXXXX | | | |
| Patient<br>ID | XXXXXXXXXX | | | |

CFB: Change from baseline. DBP: Diastolic blood pressure. SBP: Systolic blood pressure.
Relative day: Relative to day of the first dose of study medication in each treatment period.
Baseline: Defined as the assessment performed pre-dose for each treatment period.
Baseline: Defined as the last available assessment assigned to study.
Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo Seq 2 = RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg/RPL554 300 mcg/RPL

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L026

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.9.14 Vital Signs - Patients with at Least One Markedly Abnormal Finding (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.14

Vital Signs - Patients with at Least One Markedly Abnormal Finding

(Safety Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| NM-HH/AAAAMMUU |
|----------------|
| XXXXX |

CFB: Change from baseline. DBP: Diastolic Blood Pressure. SBP: Systolic Blood Pressure.

Relative day: Relative to day of the first dose of study medication in each treatment period.

Land H represents marked decrease or increase from baseline.

Baseline: Defined as the assessment performed pre-dose for each treatment period.

End of Study. Defined as the last available assessment assigned to study.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3000 mcg. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL554 300 mcg. Seq 3 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period. Only include subjects who have a markedly abnormal finding.

Output ID: L035

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Author: Jennifer Allsopp

Listing 16.2.9.15 Derived Safety Measurements (Safety Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.15

(Safety Analysis Set in Part B) Derived Safety Measurements

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

Peak Pulse Rate (bpm) (over 4 XXXXX Date/ Relative day DDMMMYYYY/xx Treatment period Treatment XXXXX XXXXXXXXXX Patient

DDMMMYYYY/xx XXXXX

Peak = Maximum post-dose value among the values collected up to timepoint of interest hours.

Relative day: Relative to day of the first dose of study medication in each treatment period.

Baseline: Defined as the assessment performed pre-dose for each treatment period.

End of Study: Defined as the last available assessment assigned to study.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL554 300 mcg. Seq 3 = RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L035

[Source: Filepath\Filename.sas] IQVIA DDMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc

Listing 16.2.9.16 Brief Physical Examination (Safety Analysis Set in Part B) Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

(Safety Analysis Set in Part B) Brief Physical Examination Listing 16.2.9.16

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | Result (if Abnormal, clinical | significant), Specify | XXXXXXXXXXXX |
|---|---|---|---|
| | | Body system | XXXXXXXXXXXXX |
| Date/Time of | examination/ | Relative day | DDMMMYYYY / HH; MM/xx |
| | | Visit | XXXXX |
| | Treatment | dnoxb | XXXXX |
| | Patient | ID | XXXXXXXXXX |

Relative day: Relative to day of the first dose of study medication in each treatment period.

BOS: End of Study, defined as the last available assessment assigned to study.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 3

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L027

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Listing 16.2.9.17 Full Physical Examination (Safety Analysis Set in Part B)

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.17

Part B Page X of Y

> (Safety Analysis Set in Part B) Full Physical Examination

> > Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| | bnormal, clinical | , Specify | XX |
|--------------|-------------------|---------------|--------------------|
| | Result (if A | significant), | XXXXXXXXXXXX |
| | | Body system | XXXXXXXXXXXX |
| Date/Time of | examination/ | Relative day | DDMMMYYYY/HH:MM/xx |
| | | Visit | XXXXX |
| | Treatment | dronb | XXXXX |
| | Patient | ID | XXXXXXXXXXX |

Relative day: Relative to day of the first dose of study medication in each treatment period.

BOS: End of Study, defined as the last wavilable assessment assigned to study.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID and treatment period.

Output ID: L027

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Version: 2.0 Date: 22JAN2021 Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B

Listing 16.2.9.18 Inhalation Training (All Randomized Analysis Set in Part B) Verona Pharma

Page X of Y Part B

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Inhalation Training Listing 16.2.9.18

(All Randomized Analysis Set in Part B)

Treatment sequence: <Seq 1/Seq 2/Seq 3/Seq 4>

| ation training/ | | |
|---------------------|---------------|--------------|
| | אפדמרדיים ממץ | DDMMMYYYY/xx |
| Inhalation training | drven: | XXXXXXX |
| Treatment | FELLOG | XXXXXXX |
| | ratient in | XXXXXXX |

Relative day: Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/PPlacebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL554 3000 mcg/RPL554 300 mcg.

Programming Notes

Order by treatment sequence (as per shell) and within group by patient ID.

Output ID: L013

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Listing 16.2.9.19 Pregnancy Urine Test Results (All Randomized Analysis Set in Part B)

Page X of Y Part B

Verona Pharma

Protocol: RPL554-MD-201

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.19

Pregnancy Urine Test Results

(All Randomized Analysis Set in Part B)

Treatment seguence: <Seg 1/Seg 2/Seg 3/Seg 4>

| Patient ID | Treatment<br>Group | Treatment Period | Urine pregnancy test performed/Date of test/Relative day | Urine pregnancy test<br>result |
|---|---|---|---|---|
| XXXXXX | XXXXXXXXX | XXXXXXX | XX/DDMMMYYYY/xx | XXXXXXX |

Relative day: Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/RPL554 1000 mcg/RPL554 1000 mcg/RPL554 300 mcg/RPL5

Programming Notes

Order by treatment group (as per shell) and within group by patient ID.

Consider only female patients.

Multiple pregnancy risk factors and multiple relevant family history will be presented as one result per row, as these are not presented spearately in Pregnancy report eCRF.

Output ID: L036

[Source: Filepath\Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAP\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp


Listing 16.2.9.20 Pregnancy Report Results (All Randomized Analysis Set in Part B)

Protocol: RPL554-MD-201 Verona Pharma

Page X of Y Part B

RPL554 pressurised Metered Dose Inhaler

Listing 16.2.9.20

Pregnancy Report Results

(All Randomized Analysis Set in Part B)

| Treatment sequence: <seq 1="" 2="" 3="" 4="" seq=""></seq> | | |
|---|---|---|
| Patient ID | Pregnancy report item | Results |
| XXXXXXXXXXXXX | Date of last menstrual period/Relative day | DDMMYYYY/xx |
| | Date of expected delivery/Relative day | DDMMYYYY/xx |
| | Overall number of previous pregnancies | XX |
| | Number of normal deliveries | XX |
| | Number of spontaneous miscarriages | XX |
| | Number of other previous pregnancies | XX |
| | Relevant pregnancy risk factors | XXXXXXXXX |
| | Relevant family history | XXXXXXXX |

Relative day: Relative to day of the first dose of study medication in each treatment period.

Seq 1 = RPL554 300 mcg/RPL554 1000 mcg/RPL554 3000 mcg/Placebo. Seq 2 = RPL554 1000 mcg/RPL554 300 mcg/RPL554 3000 mcg/RPL554 300 mcg/RP

Programming Notes

Order by treatment group (as per shell) and within group by patient ID. Consider only female patients. Williets factors and multiple relevant family history will be presented as one result per row, as these are not presented separately in Pregnancy report eCRF.

Output ID: L037

[Source: Filepath/Filename.sas] IQVIA DDMMMYYYY HH:MM

Document: \\ieedc-vnasc01\biosdata\Verona\_Pharma\RPL554\EZAA8488\Biostatistics\Documentation\SAF\Verona RPL554-MD-201 TLF Shells v2.0 - Part B


Author: Jennifer Allsopp

CONFIDENTIAL Verona Pharma plc